CLINICAL TRIAL: NCT02938520
Title: A Phase III, Randomized, Multicenter, Parallel-group, Open-Label Study Evaluating the Efficacy, Safety, and Tolerability of Long-Acting Intramuscular Cabotegravir and Rilpivirine for Maintenance of Virologic Suppression Following Switch From an Integrase Inhibitor Single Tablet Regimen in HIV-1 Infected Antiretroviral Therapy Naive Adult Participants
Brief Title: Study to Evaluate the Efficacy, Safety, and Tolerability of Long-acting Intramuscular Cabotegravir and Rilpivirine for Maintenance of Virologic Suppression Following Switch From an Integrase Inhibitor in HIV-1 Infected Therapy Naive Participants
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Janssen Pharmaceuticals (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201584; 2016-001646-25 (EudraCT Number)
Record Dates: First submitted 2016-09-15; First posted 2016-10-19 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
Keywords: Antiretroviral agent; Maintenance; rilpivirine; dolutegravir; TMC278; Triumeq; non-nucleoside reverse transcriptase inhibitor; once monthly, every 4 weeks, once daily; GSK1265744; CAB; Tivicay; Long-Acting Intramuscular rilpivirine; lamivudine; integrase inhibitor; Long-Acting Intramuscular Cabotegravir; ART naïve; cabotegravir; abacavir
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Rilpivirine; dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CAB LA + RPV LA every 4 weeks (Experimental): After Induction Phase with ABC/DTG/3TC (or DTG + two NRTIs), eligible participants will receive oral CAB 30 mg + RPV 25 mg once daily for approximately four weeks. At visit Week 4b subjects will receive an initial loading dose of CAB LA (600 mg) and RPV LA (900 mg) at Week 4b. From Week 8 onwards, subjects will receive CAB LA (400 mg) + RPV LA (600 mg) injections every 4 weeks.
  Interventions: Drug: Cabotegravir (CAB) tablet; Drug: Rilpivirine (RPV) tablet; Drug: Cabotegravir - Injectable Suspension (CAB LA); Drug: Rilpivirine - Injectable Suspension (RPV LA)
- ABC / DTG / 3TC (600 mg/50mg/300mg) once daily (Active Comparator): After the Induction Phase with ABC/DTG/3TC (or DTG + two NRTIs), eligible participants will continue to receive oral ABC/DTG/3TC (or DTG + two NRTIs) initiated during the Induction Phase for 100 weeks. At the end of the Maintenance Phase, eligible participants receiving ABC/DTG/3TC (or DTG + two NRTIs) have the option to continue in the study by switching to CAB LA + RPV LA in the Extension Phase. These participants will transition to LA dosing at either Week 100 (direct to inject) or Week 104b (if using optional oral lead-in with CAB 30 mg + RPV 25 mg once daily).
  Interventions: Drug: ABC/DTG/3TC STR - Tablet; Drug: DTG Tablet

INTERVENTIONS:
Drug: Cabotegravir (CAB) tablet — It is a white oval shaped film coated 30 mg tablets for oral administration. CAB Tablet is composed of cabotegravir sodium, lactose monohydrate, microcrystalline cellulose, hypromellose, sodium starch glycolate, magnesium stearate, and white film-coat.
  Arms: CAB LA + RPV LA every 4 weeks
Drug: Rilpivirine (RPV) tablet — It is a 25 mg tablet with off-white, round, biconvex, film-coated and debossed on one side with "TMC" and the other side with "25". Each tablet contains RPV hydrochloride, and the inactive ingredients croscarmellose sodium, lactose monohydrate, magnesium stearate, polysorbate 20, povidone K30 and silicified microcrystalline cellulose.
  Arms: CAB LA + RPV LA every 4 weeks
Drug: Cabotegravir - Injectable Suspension (CAB LA) — It is a sterile white to slightly pink suspension containing 200 mg/mL of CAB as free acid for administration by intramuscular (IM) injection. Each vial is for single-dose use containing a withdrawable volume of 2.0 mL, and does not require dilution prior to administration. CAB LA is composed of cabotegravir free acid, polysorbate 20, polyethylene glycol 3350, mannitol, and water for injection.
  Arms: CAB LA + RPV LA every 4 weeks
Drug: Rilpivirine - Injectable Suspension (RPV LA) — It is a sterile white suspension containing 300 mg/mL of RPV as the free base. The route of administration is by intramuscular (IM) injection. Each vial contains a nominal fill of 2.0 mL, and does not require dilution prior to administration. RPV LA requires refrigeration and must be protected from light. RPV LA is composed of RPV free base, poloxamer 338, sodium dihydrogen phosphate monohydrate, citric acid monohydrate, glucose monohydrate, sodium hydroxide, water for injection.
  Arms: CAB LA + RPV LA every 4 weeks
Drug: ABC/DTG/3TC STR - Tablet — It is a purple, biconvex, oval, tablet debossed with "572 Tri" on one side, film-coated tablet contains abacavir sulphate equivalent to 600 mg of abacavir, dolutegravir sodium equivalent to 50 mg dolutegravir, and 300 mg of lamivudine. The inactive ABC/DTG/3TC tablet ingredients include D-mannitol, magnesium stearate, microcrystalline cellulose, povidone, and sodium starch glycolate.
  Arms: ABC / DTG / 3TC (600 mg/50mg/300mg) once daily
Drug: DTG Tablet — It is a yellow, round, biconvex, 50 mg film-coated tablet debossed with "SV 572" on one side and "50" on the other side. Each tablet of DTG also contains the following inactive ingredients: D-mannitol, microcrystalline cellulose, povidone K29/32, sodium starch glycolate, and sodium stearyl fumarate.
  Arms: ABC / DTG / 3TC (600 mg/50mg/300mg) once daily

SUMMARY:
The First Long-Acting Injectable Regimen (FLAIR) study is being conducted to establish if human immunodeficiency virus type-1 (HIV-1) infected adult participants whose virus is virologically suppressed on an integrase inhibitor single tablet regimen (INI STR) will remain suppressed after switching to a two-drug intramuscular (IM) long-acting (LA) regimen of cabotegravir (CAB) and rilpivirine (RPV). In this study, the INI STR will be limited to abacavir/dolutegravir/lamivudine (ABC/DTG/3TC). FLAIR is a Phase 3, multi-phase, randomized, open label, active-controlled, multicenter, parallel-group, non-inferiority study in HIV-1, anti-retroviral therapy (ART)-naïve adult participants. This study is designed to demonstrate the non-inferior antiviral activity of switching to a two drug CAB LA 400 mg + RPV LA 600 mg regimen every 4 weeks (Q4W: monthly) compared to remaining on ABC/DTG/3TC over 48 weeks (4 weeks oral CAB + RPV, 44 weeks LA therapy). Participants who are HLA-B*5701 positive at Screening may enroll into the study and receive DTG plus a non-abacavir containing dual nucleoside reverse transcriptase inhibitor (NRTI) regimen. Eligible participants will enroll into the Induction Phase of the study and receive ABC/DTG/3TC for 20 weeks (Week [-20] to Day 1). Participants who have an HIV 1 ribose nucleic acid (RNA) <50 copies per milliliter (c/mL) at Week (-4) will be randomized (1:1) into the Maintenance Phase at Day 1 to either continue ABC/DTG/3TC or to discontinue ABC/DTG/3TC and begin oral therapy with CAB 30 mg + RPV 25 mg once daily for approximately 4 Weeks, followed by monthly CAB LA + RPV LA injections from visit Week 4b until study completion or withdrawal. Participants who successfully complete Week 100 (without meeting study defined withdrawal criteria and who remain virologically suppressed through Week 96: HIV-1 RNA <50 c/mL) will be given the option to switch to the LA arm in the Extension Phase (using an optional oral lead-in with CAB + RPV) or be withdrawn from the study. Participants will continue to receive injections every 4 weeks during the Extension Phase until CAB LA and RPV LA are either locally approved and commercially available, the participant no longer derives clinical benefit, the participant meets a protocol-defined reason for discontinuation, or until development of either CAB LA or RPV LA is terminated.

ELIGIBILITY:
Inclusion Criteria: - HIV-1 infected, ART-naive men or women aged 18 years or greater at the time of signing the informed consent. - HIV-1 infection as documented by Screening plasma HIV-1 RNA >=1000 c/mL; - Antiretroviral-naive (<=10 days of prior therapy with any antiretroviral agent following a diagnosis of HIV-1 infection). Any previous exposure to an HIV integrase inhibitor or non-nucleoside reverse transcriptase inhibitor will be exclusionary. - Female Participants: A female participant is eligible to participate if she is not pregnant at Screening and first day of Induction Phase (as confirmed by a negative serum human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies: Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation; Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; Hysterectomy; Documented Bilateral Oophorectomy; Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication, throughout the study, and for at least 30 days after discontinuation of all oral study medications and for at least 52 weeks after discontinuation of CAB LA and RPV LA. The investigator is responsible for ensuring that participants understand how to properly use these methods of contraception. All participants in the study should be counseled on safer sexual practices including the use and benefit/risk of effective barrier methods (e.g., male condom) and on the risk of HIV transmission to an uninfected partner. - Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol. - In France, a participant will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria: - Women who are pregnant, breastfeeding, or plan to become pregnant or breastfeed during the study. - Any evidence at Screening of an active Centers for Disease and Prevention Control (CDC) Stage 3 disease, except cutaneous Kaposi's sarcoma not requiring systemic therapy or historic or current cluster of differentiation4+ (CD4+) cell count <200 cells/ cubic millimeter (mm^3) are not exclusionary. - Participants with known moderate to severe hepatic impairment. - Any pre-existing physical or mental condition (including substance abuse disorder) which, in the opinion of the Investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant. - Participants determined by the Investigator to have a high risk of seizures, including participants with an unstable or poorly controlled seizure disorder. A participant with a prior history of seizure may be considered for enrolment if the Investigator believes the risk of seizure recurrence is low. All cases of prior seizure history should be discussed with the Medical Monitor prior to enrolment. - Participant who, in the investigator's judgment, poses a significant suicide risk. Participant's recent history of suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk. - The participant has a tattoo or other dermatological condition overlying the gluteus region which may interfere with interpretation of injection site reactions. - Evidence of Hepatitis B virus (HBV) infection based on the results of testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti HBc), Hepatitis B surface antibody (anti-HBs) and HBV dioxyribose nucleic acid (DNA) as follows: Participants positive for HBsAg are excluded; Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded. Note: Participants positive for anti-HBc (negative HBsAg status) and positive for anti-HBs (past and/or current evidence) are immune to HBV and are not excluded. - Asymptomatic individuals with chronic hepatitis C virus (HCV) infection will not be excluded, however Investigators must carefully assess if therapy specific for HCV infection is required; participants who are anticipated to require HCV treatment prior to Week 48 of the Maintenance Phase must be excluded. HCV treatment on study may be permitted post Week 48, following consultation with the Medical Monitor. Participants with HCV co-infection will be allowed entry into Phase 3 studies if: Liver enzymes meet entry criteria; HCV Disease has undergone appropriate work-up, HCV is not advanced, and will not require treatment prior to the Week 48 visit. Additional information (where available) on participants with HCV co-infection at screening should include results from any liver biopsy, fibroscan, ultrasound, or other fibrosis evaluation, history of cirrhosis or other decompensated liver disease, prior treatment, and timing/plan for HCV treatment. In the event that recent biopsy or imaging data is not available or is inconclusive, the Fib-4 score will be used to verify eligibility. A Fib-4 score > 3.25 is exclusionary; Fib-4 scores 1.45 - 3.25 requires Medical Monitor consultation. Fibrosis 4 Score Formula: (Age x AST)/(Platelets x [square root of ALT]). - Unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment). - History of liver cirrhosis with or without hepatitis viral co-infection. - Ongoing or clinically relevant pancreatitis. - All participants will be screened for syphilis (rapid plasma reagin [RPR]). Participants with untreated syphilis infection, defined as a positive RPR without clear documentation of treatment, are excluded. Participants with a positive RPR test who have not been treated may be rescreened at least 30 days after completion of antibiotic treatment for syphilis. - Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical, anal or penile intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the study Medical Monitor for inclusion of the participant prior to enrollment. - Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the drug or render the participant unable to receive study medication. - History or presence of allergy or intolerance to the study drugs or their components or drugs of their class. In addition, if heparin is used during pharmacokinetic sampling (PK) sampling, participants with a history of sensitivity to heparin or heparin-induced thrombocytopenia must not be enrolled. - Current or anticipated need for chronic anti-coagulation. - Alanine aminotransferase (ALT) >=3 times upper limit normal (ULN). - Clinically significant cardiovascular disease, as defined by history/evidence of congestive heart failure, symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease. - Exposure to an experimental drug and/or experimental vaccine within 28 days or 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of investigational product (IP). - Treatment with any of the following agents within 28 days of Screening: radiation therapy; cytotoxic chemotherapeutic agents; tuberculosis (TB) therapy, with the exception of treatment of latent TB with isoniazid; Immunomodulators that alter immune responses (such as chronic systemic corticosteroids, interleukins, or interferons). Note: Participants using short-term (e.g. =<21 day) systemic corticosteroid treatment, topical, inhaled or intranasal corticosteroids are eligible for enrollment. - Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening. - Treatment with any agent, except recognized ART as allowed above, with documented activity against HIV-1 within 28 days of the first dose of IP. - Use of medications which are associated with Torsades de Pointes - Any evidence of primary resistance to non-nuclease reverse transcriptase inhibitors (NNRTIs) (except for K103N which is allowed), or any known resistance to INIs from historical resistance test results. Note: re-tests of Screening genotypes are allowed only at the discretion of the study virologist. - Participants who are HLA-B*5701 positive and are unable to use an nuclease reverse transcriptase inhibitors (NRTI) backbone that does not contain abacavir (participants who are HLA-B*5701 positive may be enrolled if they use a NRTI backbone that does not contain abacavir; HLA-B*5701 positive participants may be excluded from the study if local provision of an alternate NRTI backbone is not possible). - Any verified Grade 4 laboratory abnormality. A single repeat test is allowed during the Screening Phase to verify a result. - Any acute laboratory abnormality at Screening, which, in the opinion of the Investigator, would preclude the participant's participation in the study of an investigational compound. - Participant has estimated creatinine clearance <50 mL/min/1.73m^2 via the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation. - Participants who are currently participating in or anticipate to be selected for any other interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (85):
- United States (24):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Camden, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, Lynchburg, Virginia
- Canada (4):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (4):
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
- Germany (7):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Bonn
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Hanover
  - GSK Investigational Site, München
- Italy (4):
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Monza MB
  - GSK Investigational Site, Roma
- Japan (3):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Netherlands (4):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Utrecht
- Russia (11):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Lipetsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Oryol
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Toliyatti
  - GSK Investigational Site, Yekaterinburg
- South Africa (7):
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Middelburg
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Winnie Mandela
- Spain (13):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Elche Alicante
  - GSK Investigational Site, Ferrol
  - GSK Investigational Site, Granada
  - GSK Investigational Site, La Laguna Santa Cruz
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, San SebastiAn de Los Rey
  - GSK Investigational Site, Santa Cruz de Tenerife
  - GSK Investigational Site, Santander
- United Kingdom (4):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Coventry
  - GSK Investigational Site, Leeds Yorkshire
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20364

REFERENCES:
- [Background] Orkin C, Arasteh K, Gorgolas Hernandez-Mora M, Pokrovsky V, Overton ET, Girard PM, Oka S, Walmsley S, Bettacchi C, Brinson C, Philibert P, Lombaard J, St Clair M, Crauwels H, Ford SL, Patel P, Chounta V, D'Amico R, Vanveggel S, Dorey D, Cutrell A, Griffith S, Margolis DA, Williams PE, Parys W, Smith KY, Spreen WR. Long-Acting Cabotegravir and Rilpivirine after Oral Induction for HIV-1 Infection. N Engl J Med. 2020 Mar 19;382(12):1124-1135. doi: 10.1056/NEJMoa1909512. Epub 2020 Mar 4. PMID 32130806
- [Derived] D'Amico R, Han K, Min S, DeMoor R, St Clair M, Ford SL, Harrington C, Bernal-Morell E, Lombaard J, Crauwels H, Kolobova I, Patel N, Jamil N, Van Solingen-Ristea R, Acuipil C, Spreen W. Subcutaneous injections of cabotegravir plus rilpivirine long-acting in virally suppressed adults with HIV-1. AIDS. 2025 Dec 1;39(15):2182-2190. doi: 10.1097/QAD.0000000000004310. Epub 2025 Oct 21. PMID 40779489
- [Derived] Okesanya OJ, Ayeni RA, Amadin P, Ngwoke I, Amisu BO, Ukoaka BM, Ahmed MM, Oso TA, Musa SS, Lucero-Prisno DE. Advances in HIV Treatment and Vaccine Development: Emerging Therapies and Breakthrough Strategies for Long-Term Control. AIDS Res Treat. 2025 Jul 4;2025:6829446. doi: 10.1155/arat/6829446. eCollection 2025. PMID 40655875
- [Derived] Elliot ER, Polli JW, Patel P, Garside L, Grove R, Barnett V, Roberts J, Byrapuneni S, Crauwels H, Ford SL, Van Solingen-Ristea R, Birmingham E, D'Amico R, Baugh B, van Wyk J. Efficacy, Safety, and Pharmacokinetics by Body Mass Index Category in Phase 3/3b Long-Acting Cabotegravir Plus Rilpivirine Trials. J Infect Dis. 2024 Jul 25;230(1):e34-e42. doi: 10.1093/infdis/jiad580. PMID 39052748
- [Derived] Chounta V, Byrnes HF, Henry-Szatkowski M, Browning D, Donatti C, Lambert J. Psychometric Validation of the Perception of Injection (PIN) Questionnaire Using Data From Two Phase III, Open-Label, Active-Controlled, Non-Inferiority Studies in People Living With HIV. Adv Ther. 2023 Dec;40(12):5300-5314. doi: 10.1007/s12325-023-02656-1. Epub 2023 Sep 30. PMID 37776478
- [Derived] Moreno S, Rivero A, Ventayol P, Falco V, Torralba M, Schroeder M, Neches V, Vallejo-Aparicio LA, Mackenzie I, Turner M, Harrison C. Cabotegravir and Rilpivirine Long-Acting Antiretroviral Therapy Administered Every 2 Months is Cost-Effective for the Treatment of HIV-1 in Spain. Infect Dis Ther. 2023 Aug;12(8):2039-2055. doi: 10.1007/s40121-023-00840-y. Epub 2023 Jul 14. PMID 37452174
- [Derived] Masia M, Fernandez-Gonzalez M, Agullo V, Mascarell P, Padilla S, Garcia-Abellan J, Gutierrez F. Human Immunodeficiency Virus Type 1 RNA Levels in Rectal and Seminal Compartments After Switching to Long-Acting Cabotegravir Plus Rilpivirine: A Longitudinal Study. Clin Infect Dis. 2023 Feb 8;76(3):e748-e751. doi: 10.1093/cid/ciac676. PMID 35986671
- [Derived] Chounta V, Snedecor SJ, Wu S, Van de Velde N. Indirect comparison of 48-week efficacy and safety of long-acting cabotegravir and rilpivirine maintenance every 8 weeks with daily oral standard of care antiretroviral therapy in participants with virologically suppressed HIV-1-infection. BMC Infect Dis. 2022 May 4;22(1):428. doi: 10.1186/s12879-022-07243-3. PMID 35508986
- [Derived] Jeffrey JL, St Clair M, Wang P, Wang C, Li Z, Beloor J, Talarico C, Fridell R, Krystal M, White CT, Griffith S, D'Amico R, Smith K, Van Eygen V, Vingerhoets J, Vandermeulen K, Spreen W, van Lunzen J. Impact of Integrase Sequences from HIV-1 Subtypes A6/A1 on the In Vitro Potency of Cabotegravir or Rilpivirine. Antimicrob Agents Chemother. 2022 Mar 15;66(3):e0170221. doi: 10.1128/AAC.01702-21. Epub 2022 Jan 3. PMID 34978890
- [Derived] Orkin C, Bernal Morell E, Tan DHS, Katner H, Stellbrink HJ, Belonosova E, DeMoor R, Griffith S, Thiagarajah S, Van Solingen-Ristea R, Ford SL, Crauwels H, Patel P, Cutrell A, Smith KY, Vandermeulen K, Birmingham E, St Clair M, Spreen WR, D'Amico R. Initiation of long-acting cabotegravir plus rilpivirine as direct-to-injection or with an oral lead-in in adults with HIV-1 infection: week 124 results of the open-label phase 3 FLAIR study. Lancet HIV. 2021 Nov;8(11):e668-e678. doi: 10.1016/S2352-3018(21)00184-3. Epub 2021 Oct 14. PMID 34656207
- [Derived] Orkin C, Oka S, Philibert P, Brinson C, Bassa A, Gusev D, Degen O, Garcia JG, Morell EB, Tan DHS, D'Amico R, Dorey D, Griffith S, Thiagarajah S, St Clair M, Van Solingen-Ristea R, Crauwels H, Ford SL, Patel P, Chounta V, Vanveggel S, Cutrell A, Van Eygen V, Vandermeulen K, Margolis DA, Smith KY, Spreen WR. Long-acting cabotegravir plus rilpivirine for treatment in adults with HIV-1 infection: 96-week results of the randomised, open-label, phase 3 FLAIR study. Lancet HIV. 2021 Apr;8(4):e185-e196. doi: 10.1016/S2352-3018(20)30340-4. PMID 33794181
- [Derived] Rizzardini G, Overton ET, Orkin C, Swindells S, Arasteh K, Gorgolas Hernandez-Mora M, Pokrovsky V, Girard PM, Oka S, Andrade-Villanueva JF, Richmond GJ, Baumgarten A, Masia M, Latiff G, Griffith S, Harrington CM, Hudson KJ, St Clair M, Talarico CL, Patel P, Cutrell A, Van Eygen V, D'Amico R, Mrus JM, Wu S, Ford SL, Chow K, Roberts J, Wills A, Walters N, Vanveggel S, Van Solingen-Ristea R, Crauwels H, Smith KY, Spreen WR, Margolis DA. Long-Acting Injectable Cabotegravir + Rilpivirine for HIV Maintenance Therapy: Week 48 Pooled Analysis of Phase 3 ATLAS and FLAIR Trials. J Acquir Immune Defic Syndr. 2020 Dec 1;85(4):498-506. doi: 10.1097/QAI.0000000000002466. PMID 33136751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-inferiority study evaluated antiviral activity of switching to intramuscular long acting carbotegravir (CAB) and rilpivirine (RPV) every 4 weeks compared to continuation of abacavir (ABC)/dolutegravir (DTG)/lamivudine (3TC) over 48 weeks in virologically suppressed participants with human immunodeficiency type 1 infection
Pre-assignment Details: A total of 631 participants were enrolled into the Induction Phase of the study. 566 participants were subsequently randomized. Two randomized participants did not receive study treatment. This study was conducted in 11 countries. The results presented are based on Week 48 primary analysis
Groups:
- CAB LA + RPV LA (Q4W): Participants who received ABC/DTG/3TC for 20 Weeks (Week [-20] to Day 1) in the Induction Phase and who have an HIV-1 ribonucleic acid (RNA) <50 copies per millilter (c/mL) at Week (-4) entered Maintenance Phase (Day 1 to Week 100) to begin oral therapy with CAB 30 milligram (mg) + RPV 25 mg once daily for 4 Weeks. At Week 4b visit, participants received last dose of oral CAB + RPV and first dose CAB LA 600 mg + RPV LA 900 mg injections. Participants received intramuscular (IM) injections of CAB LA 400 mg and RPV LA 600 mg at Week 8 and every four weeks (Q4W) through Week 100. After completion of Maintenance Phase, participants who chose to enter Extension Phase will continue to receive both CAB LA and RPV LA. Participants withdrawn from study treatment who received at least one CAB LA+RPV LA injection were required to enter a 52-week long term follow-up (LTFU) period.
- ABC/ DTG/ 3TC: During Maintenance Phase (Day 1 to Week 100), participants continued to receive ABC/DTG/3TC. After completion of Maintenance Phase, participants who chose to enter the Extension Phase have the option to complete the study or switch to CAB LA+RPV LA
Period: Overall Study
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Started | 283 | 283
Completed | 0 | 0
Not Completed | 283 | 283
Not completed — On-going at the time of analysis | 258 | 261
Not completed — Physician Decision | 2 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Protocol Violation | 0 | 1
Not completed — Lack of Efficacy | 5 | 3
Not completed — Adverse Event | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC | Total
Number analyzed (Participants) | 283 | 283 | 566
Age, Continuous [Mean (Standard Deviation); unit: Years] — Intent-to-Treat Exposed
  Years | 35.9 (10.17) | 36.0 (9.82) | 35.9 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants] — Intent-to-Treat Exposed
  Participants
    Female | 63 | 64 | 127
    Male | 220 | 219 | 439
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 3 | 6 | 9
  Asian-Central/South Asian Heritage | 2 | 1 | 3
  Asian-East Asian Heritage | 1 | 2 | 3
  Asian-South East Asian Heritage | 1 | 0 | 1
  Asian-Japanese Heritage | 8 | 12 | 20
  Black or African American | 47 | 56 | 103
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  White-Arabic/North African Heritage | 5 | 3 | 8
  White-White /Caucasian/European Heritage | 211 | 198 | 409
  Multiple | 4 | 3 | 7
  Missing | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Virologic Failure (HIV-1 Ribonucleic Acid [RNA] >=50 Copies Per Millilter [mL]) Using Snapshot Algorithm at Week 48
Description: Percentage of participants with virologic failure endpoint (HIV-1 RNA>=50 c/mL) as per Food and Drug Administration (FDA) snapshot algorithm at Week 48 was assessed to demonstrate the noninferior antiviral activity of switching to intramuscular (IM) CAB LA+RPV LA every 4 weeks compared to continuation of ABC/DTG/3TC regimen over 48 weeks in HIV-1 infected ARTexperienced participants. The HIV-1 RNA >=50 copies/mL per snapshot algorithm was determined by the last on-treatment HIV-1 RNA measurement within the Week 48 analysis visit window (+/- 6 weeks) or at time of discontinuation (if discontinuation occurred prior to Week 48 for reasons other than Adverse Event).
Time Frame: Week 48
Population: Intent-to treat exposed (ITT-E) participants included all randomized participants who received at least one dose of Investigational Product (IP) during the Maintenance Phase. Participants were analyzed according to the randomized treatment regardless of what treatment actually received.
Measure: Number; unit: Percentage of Participants
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Percentage of Participants | 2.1 | 2.5
Statistical Analysis 1: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Non-Inferiority — Non-inferiority in the proportion of participants with virologic failure at Week 48 (per FDA's snapshot algorithm for assessing HIV-1 RNA >=50 c/mL) can be concluded if the upper bound of a two-sided 95% confidence interval (CI) for the difference in failure rates between the two treatment arms (CAB - ABC/DTG/3TC) is less than 6%; Adjusted difference in proportion = -0.4, 95% CI 2-sided [-2.8 to 2.1]; Adjusted difference in proportion was based on Cochran-Mantel Haenszel stratified analysis adjusting for the following baseline stratification factors: sex at birth (Male, Female) and Induction Baseline (Week -20) HIV-1 RNA (<100,000 >=100,000 c/mL)

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL Using Snapshot Algorithm at Week 48
Description: Percentage of participants with plasma HIV-1 RNA <50 copies/mL at Week 48 using FDA snapshot algorithm was assessed to demonstrate antiviral and immunologic activity of switching to IM CAB LA+RPV LA every 4 weeks compared to continuation of ABC/DTG/3TC. The HIV-1 RNA <50 copies/mL per snapshot algorithm was determined by last on-treatment HIV-1 RNA measurement within the Week 48 analysis visit window (+/- 6 weeks). Participants with no data in the analysis window were classificated as non-responders.
Time Frame: Week 48
Population: ITT-E Population
Measure: Number; unit: Percentage of Participants
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Percentage of Participants | 94 | 93
Statistical Analysis 1: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Non-Inferiority — Non-inferiority in the proportion of participants with HIV-1 RNA<50 c/mL at Week 48 (per FDA's snapshot algorithm) can be concluded if the lower bound of a two-sided 95% confidence interval for the difference in success rates between the two treatment arms (CAB - ABC/DTG/3TC) is more than -10%; Adjusted difference in proportion = 0.4, 95% CI 2-sided [-3.7 to 4.5] — Adjusted difference in proportion was based on Cochran-Mantel Haenszel stratified analysis adjusting for the following baseline stratification factors: sex at birth (Male, Female) and Induction Baseline (Week -20) HIV-1 RNA (<100,000 >=100,000 c/mL)

3. Secondary Outcome: Number of Participants With HIV-1 RNA <200 Copies/mL Using Snapshot Algorithm at Week 48
Description: Percentage of participants with plasma HIV-1 RNA <200 copies/mL at Week 48 using the snapshot algorithm was assessed based on the antiviral and immunologic activity of switching to IM CAB LA+RPV LA every 4 weeks compared to continuation of ABC/DTG/3TC
Time Frame: Week 48
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Percentage of Participants | 94 [91 to 97] | 94 [91 to 97]

4. Secondary Outcome: Number of Participants With Confirmed Virologic Failure (CVF) During the Maintenance Phase
Description: The CVF is defined as rebound as indicated by two consecutive plasma HIV-1-RNA levels >=200 copies/mL after prior suppression to <200 copies/mL.
Time Frame: Week 48
Population: ITT-E Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Participants | 4 | 3

5. Secondary Outcome: Absolute Values for Plasma HIV-1 RNA at Week 48
Description: Plasma for quantitative HIV-1 RNA were collected at indicated time points. Logarithm to base 10 (log10) values for plasma HIV-1 RNA has been presented.
Time Frame: Week 48
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
log10 copies/mL | 1.513 (0.0954) | 1.518 (0.1152)

6. Secondary Outcome: Change From Baseline Values for Plasma HIV-1 RNA at Week 48
Description: Baseline value is defined as the last available recorded value up to and including the date of first Maintenance Phase dose of IP. Change from Baseline was defined as: HIV-1 RNA(log 10) at Week 48 minus HIV-1 RNA(log 10) at Baseline.
Time Frame: Baseline (Day 1) and at Week 48
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
log10 copies/mL | -0.006 (0.1026) | 0.001 (0.1435)

7. Secondary Outcome: Absolute Values for CD4+ Lymphocyte Count at Week 48
Description: Blood samples were collected and CD4+ cell count assessment by flow cyclometry was carried out to evaluate the immunologic activity of switching to IM CAB LA+RPV LA every 4 weeks compared to ABC/DTG/3TC
Time Frame: Week 48
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Cells per cubic millimeter | 703.2 (285.75) | 731.2 (272.49)

8. Secondary Outcome: Change From Baseline Values for CD4+ Lymphocyte Count at Week 48
Description: Blood samples were collected and CD4+ cell count assessment by flow cyclometry was carried out to evaluate the immunologic activity of switching to IM CAB LA+RPV LA every 4 weeks compared to ABC/DTG/3TC. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance Phase dose of IP. Change from Baseline was defined as post-dose visit value at Week 48 minus Maintenance Baseline value.
Time Frame: Baseline (Day 1) and Week 48
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Cells per cubic millimeter | 40.2 (195.17) | 79.9 (194.55)

9. Secondary Outcome: Number of Participants With Disease Progression
Description: Data for participants who experienced disease progression to Centers for Disease Control and Prevention (CDC) Stage III or death has been presented. CDC stage is derived according to lowest post baseline CD4+ T-lympohocyte count and/or occurrence of AIDS-defining conditons (per 2014 CDC criteria).
Time Frame: Day 1 up to an average of 59 weeks
Population: ITT-E Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Participants | 9 | 11

10. Secondary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence temporally associated with the use of a study treatment, whether or not considered related to study treatment. A SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per medical or scientific judgment. Safety Population: all randomized participants who received at least 1 dose of IP during maintenance phase and assessed according to actual treatment received. All Maintenance Phase AEs was presented including AEs with start date occurring on/after date of 1st dose of randomized treatment, up to and including start date of LTFU antiretroviral therapy for participants who discontinued from Q4W arm. Non-SAE counts in >=5% of participants within any arm is reported
Time Frame: Day 1 up to an average of 59 Weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Participants
  Any non-SAE | 252 | 138
  Any SAE | 18 | 12

11. Secondary Outcome: Number of Participants With Severity of Adverse Events
Description: Severity of adverse events (AEs) were defined as per The Division of acquired immuno deficiency syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table) Version 2.0, November 2014. Severity grades for AEs were as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (Potentially life-threatening) and Grade 5 were all deaths related to an AE. All Maintenance Phase adverse events have been presented, which includes AEs with start date occuring on or after the date of first dose of randomized study treatment, up to and including the start date of LTFU antiretroviral therapy for participants who discontinued from the Q4W arm.
Time Frame: Up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Participants
  Grade 1 | 93 | 119
  Grade 2 | 143 | 95
  Grade 3 | 23 | 10
  Grade 4 | 8 | 1
  Grade 5 | 0 | 0

12. Secondary Outcome: Absolute Values for Hematology Parameters Over Time Including Week 48: Basophils, Eosinophils, Leukocytes, Lymphocytes, Neutrophils, Monocytes, and Platelets
Description: Blood samples were collected for the analysis of hematology parameters including basophil, eosinophils, leukocytes, lymphocytes, neutrophils, monocytes, and platelets at indicated time points.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: 10^9 cells per Liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
10^9 cells per Liter
  Basophils, Baseline (Day 1), n=283, 283 | 0.022 (0.0124) | 0.022 (0.0138)
  Basophils, Week 4, n=277, 270: number analyzed (Participants) | 277 | 270
  Basophils, Week 4, n=277, 270 | 0.024 (0.0136) | 0.024 (0.0142)
  Basophils, Week 8, n=210, 272: number analyzed (Participants) | 210 | 272
  Basophils, Week 8, n=210, 272 | 0.023 (0.0135) | 0.023 (0.0122)
  Basophils, Week 12, n=267, 272: number analyzed (Participants) | 267 | 272
  Basophils, Week 12, n=267, 272 | 0.025 (0.0166) | 0.023 (0.0144)
  Basophils, Week 16, n=247, 259: number analyzed (Participants) | 247 | 259
  Basophils, Week 16, n=247, 259 | 0.030 (0.0212) | 0.028 (0.0209)
  Basophils, Week 20, n=247, 259: number analyzed (Participants) | 247 | 259
  Basophils, Week 20, n=247, 259 | 0.035 (0.0254) | 0.032 (0.0256)
  Basophils, Week 24, n=256, 260: number analyzed (Participants) | 256 | 260
  Basophils, Week 24, n=256, 260 | 0.037 (0.0245) | 0.036 (0.0256)
  Basophils, Week 28, n=239, 258: number analyzed (Participants) | 239 | 258
  Basophils, Week 28, n=239, 258 | 0.039 (0.0249) | 0.038 (0.0247)
  Basophils, Week 32, n=246, 263: number analyzed (Participants) | 246 | 263
  Basophils, Week 32, n=246, 263 | 0.044 (0.0254) | 0.038 (0.0246)
  Basophils, Week 36, n=250, 259: number analyzed (Participants) | 250 | 259
  Basophils, Week 36, n=250, 259 | 0.042 (0.0237) | 0.040 (0.0250)
  Basophils, Week 40, n=244, 245: number analyzed (Participants) | 244 | 245
  Basophils, Week 40, n=244, 245 | 0.041 (0.0248) | 0.041 (0.0252)
  Basophils, Week 44, n=249, 260: number analyzed (Participants) | 249 | 260
  Basophils, Week 44, n=249, 260 | 0.040 (0.0246) | 0.040 (0.0257)
  Basophils, Week 48, n=239, 258: number analyzed (Participants) | 239 | 258
  Basophils, Week 48, n=239, 258 | 0.038 (0.0214) | 0.038 (0.0246)
  Eosinophils, Baseline (Day 1), n=283, 283 | 0.142 (0.1238) | 0.141 (0.1449)
  Eosinophils, Week 4, n=277, 270: number analyzed (Participants) | 277 | 270
  Eosinophils, Week 4, n=277, 270 | 0.164 (0.1470) | 0.154 (0.1535)
  Eosinophils, Week 8, n=210, 272: number analyzed (Participants) | 210 | 272
  Eosinophils, Week 8, n=210, 272 | 0.169 (0.1401) | 0.150 (0.1393)
  Eosinophils, Week 12, n=267, 272: number analyzed (Participants) | 267 | 272
  Eosinophils, Week 12, n=267, 272 | 0.165 (0.1375) | 0.157 (0.1481)
  Eosinophils, Week 16, n=247, 259: number analyzed (Participants) | 247 | 259
  Eosinophils, Week 16, n=247, 259 | 0.177 (0.1538) | 0.162 (0.1434)
  Eosinophils, Week 20, n=247, 259: number analyzed (Participants) | 247 | 259
  Eosinophils, Week 20, n=247, 259 | 0.185 (0.1617) | 0.166 (0.1675)
  Eosinophils, Week 24, n=256, 260: number analyzed (Participants) | 256 | 260
  Eosinophils, Week 24, n=256, 260 | 0.193 (0.1591) | 0.172 (0.1518)
  Eosinophils, Week 28, n=239, 258: number analyzed (Participants) | 239 | 258
  Eosinophils, Week 28, n=239, 258 | 0.206 (0.1634) | 0.179 (0.1659)
  Eosinophils, Week 32, n=246, 263: number analyzed (Participants) | 246 | 263
  Eosinophils, Week 32, n=246, 263 | 0.206 (0.1779) | 0.169 (0.1466)
  Eosinophils, Week 36, n=250, 259: number analyzed (Participants) | 250 | 259
  Eosinophils, Week 36, n=250, 259 | 0.209 (0.2043) | 0.172 (0.1540)
  Eosinophils, Week 40, n=244, 245: number analyzed (Participants) | 244 | 245
  Eosinophils, Week 40, n=244, 245 | 0.203 (0.1837) | 0.174 (0.1495)
  Eosinophils, Week 44, n=249, 260: number analyzed (Participants) | 249 | 260
  Eosinophils, Week 44, n=249, 260 | 0.198 (0.1867) | 0.180 (0.1723)
  Eosinophils, Week 48, n=239, 258: number analyzed (Participants) | 239 | 258
  Eosinophils, Week 48, n=239, 258 | 0.182 (0.1508) | 0.172 (0.1533)
  Leukocytes, Baseline (Day 1), n=283, 283 | 5.82 (1.792) | 5.68 (1.684)
  Leukocytes, Week 4, n=279, 272: number analyzed (Participants) | 279 | 272
  Leukocytes, Week 4, n=279, 272 | 6.41 (1.989) | 6.11 (1.770)
  Leukocytes, Week 8, n=211, 275: number analyzed (Participants) | 211 | 275
  Leukocytes, Week 8, n=211, 275 | 6.04 (1.806) | 6.00 (1.714)
  Leukocytes, Week 12, n=270, 275: number analyzed (Participants) | 270 | 275
  Leukocytes, Week 12, n=270, 275 | 5.88 (1.590) | 6.08 (1.836)
  Leukocytes, Week 16, n=252, 265: number analyzed (Participants) | 252 | 265
  Leukocytes, Week 16, n=252, 265 | 6.08 (2.045) | 6.11 (1.887)
  Leukocytes, Week 20, n=254, 265: number analyzed (Participants) | 254 | 265
  Leukocytes, Week 20, n=254, 265 | 6.08 (1.788) | 6.15 (1.926)
  Leukocytes, Week 24, n=258, 264: number analyzed (Participants) | 258 | 264
  Leukocytes, Week 24, n=258, 264 | 6.11 (1.841) | 6.16 (2.046)
  Leukocytes, Week 28, n=244, 263: number analyzed (Participants) | 244 | 263
  Leukocytes, Week 28, n=244, 263 | 6.17 (1.929) | 6.17 (1.939)
  Leukocytes, Week 32, n=253, 266: number analyzed (Participants) | 253 | 266
  Leukocytes, Week 32, n=253, 266 | 6.07 (1.925) | 6.12 (1.918)
  Leukocytes, Week 36, n=252, 259: number analyzed (Participants) | 252 | 259
  Leukocytes, Week 36, n=252, 259 | 6.11 (1.992) | 6.23 (2.104)
  Leukocytes, Week 40, n=246, 253: number analyzed (Participants) | 246 | 253
  Leukocytes, Week 40, n=246, 253 | 5.96 (1.773) | 6.12 (2.076)
  Leukocytes, Week 44, n=256, 262: number analyzed (Participants) | 256 | 262
  Leukocytes, Week 44, n=256, 262 | 6.03 (2.000) | 6.19 (1.970)
  Leukocytes, Week 48, n=243, 260: number analyzed (Participants) | 243 | 260
  Leukocytes, Week 48, n=243, 260 | 5.85 (1.884) | 5.99 (1.986)
  Lymphocytes, Baseline (Day 1), n=283, 283 | 2.022 (0.6893) | 1.957 (0.6408)
  Lymphocytes, Week 4, n=277, 270: number analyzed (Participants) | 277 | 270
  Lymphocytes, Week 4, n=277, 270 | 2.227 (0.7321) | 2.197 (0.7198)
  Lymphocytes, Week 8, n=210, 272: number analyzed (Participants) | 210 | 272
  Lymphocytes, Week 8, n=210, 272 | 2.102 (0.6980) | 2.110 (0.7015)
  Lymphocytes, Week 12, n=267, 272: number analyzed (Participants) | 267 | 272
  Lymphocytes, Week 12, n=267, 272 | 2.032 (0.6095) | 2.117 (0.7162)
  Lymphocytes, Week 16, n=247, 259: number analyzed (Participants) | 247 | 259
  Lymphocytes, Week 16, n=247, 259 | 2.028 (0.6931) | 2.130 (0.7245)
  Lymphocytes, Week 20, n=247, 259: number analyzed (Participants) | 247 | 259
  Lymphocytes, Week 20, n=247, 259 | 2.028 (0.6284) | 2.121 (0.6995)
  Lymphocytes, Week 24, n=256, 260: number analyzed (Participants) | 256 | 260
  Lymphocytes, Week 24, n=256, 260 | 2.014 (0.6456) | 2.111 (0.7092)
  Lymphocytes, Week 28, n=239, 258: number analyzed (Participants) | 239 | 258
  Lymphocytes, Week 28, n=239, 258 | 2.051 (0.6592) | 2.106 (0.6679)
  Lymphocytes, Week 32, n=246, 263: number analyzed (Participants) | 246 | 263
  Lymphocytes, Week 32, n=246, 263 | 2.037 (0.6543) | 2.112 (0.6950)
  Lymphocytes, Week 36, n=250, 259: number analyzed (Participants) | 250 | 259
  Lymphocytes, Week 36, n=250, 259 | 2.023 (0.6878) | 2.098 (0.6921)
  Lymphocytes, Week 40, n=244, 245: number analyzed (Participants) | 244 | 245
  Lymphocytes, Week 40, n=244, 245 | 2.021 (0.6646) | 2.030 (0.6357)
  Lymphocytes, Week 44, n=249, 260: number analyzed (Participants) | 249 | 260
  Lymphocytes, Week 44, n=249, 260 | 1.997 (0.6748) | 2.068 (0.6754)
  Lymphocytes, Week 48, n=239, 258: number analyzed (Participants) | 239 | 258
  Lymphocytes, Week 48, n=239, 258 | 1.926 (0.6126) | 2.003 (0.7651)
  Monocytes, Baseline (Day 1), n=283, 283 | 0.382 (0.1666) | 0.366 (0.1705)
  Monocytes, Week 4, n=277, 270: number analyzed (Participants) | 277 | 270
  Monocytes, Week 4, n=277, 270 | 0.422 (0.1778) | 0.398 (0.1778)
  Monocytes, Week 8, n=210, 272: number analyzed (Participants) | 210 | 272
  Monocytes, Week 8, n=210, 272 | 0.415 (0.1824) | 0.380 (0.1771)
  Monocytes, Week 12, n=267, 272: number analyzed (Participants) | 267 | 272
  Monocytes, Week 12, n=267, 272 | 0.395 (0.1662) | 0.383 (0.1570)
  Monocytes, Week 16, n=247, 259: number analyzed (Participants) | 247 | 259
  Monocytes, Week 16, n=247, 259 | 0.438 (0.1859) | 0.409 (0.1810)
  Monocytes, Week 20, n=247, 259: number analyzed (Participants) | 247 | 259
  Monocytes, Week 20, n=247, 259 | 0.455 (0.1927) | 0.423 (0.1904)
  Monocytes, Week 24, n=256, 260: number analyzed (Participants) | 256 | 260
  Monocytes, Week 24, n=256, 260 | 0.438 (0.1859) | 0.438 (0.1897)
  Monocytes, Week 28, n=239, 258: number analyzed (Participants) | 239 | 258
  Monocytes, Week 28, n=239, 258 | 0.471 (0.1916) | 0.447 (0.2003)
  Monocytes, Week 32, n=246, 263: number analyzed (Participants) | 246 | 263
  Monocytes, Week 32, n=246, 263 | 0.462 (0.1898) | 0.459 (0.2107)
  Monocytes, Week 36, n=250, 259: number analyzed (Participants) | 250 | 259
  Monocytes, Week 36, n=250, 259 | 0.458 (0.2116) | 0.456 (0.2021)
  Monocytes, Week 40, n=244, 245: number analyzed (Participants) | 244 | 245
  Monocytes, Week 40, n=244, 245 | 0.438 (0.1740) | 0.442 (0.2038)
  Monocytes, Week 44, n=249, 260: number analyzed (Participants) | 249 | 260
  Monocytes, Week 44, n=249, 260 | 0.440 (0.1907) | 0.428 (0.1965)
  Monocytes, Week 48, n=239, 258: number analyzed (Participants) | 239 | 258
  Monocytes, Week 48, n=239, 258 | 0.402 (0.1911) | 0.396 (0.1857)
  Neutrophils, Baseline (Day 1), n=283, 283 | 3.246 (1.3715) | 3.205 (1.2803)
  Neutrophils, Week 4, n=277, 270: number analyzed (Participants) | 277 | 270
  Neutrophils, Week 4, n=277, 270 | 3.573 (1.5681) | 3.342 (1.3344)
  Neutrophils, Week 8, n=210, 272: number analyzed (Participants) | 210 | 272
  Neutrophils, Week 8, n=210, 272 | 3.334 (1.3166) | 3.316 (1.3588)
  Neutrophils, Week 12, n=267, 272: number analyzed (Participants) | 267 | 272
  Neutrophils, Week 12, n=267, 272 | 3.271 (1.2151) | 3.379 (1.4884)
  Neutrophils, Week 16, n=247, 259: number analyzed (Participants) | 247 | 259
  Neutrophils, Week 16, n=247, 259 | 3.410 (1.7208) | 3.432 (1.5052)
  Neutrophils, Week 20, n=247, 259: number analyzed (Participants) | 247 | 259
  Neutrophils, Week 20, n=247, 259 | 3.406 (1.4209) | 3.433 (1.5620)
  Neutrophils, Week 24, n=256, 260: number analyzed (Participants) | 256 | 260
  Neutrophils, Week 24, n=256, 260 | 3.428 (1.4938) | 3.424 (1.6766)
  Neutrophils, Week 28, n=239, 258: number analyzed (Participants) | 239 | 258
  Neutrophils, Week 28, n=239, 258 | 3.439 (1.5379) | 3.423 (1.5514)
  Neutrophils, Week 32, n=246, 263: number analyzed (Participants) | 246 | 263
  Neutrophils, Week 32, n=246, 263 | 3.367 (1.5670) | 3.392 (1.4892)
  Neutrophils, Week 36, n=250, 259: number analyzed (Participants) | 250 | 259
  Neutrophils, Week 36, n=250, 259 | 3.388 (1.5215) | 3.468 (1.6269)
  Neutrophils, Week 40, n=244, 245: number analyzed (Participants) | 244 | 245
  Neutrophils, Week 40, n=244, 245 | 3.274 (1.3654) | 3.477 (1.7021)
  Neutrophils, Week 44, n=249, 260: number analyzed (Participants) | 249 | 260
  Neutrophils, Week 44, n=249, 260 | 3.398 (1.5679) | 3.503 (1.5486)
  Neutrophils, Week 48, n=239, 258: number analyzed (Participants) | 239 | 258
  Neutrophils, Week 48, n=239, 258 | 3.309 (1.4923) | 3.419 (1.5186)
  Platelets, Baseline (Day 1), n=283, 282: number analyzed (Participants) | 283 | 282
  Platelets, Baseline (Day 1), n=283, 282 | 226.7 (55.39) | 230.6 (58.33)
  Platelets, Week 4, n=278, 269: number analyzed (Participants) | 278 | 269
  Platelets, Week 4, n=278, 269 | 233.1 (56.85) | 233.4 (56.56)
  Platelets, Week 8, n=207, 273: number analyzed (Participants) | 207 | 273
  Platelets, Week 8, n=207, 273 | 226.9 (53.23) | 232.0 (56.31)
  Platelets, Week 12, n=269, 271: number analyzed (Participants) | 269 | 271
  Platelets, Week 12, n=269, 271 | 226.6 (55.07) | 235.5 (57.26)
  Platelets, Week 16, n=251, 263: number analyzed (Participants) | 251 | 263
  Platelets, Week 16, n=251, 263 | 225.5 (55.49) | 239.9 (70.40)
  Platelets, Week 20, n=255, 264: number analyzed (Participants) | 255 | 264
  Platelets, Week 20, n=255, 264 | 233.8 (60.98) | 243.4 (62.06)
  Platelets, Week 24, n=256, 261: number analyzed (Participants) | 256 | 261
  Platelets, Week 24, n=256, 261 | 233.9 (58.12) | 244.2 (59.95)
  Platelets, Week 28, n=245, 258: number analyzed (Participants) | 245 | 258
  Platelets, Week 28, n=245, 258 | 233.7 (61.56) | 247.2 (63.18)
  Platelets, Week 32, n=249, 262: number analyzed (Participants) | 249 | 262
  Platelets, Week 32, n=249, 262 | 235.0 (62.74) | 245.3 (60.25)
  Platelets, Week 36, n=248, 259: number analyzed (Participants) | 248 | 259
  Platelets, Week 36, n=248, 259 | 237.3 (58.56) | 248.1 (59.57)
  Platelets, Week 40, n=244, 254: number analyzed (Participants) | 244 | 254
  Platelets, Week 40, n=244, 254 | 233.9 (56.93) | 247.4 (63.85)
  Platelets, Week 44, n=254, 261: number analyzed (Participants) | 254 | 261
  Platelets, Week 44, n=254, 261 | 236.7 (58.18) | 249.5 (71.56)
  Platelets, Week 48, n=240, 255: number analyzed (Participants) | 240 | 255
  Platelets, Week 48, n=240, 255 | 232.8 (57.07) | 246.0 (70.35)

13. Secondary Outcome: Absolute Values for Hematology Parameters Over Time Including Week 48: Erythrocyte Mean Corpuscular Volume
Description: Blood samples were collected for the analysis of hematology parameter including erythrocyte mean corpuscular volume at indicated timepoints.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Femtoliters
  Baseline (Day 1), n=283, 283 | 94.8 (4.94) | 94.3 (5.69)
  Week 4, n=279, 273: number analyzed (Participants) | 279 | 273
  Week 4, n=279, 273 | 94.1 (4.77) | 94.6 (5.85)
  Week 8, n=211, 275: number analyzed (Participants) | 211 | 275
  Week 8, n=211, 275 | 92.3 (4.86) | 94.6 (5.78)
  Week 12, n=270, 275: number analyzed (Participants) | 270 | 275
  Week 12, n=270, 275 | 91.0 (4.64) | 94.0 (5.81)
  Week 16, n=254, 265: number analyzed (Participants) | 254 | 265
  Week 16, n=254, 265 | 89.9 (4.43) | 94.1 (5.78)
  Week 20, n=255, 267: number analyzed (Participants) | 255 | 267
  Week 20, n=255, 267 | 89.3 (4.46) | 93.9 (5.64)
  Week 24, n=259, 264: number analyzed (Participants) | 259 | 264
  Week 24, n=259, 264 | 89.4 (4.33) | 93.8 (5.69)
  Week 28, n=246, 265: number analyzed (Participants) | 246 | 265
  Week 28, n=246, 265 | 89.3 (4.64) | 93.5 (5.78)
  Week 32, n=254, 267: number analyzed (Participants) | 254 | 267
  Week 32, n=254, 267 | 89.6 (4.69) | 93.6 (5.90)
  Week 36, n=252, 261: number analyzed (Participants) | 252 | 261
  Week 36, n=252, 261 | 89.5 (4.65) | 94.1 (5.65)
  Week 40, n=246, 255: number analyzed (Participants) | 246 | 255
  Week 40, n=246, 255 | 90.3 (4.62) | 94.4 (6.09)
  Week 44, n=256, 262: number analyzed (Participants) | 256 | 262
  Week 44, n=256, 262 | 90.7 (5.05) | 94.6 (6.32)
  Week 48, n=243, 260: number analyzed (Participants) | 243 | 260
  Week 48, n=243, 260 | 91.2 (5.21) | 95.4 (6.60)

14. Secondary Outcome: Absolute Values for Hematology Parameters Over Time Including Week 48: Erythrocytes
Description: Blood samples were collected for the analysis of hematology parameters including erythrocytes at indicated timepoints.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^12 cells per Liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
10^12 cells per Liter
  Baseline (Day 1), n=283, 283 | 4.59 (0.434) | 4.65 (0.412)
  Week 4, n=279, 273: number analyzed (Participants) | 279 | 273
  Week 4, n=279, 273 | 4.67 (0.423) | 4.62 (0.406)
  Week 8, n=211, 275: number analyzed (Participants) | 211 | 275
  Week 8, n=211, 275 | 4.76 (0.435) | 4.67 (0.410)
  Week 12, n=270, 275: number analyzed (Participants) | 270 | 275
  Week 12, n=270, 275 | 4.82 (0.435) | 4.66 (0.419)
  Week 16, n=254, 265: number analyzed (Participants) | 254 | 265
  Week 16, n=254, 265 | 4.87 (0.430) | 4.66 (0.407)
  Week 20, n=255, 267: number analyzed (Participants) | 255 | 267
  Week 20, n=255, 267 | 4.89 (0.418) | 4.64 (0.410)
  Week 24, n=259, 264: number analyzed (Participants) | 259 | 264
  Week 24, n=259, 264 | 4.87 (0.418) | 4.67 (0.425)
  Week 28, n=246, 265: number analyzed (Participants) | 246 | 265
  Week 28, n=246, 265 | 4.87 (0.416) | 4.69 (0.395)
  Week 32, n=254, 267: number analyzed (Participants) | 254 | 267
  Week 32, n=254, 267 | 4.83 (0.435) | 4.66 (0.418)
  Week 36, n=252, 261: number analyzed (Participants) | 252 | 261
  Week 36, n=252, 261 | 4.82 (0.403) | 4.64 (0.395)
  Week 40, n=246, 255: number analyzed (Participants) | 246 | 255
  Week 40, n=246, 255 | 4.81 (0.407) | 4.63 (0.409)
  Week 44, n=256, 262: number analyzed (Participants) | 256 | 262
  Week 44, n=256, 262 | 4.79 (0.425) | 4.59 (0.403)
  Week 48, n=243, 260: number analyzed (Participants) | 243 | 260
  Week 48, n=243, 260 | 4.74 (0.443) | 4.59 (0.437)

15. Secondary Outcome: Absolute Values for Hematology Parameters Over Time Including Week 48: Hemoglobin
Description: Blood samples were collected for the analysis of hematology parameter including hemoglobin at indicated timepoints.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Grams per liter
  Baseline (Day 1), n=283, 283 | 142.5 (13.59) | 143.1 (13.51)
  Week 4, n=279, 273: number analyzed (Participants) | 279 | 273
  Week 4, n=279, 273 | 144.3 (13.34) | 143.4 (13.47)
  Week 8, n=211, 275: number analyzed (Participants) | 211 | 275
  Week 8, n=211, 275 | 143.9 (13.84) | 144.7 (13.59)
  Week 12, n=270, 275: number analyzed (Participants) | 270 | 275
  Week 12, n=270, 275 | 144.5 (13.89) | 144.7 (14.66)
  Week 16, n=254, 265: number analyzed (Participants) | 254 | 265
  Week 16, n=254, 265 | 145.3 (13.52) | 144.6 (13.88)
  Week 20, n=255, 267: number analyzed (Participants) | 255 | 267
  Week 20, n=255, 267 | 145.4 (12.69) | 144.8 (13.87)
  Week 24, n=259, 264: number analyzed (Participants) | 259 | 264
  Week 24, n=259, 264 | 145.0 (13.14) | 145.3 (14.07)
  Week 28, n=246, 265: number analyzed (Participants) | 246 | 265
  Week 28, n=246, 265 | 145.3 (12.80) | 146.5 (14.17)
  Week 32, n=254, 267: number analyzed (Participants) | 254 | 267
  Week 32, n=254, 267 | 145.1 (13.37) | 146.2 (14.80)
  Week 36, n=252, 261: number analyzed (Participants) | 252 | 261
  Week 36, n=252, 261 | 144.6 (12.27) | 146.2 (13.85)
  Week 40, n=246, 255: number analyzed (Participants) | 246 | 255
  Week 40, n=246, 255 | 145.9 (12.32) | 146.2 (13.85)
  Week 44, n=256, 262: number analyzed (Participants) | 256 | 262
  Week 44, n=256, 262 | 145.1 (12.79) | 145.0 (14.13)
  Week 48, n=243, 260: number analyzed (Participants) | 243 | 260
  Week 48, n=243, 260 | 143.8 (13.56) | 145.4 (14.56)

16. Secondary Outcome: Absolute Values for Hematology Parameters Over Time Including Week 48: Hematocrit
Description: Blood samples were collected for the analysis of hematology parameters including hematocrit at indicated timepoints.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Proportion of red blood cells in blood
  Baseline (Day 1), n=283, 283 | 0.4341 (0.03889) | 0.4370 (0.03887)
  Week 4, n=279, 273: number analyzed (Participants) | 279 | 273
  Week 4, n=279, 273 | 0.4387 (0.03809) | 0.4363 (0.03832)
  Week 8, n=211, 275: number analyzed (Participants) | 211 | 275
  Week 8, n=211, 275 | 0.4382 (0.04056) | 0.4403 (0.03978)
  Week 12, n=270, 275: number analyzed (Participants) | 270 | 275
  Week 12, n=270, 275 | 0.4377 (0.04020) | 0.4373 (0.04144)
  Week 16, n=254, 265: number analyzed (Participants) | 254 | 265
  Week 16, n=254, 265 | 0.4366 (0.03769) | 0.4371 (0.03890)
  Week 20, n=255, 267: number analyzed (Participants) | 255 | 267
  Week 20, n=255, 267 | 0.4363 (0.03574) | 0.4349 (0.03839)
  Week 24, n=259, 264: number analyzed (Participants) | 259 | 264
  Week 24, n=259, 264 | 0.4351 (0.03580) | 0.4366 (0.03901)
  Week 28, n=246, 265: number analyzed (Participants) | 246 | 265
  Week 28, n=246, 265 | 0.4342 (0.03519) | 0.4374 (0.03867)
  Week 32, n=254, 267: number analyzed (Participants) | 254 | 267
  Week 32, n=254, 267 | 0.4318 (0.03623) | 0.4347 (0.04025)
  Week 36, n=252, 261: number analyzed (Participants) | 252 | 261
  Week 36, n=252, 261 | 0.4301 (0.03392) | 0.4349 (0.03774)
  Week 40, n=246, 255: number analyzed (Participants) | 246 | 255
  Week 40, n=246, 255 | 0.4328 (0.03433) | 0.4358 (0.03845)
  Week 44, n=256, 262: number analyzed (Participants) | 256 | 262
  Week 44, n=256, 262 | 0.4332 (0.03570) | 0.4328 (0.03847)
  Week 48, n=243, 260: number analyzed (Participants) | 243 | 260
  Week 48, n=243, 260 | 0.4310 (0.03875) | 0.4361 (0.04156)

17. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Over Time Including Week 48: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST) and Creatinine Kinase (CK)
Description: Blood samples were collected for the analysis of clinical chemistry parameters including ALT, ALP, AST and CK at indicated timepoints.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
International units per liter
  ALT, Baseline (Day 1), n=283, 283 | 28.7 (125.27) | 19.5 (14.76)
  ALT, Week 4, n=281, 277: number analyzed (Participants) | 281 | 277
  ALT, Week 4, n=281, 277 | 25.1 (64.74) | 17.9 (11.10)
  ALT, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  ALT, Week 8, n=212, 278 | 20.8 (17.43) | 18.4 (11.34)
  ALT, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  ALT, Week 12, n=270, 276 | 21.4 (16.94) | 19.2 (11.29)
  ALT, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  ALT, Week 16, n=255, 269 | 21.6 (17.61) | 20.3 (13.34)
  ALT, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  ALT, Week 20, n=260, 272 | 25.8 (72.51) | 19.6 (15.78)
  ALT, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  ALT, Week 24, n=261, 268 | 23.9 (31.14) | 19.1 (11.91)
  ALT, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  ALT, Week 28, n=253, 268 | 22.5 (19.78) | 19.6 (10.73)
  ALT, Week 32, n=256, 268: number analyzed (Participants) | 256 | 268
  ALT, Week 32, n=256, 268 | 38.5 (293.55) | 19.0 (11.56)
  ALT, Week 36, n=255, 261: number analyzed (Participants) | 255 | 261
  ALT, Week 36, n=255, 261 | 20.3 (13.92) | 21.2 (31.68)
  ALT, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  ALT, Week 40, n=250, 266 | 20.9 (17.32) | 19.5 (12.35)
  ALT, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  ALT, Week 44, n=258, 263 | 22.2 (27.14) | 19.8 (17.43)
  ALT, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  ALT, Week 48, n=247, 262 | 20.1 (21.78) | 19.7 (16.58)
  ALP, Baseline (Day 1), n=283, 283 | 66.5 (22.06) | 67.1 (22.98)
  ALP, Week 4, n=281, 277: number analyzed (Participants) | 281 | 277
  ALP, Week 4, n=281, 277 | 66.2 (19.56) | 65.5 (17.07)
  ALP, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  ALP, Week 8, n=212, 278 | 66.8 (18.82) | 66.3 (17.49)
  ALP, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  ALP, Week 12, n=270, 276 | 66.8 (19.80) | 66.1 (17.23)
  ALP, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  ALP, Week 16, n=255, 269 | 66.7 (19.96) | 66.1 (17.89)
  ALP, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  ALP, Week 20, n=260, 272 | 67.6 (19.11) | 65.6 (16.71)
  ALP, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  ALP, Week 24, n=261, 268 | 67.1 (19.68) | 66.1 (17.96)
  ALP, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  ALP, Week 28, n=253, 268 | 67.4 (20.05) | 67.5 (18.07)
  ALP, Week 32, n=256, 268: number analyzed (Participants) | 256 | 268
  ALP, Week 32, n=256, 268 | 68.0 (22.17) | 66.6 (17.65)
  ALP, Week 36, n=255, 261: number analyzed (Participants) | 255 | 261
  ALP, Week 36, n=255, 261 | 69.5 (26.86) | 68.3 (20.19)
  ALP, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  ALP, Week 40, n=250, 266 | 67.4 (18.94) | 67.7 (18.30)
  ALP, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  ALP, Week 44, n=258, 263 | 67.7 (18.59) | 68.2 (18.62)
  ALP, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  ALP, Week 48, n=247, 262 | 66.4 (17.95) | 67.7 (18.15)
  AST, Baseline (Day 1), n=283, 283 | 28.8 (90.66) | 22.5 (14.80)
  AST, Week 4, n=281, 277: number analyzed (Participants) | 281 | 277
  AST, Week 4, n=281, 277 | 25.1 (32.67) | 20.9 (8.47)
  AST, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  AST, Week 8, n=212, 278 | 23.6 (20.85) | 20.5 (6.26)
  AST, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  AST, Week 12, n=270, 276 | 22.8 (10.38) | 21.0 (8.14)
  AST, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  AST, Week 16, n=255, 269 | 23.0 (10.71) | 22.8 (14.03)
  AST, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  AST, Week 20, n=260, 272 | 25.3 (32.64) | 22.7 (23.48)
  AST, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  AST, Week 24, n=261, 268 | 25.9 (25.16) | 21.2 (9.73)
  AST, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  AST, Week 28, n=253, 268 | 24.8 (16.50) | 21.7 (10.61)
  AST, Week 32, n=256, 268: number analyzed (Participants) | 256 | 268
  AST, Week 32, n=256, 268 | 37.1 (233.23) | 20.7 (6.42)
  AST, Week 36, n=255, 261: number analyzed (Participants) | 255 | 261
  AST, Week 36, n=255, 261 | 23.0 (12.44) | 22.4 (17.37)
  AST, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  AST, Week 40, n=250, 266 | 23.1 (12.22) | 21.0 (6.51)
  AST, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  AST, Week 44, n=258, 263 | 24.4 (15.66) | 21.9 (13.25)
  AST Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  AST Week 48, n=247, 262 | 22.3 (10.98) | 23.5 (42.49)
  CK, Baseline (Day 1), n=283, 283 | 197.8 (291.21) | 199.8 (482.84)
  CK, Week 4, n=280, 277: number analyzed (Participants) | 280 | 277
  CK, Week 4, n=280, 277 | 230.2 (447.94) | 173.0 (220.54)
  CK, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  CK, Week 8, n=212, 278 | 258.0 (928.82) | 152.9 (146.05)
  CK, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  CK, Week 12, n=270, 276 | 201.8 (348.13) | 182.6 (387.61)
  CK, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  CK, Week 16, n=255, 269 | 179.7 (248.71) | 234.0 (576.62)
  CK, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  CK, Week 20, n=260, 272 | 215.7 (539.34) | 258.9 (1109.04)
  CK, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  CK, Week 24, n=261, 268 | 248.6 (628.44) | 183.1 (368.02)
  CK, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  CK, Week 28, n=253, 268 | 252.7 (673.98) | 194.5 (506.24)
  CK, Week 32, n=256, 268: number analyzed (Participants) | 256 | 268
  CK, Week 32, n=256, 268 | 175.8 (223.16) | 160.0 (176.09)
  CK, Week 36, n=254, 261: number analyzed (Participants) | 254 | 261
  CK, Week 36, n=254, 261 | 219.0 (507.30) | 215.2 (460.38)
  CK, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  CK, Week 40, n=250, 266 | 220.5 (507.68) | 149.5 (115.14)
  CK, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  CK, Week 44, n=258, 263 | 254.0 (477.19) | 181.9 (428.28)
  CK, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  CK, Week 48, n=247, 262 | 185.5 (227.54) | 323.6 (2637.27)

18. Secondary Outcome: Absolute Values for Clinical Chemistry Parameter Over Time Including Week 48: Albumin
Description: Blood samples were collected for the analysis of clinical chemistry parameter-albumin at indicated timepoints.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Grams per liter
  Baseline (Day 1), n=283, 283 | 43.8 (3.04) | 44.1 (2.80)
  Week 4, n=280, 277: number analyzed (Participants) | 280 | 277
  Week 4, n=280, 277 | 43.7 (3.03) | 43.8 (2.70)
  Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Week 8, n=212, 278 | 43.5 (2.85) | 43.9 (2.76)
  Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Week 12, n=270, 276 | 43.7 (3.06) | 44.1 (2.87)
  Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  Week 16, n=255, 269 | 44.1 (2.99) | 44.0 (2.78)
  Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  Week 20, n=260, 272 | 44.1 (3.11) | 43.9 (2.72)
  Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  Week 24, n=261, 268 | 44.3 (3.08) | 44.2 (2.60)
  Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Week 28, n=253, 268 | 44.4 (3.09) | 44.5 (2.66)
  Week 32, n=255, 268: number analyzed (Participants) | 255 | 268
  Week 32, n=255, 268 | 44.6 (3.17) | 44.4 (2.76)
  Week 36, n=254, 261: number analyzed (Participants) | 254 | 261
  Week 36, n=254, 261 | 44.1 (3.05) | 44.3 (2.63)
  Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Week 40, n=250, 266 | 44.8 (3.02) | 44.5 (2.76)
  Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Week 44, n=258, 263 | 44.7 (2.98) | 44.4 (2.71)
  Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Week 48, n=247, 262 | 44.6 (2.98) | 44.6 (2.86)

19. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Over Time Including Week 48: Bilirubin, Direct Bilirubin and Creatinine
Description: Blood samples were collected for the analysis of clinical chemistry parameters including bilirubin, creatinine and direct bilirubin at indicated timepoints.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Micromoles per liter
  Bilirubin, Baseline (Day 1), n=283, 283 | 9.3 (5.12) | 9.4 (4.68)
  Bilirubin, Week 4, n=281, 277: number analyzed (Participants) | 281 | 277
  Bilirubin, Week 4, n=281, 277 | 10.7 (6.37) | 8.9 (4.40)
  Bilirubin, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Bilirubin, Week 8, n=212, 278 | 10.1 (4.62) | 8.8 (3.85)
  Bilirubin, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Bilirubin, Week 12, n=270, 276 | 10.5 (5.45) | 8.6 (3.53)
  Bilirubin, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  Bilirubin, Week 16, n=255, 269 | 10.6 (5.49) | 8.7 (3.74)
  Bilirubin, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  Bilirubin, Week 20, n=260, 272 | 10.3 (5.29) | 8.5 (3.40)
  Bilirubin, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  Bilirubin, Week 24, n=261, 268 | 10.0 (5.09) | 8.9 (3.86)
  Bilirubin, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Bilirubin, Week 28, n=253, 268 | 10.4 (5.67) | 8.6 (3.90)
  Bilirubin, Week 32, n=256, 268: number analyzed (Participants) | 256 | 268
  Bilirubin, Week 32, n=256, 268 | 10.5 (7.86) | 8.7 (3.95)
  Bilirubin, Week 36, n=255, 260: number analyzed (Participants) | 255 | 260
  Bilirubin, Week 36, n=255, 260 | 9.9 (6.35) | 8.5 (3.42)
  Bilirubin, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Bilirubin, Week 40, n=250, 266 | 10.2 (5.26) | 8.5 (3.52)
  Bilirubin, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Bilirubin, Week 44, n=258, 263 | 10.3 (5.15) | 8.8 (3.78)
  Bilirubin, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Bilirubin, Week 48, n=247, 262 | 10.3 (5.23) | 8.9 (3.71)
  Direct bilirubin, Baseline (Day 1), n=283, 283 | 2.3 (1.32) | 2.2 (1.09)
  Direct bilirubin, Week 4, n=277, 277: number analyzed (Participants) | 277 | 277
  Direct bilirubin, Week 4, n=277, 277 | 2.4 (1.47) | 2.1 (1.08)
  Direct bilirubin, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Direct bilirubin, Week 8, n=212, 278 | 2.4 (1.17) | 2.1 (0.93)
  Direct bilirubin, Week 12, n=269, 273: number analyzed (Participants) | 269 | 273
  Direct bilirubin, Week 12, n=269, 273 | 2.5 (1.26) | 2.1 (0.91)
  Direct bilirubin, Week 16, n=254, 268: number analyzed (Participants) | 254 | 268
  Direct bilirubin, Week 16, n=254, 268 | 2.4 (1.46) | 2.1 (0.95)
  Direct bilirubin, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  Direct bilirubin, Week 20, n=260, 272 | 2.4 (1.54) | 2.1 (0.90)
  Direct bilirubin, Week 24, n=260, 266: number analyzed (Participants) | 260 | 266
  Direct bilirubin, Week 24, n=260, 266 | 2.3 (1.20) | 2.1 (0.96)
  Direct bilirubin, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Direct bilirubin, Week 28, n=253, 268 | 2.5 (1.29) | 2.1 (0.94)
  Direct bilirubin, Week 32, n=256, 268: number analyzed (Participants) | 256 | 268
  Direct bilirubin, Week 32, n=256, 268 | 2.5 (3.48) | 2.1 (0.94)
  Direct bilirubin, Week 36, n=255, 260: number analyzed (Participants) | 255 | 260
  Direct bilirubin, Week 36, n=255, 260 | 2.4 (2.24) | 2.0 (0.89)
  Direct bilirubin, Week 40, n=249, 266: number analyzed (Participants) | 249 | 266
  Direct bilirubin, Week 40, n=249, 266 | 2.3 (1.29) | 2.1 (0.98)
  Direct bilirubin, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Direct bilirubin, Week 44, n=258, 263 | 2.4 (1.34) | 2.1 (0.95)
  Direct bilirubin, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Direct bilirubin, Week 48, n=247, 262 | 2.3 (1.26) | 2.2 (1.00)
  Creatinine, Baseline (Day 1), n=283, 283 | 89.00 (16.061) | 85.80 (15.660)
  Creatinine, Week 4, n=280, 277: number analyzed (Participants) | 280 | 277
  Creatinine, Week 4, n=280, 277 | 82.99 (15.599) | 86.43 (14.655)
  Creatinine, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Creatinine, Week 8, n=212, 278 | 79.50 (14.103) | 85.50 (15.925)
  Creatinine, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Creatinine, Week 12, n=270, 276 | 79.25 (14.433) | 84.63 (15.155)
  Creatinine, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  Creatinine, Week 16, n=255, 269 | 79.58 (14.509) | 85.18 (14.997)
  Creatinine, Week 20, n=261, 272: number analyzed (Participants) | 261 | 272
  Creatinine, Week 20, n=261, 272 | 78.50 (13.966) | 85.02 (15.488)
  Creatinine, Week 24, n=262, 268: number analyzed (Participants) | 262 | 268
  Creatinine, Week 24, n=262, 268 | 79.10 (15.340) | 85.05 (14.690)
  Creatinine, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Creatinine, Week 28, n=253, 268 | 78.79 (14.741) | 84.38 (15.023)
  Creatinine, Week 32, n=255, 268: number analyzed (Participants) | 255 | 268
  Creatinine, Week 32, n=255, 268 | 78.89 (14.558) | 84.50 (15.047)
  Creatinine, Week 36, n=254, 262: number analyzed (Participants) | 254 | 262
  Creatinine, Week 36, n=254, 262 | 79.58 (14.973) | 84.75 (14.352)
  Creatinine, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Creatinine, Week 40, n=250, 266 | 79.50 (15.615) | 84.70 (14.808)
  Creatinine, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Creatinine, Week 44, n=258, 263 | 80.04 (15.401) | 83.90 (14.604)
  Creatinine, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Creatinine, Week 48, n=247, 262 | 79.95 (15.613) | 90.88 (87.655)

20. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters: Total Carbon-dioxide (CO2), Chloride, Glucose, Phosphate, Potassium, Sodium and Urea Over Time Including Week 48
Description: Blood samples were collected for the analysis of clinical chemistry parameters which includes total CO2, chloride, glucose, phosphate, potassium, sodium and urea at indicated timepoints.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Millimoles per liter
  CO2, Baseline (Day 1), n=283, 283 | 22.4 (2.24) | 22.4 (2.10)
  CO2, Week 4, n=280, 276: number analyzed (Participants) | 280 | 276
  CO2, Week 4, n=280, 276 | 23.0 (2.29) | 22.6 (2.28)
  CO2, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  CO2, Week 8, n=212, 278 | 22.8 (2.07) | 22.3 (2.27)
  CO2, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  CO2, Week 12, n=270, 276 | 22.6 (2.50) | 22.2 (2.34)
  CO2, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  CO2, Week 16, n=255, 269 | 22.9 (2.40) | 22.3 (2.50)
  CO2, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  CO2, Week 20, n=260, 272 | 22.8 (2.30) | 22.4 (2.32)
  CO2, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  CO2, Week 24, n=261, 268 | 23.0 (2.71) | 22.8 (2.19)
  CO2, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  CO2, Week 28, n=253, 268 | 23.0 (2.31) | 22.8 (2.47)
  CO2, Week 32, n=255, 268: number analyzed (Participants) | 255 | 268
  CO2, Week 32, n=255, 268 | 23.0 (2.31) | 22.7 (2.35)
  CO2, Week 36, n=253, 261: number analyzed (Participants) | 253 | 261
  CO2, Week 36, n=253, 261 | 23.1 (2.37) | 22.5 (2.26)
  CO2, Week 40, n=249, 265: number analyzed (Participants) | 249 | 265
  CO2, Week 40, n=249, 265 | 22.8 (2.34) | 22.6 (2.39)
  CO2, Week 44, n=257, 263: number analyzed (Participants) | 257 | 263
  CO2, Week 44, n=257, 263 | 22.9 (2.34) | 22.4 (2.12)
  CO2, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  CO2, Week 48, n=247, 262 | 22.5 (2.18) | 22.3 (2.04)
  Chloride, Baseline (Day 1), n=283, 283 | 104.6 (2.32) | 104.3 (2.32)
  Chloride, Week 4, n=280, 277: number analyzed (Participants) | 280 | 277
  Chloride, Week 4, n=280, 277 | 104.6 (2.22) | 104.7 (2.13)
  Chloride, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Chloride, Week 8, n=212, 278 | 104.7 (1.96) | 104.6 (2.32)
  Chloride, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Chloride, Week 12, n=270, 276 | 104.6 (2.16) | 104.7 (2.35)
  Chloride, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  Chloride, Week 16, n=255, 269 | 104.4 (2.31) | 104.7 (2.24)
  Chloride, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  Chloride, Week 20, n=260, 272 | 104.3 (2.28) | 104.7 (2.06)
  Chloride, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  Chloride, Week 24, n=261, 268 | 104.4 (2.33) | 104.5 (2.42)
  Chloride, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Chloride, Week 28, n=253, 268 | 104.5 (2.20) | 104.5 (2.28)
  Chloride, Week 32, n=255, 268: number analyzed (Participants) | 255 | 268
  Chloride, Week 32, n=255, 268 | 104.4 (2.46) | 104.5 (2.33)
  Chloride, Week 36, n=254, 261: number analyzed (Participants) | 254 | 261
  Chloride, Week 36, n=254, 261 | 104.4 (2.42) | 104.7 (2.20)
  Chloride, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Chloride, Week 40, n=250, 266 | 104.8 (2.55) | 104.7 (2.25)
  Chloride, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Chloride, Week 44, n=258, 263 | 104.7 (2.19) | 105.0 (2.22)
  Chloride, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Chloride, Week 48, n=247, 262 | 104.7 (2.21) | 104.7 (2.28)
  Glucose, Baseline (Day 1), n=283, 283 | 5.21 (1.632) | 5.17 (0.932)
  Glucose, Week 4, n=236, 230: number analyzed (Participants) | 236 | 230
  Glucose, Week 4, n=236, 230 | 5.27 (1.322) | 5.23 (0.734)
  Glucose, Week 8, n=172, 227: number analyzed (Participants) | 172 | 227
  Glucose, Week 8, n=172, 227 | 5.31 (1.347) | 5.19 (0.644)
  Glucose, Week 12, n=229, 216: number analyzed (Participants) | 229 | 216
  Glucose, Week 12, n=229, 216 | 5.26 (0.911) | 5.27 (0.616)
  Glucose, Week 16, n=204, 213: number analyzed (Participants) | 204 | 213
  Glucose, Week 16, n=204, 213 | 5.36 (1.804) | 5.28 (0.801)
  Glucose, Week 20, n=209, 218: number analyzed (Participants) | 209 | 218
  Glucose, Week 20, n=209, 218 | 5.32 (0.735) | 5.26 (0.634)
  Glucose, Week 24, n=221, 214: number analyzed (Participants) | 221 | 214
  Glucose, Week 24, n=221, 214 | 5.35 (1.219) | 5.21 (0.634)
  Glucose, Week 28, n=207, 211: number analyzed (Participants) | 207 | 211
  Glucose, Week 28, n=207, 211 | 5.35 (1.633) | 5.23 (0.614)
  Glucose, Week 32, n=201, 213: number analyzed (Participants) | 201 | 213
  Glucose, Week 32, n=201, 213 | 5.44 (1.355) | 5.27 (0.600)
  Glucose, Week 36, n=199, 204: number analyzed (Participants) | 199 | 204
  Glucose, Week 36, n=199, 204 | 5.35 (0.797) | 5.31 (0.960)
  Glucose, Week 40, n=203, 202: number analyzed (Participants) | 203 | 202
  Glucose, Week 40, n=203, 202 | 5.44 (1.319) | 5.35 (0.753)
  Glucose, Week 44, n=208, 202: number analyzed (Participants) | 208 | 202
  Glucose, Week 44, n=208, 202 | 5.34 (0.991) | 5.35 (0.709)
  Glucose, Week 48, n=248, 251: number analyzed (Participants) | 248 | 251
  Glucose, Week 48, n=248, 251 | 5.22 (0.895) | 5.22 (0.690)
  Phosphate, Baseline (Day 1), n=283, 283 | 1.103 (0.1747) | 1.097 (0.1765)
  Phosphate, Week 4, n=279, 277: number analyzed (Participants) | 279 | 277
  Phosphate, Week 4, n=279, 277 | 1.137 (0.1774) | 1.112 (0.1850)
  Phosphate, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Phosphate, Week 8, n=212, 278 | 1.096 (0.1742) | 1.114 (0.1858)
  Phosphate, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Phosphate, Week 12, n=270, 276 | 1.097 (0.1802) | 1.106 (0.1876)
  Phosphate, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  Phosphate, Week 16, n=255, 269 | 1.104 (0.1806) | 1.119 (0.1823)
  Phosphate, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  Phosphate, Week 20, n=260, 272 | 1.078 (0.1843) | 1.114 (0.1812)
  Phosphate, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  Phosphate, Week 24, n=261, 268 | 1.106 (0.1797) | 1.109 (0.1791)
  Phosphate, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Phosphate, Week 28, n=253, 268 | 1.094 (0.1814) | 1.119 (0.1893)
  Phosphate, Week 32, n=255, 268: number analyzed (Participants) | 255 | 268
  Phosphate, Week 32, n=255, 268 | 1.105 (0.1769) | 1.104 (0.1945)
  Phosphate, Week 36, n=254, 261: number analyzed (Participants) | 254 | 261
  Phosphate, Week 36, n=254, 261 | 1.102 (0.1862) | 1.122 (0.1872)
  Phosphate, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Phosphate, Week 40, n=250, 266 | 1.093 (0.1699) | 1.114 (0.1837)
  Phosphate, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Phosphate, Week 44, n=258, 263 | 1.096 (0.1851) | 1.120 (0.1903)
  Phosphate, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Phosphate, Week 48, n=247, 262 | 1.096 (0.1888) | 1.120 (0.2341)
  Potassium, Baseline (Day 1), n=283, 283 | 4.12 (0.301) | 4.14 (0.288)
  Potassium, Week 4, n=280, 277: number analyzed (Participants) | 280 | 277
  Potassium, Week 4, n=280, 277 | 4.27 (0.308) | 4.20 (0.327)
  Potassium, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Potassium, Week 8, n=212, 278 | 4.22 (0.302) | 4.22 (0.343)
  Potassium, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Potassium, Week 12, n=270, 276 | 4.21 (0.305) | 4.19 (0.282)
  Potassium, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  Potassium, Week 16, n=255, 269 | 4.21 (0.283) | 4.18 (0.303)
  Potassium, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  Potassium, Week 20, n=260, 272 | 4.21 (0.320) | 4.19 (0.313)
  Potassium, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  Potassium, Week 24, n=261, 268 | 4.24 (0.322) | 4.21 (0.312)
  Potassium, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Potassium, Week 28, n=253, 268 | 4.20 (0.298) | 4.23 (0.294)
  Potassium, Week 32, n=255, 268: number analyzed (Participants) | 255 | 268
  Potassium, Week 32, n=255, 268 | 4.21 (0.295) | 4.21 (0.315)
  Potassium, Week 36, n=254, 261: number analyzed (Participants) | 254 | 261
  Potassium, Week 36, n=254, 261 | 4.21 (0.314) | 4.22 (0.314)
  Potassium, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Potassium, Week 40, n=250, 266 | 4.19 (0.301) | 4.20 (0.305)
  Potassium, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Potassium, Week 44, n=258, 263 | 4.21 (0.302) | 4.21 (0.324)
  Potassium, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Potassium, Week 48, n=247, 262 | 4.13 (0.288) | 4.17 (0.449)
  Sodium, Baseline (Day 1), n=283, 283 | 139.2 (1.89) | 139.2 (1.76)
  Sodium, Week 4, n=280, 277: number analyzed (Participants) | 280 | 277
  Sodium, Week 4, n=280, 277 | 139.5 (1.98) | 139.4 (1.83)
  Sodium, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Sodium, Week 8, n=212, 278 | 139.4 (1.78) | 139.3 (1.86)
  Sodium, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Sodium, Week 12, n=270, 276 | 139.5 (1.80) | 139.3 (1.84)
  Sodium, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  Sodium, Week 16, n=255, 269 | 139.4 (1.76) | 139.4 (1.94)
  Sodium, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  Sodium, Week 20, n=260, 272 | 139.4 (1.75) | 139.5 (1.77)
  Sodium, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  Sodium, Week 24, n=261, 268 | 139.3 (1.82) | 139.4 (1.95)
  Sodium, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Sodium, Week 28, n=253, 268 | 139.4 (1.80) | 139.5 (1.83)
  Sodium, Week 32, n=255, 268: number analyzed (Participants) | 255 | 268
  Sodium, Week 32, n=255, 268 | 139.4 (1.83) | 139.4 (1.72)
  Sodium, Week 36, n=254, 261: number analyzed (Participants) | 254 | 261
  Sodium, Week 36, n=254, 261 | 139.3 (1.87) | 139.5 (1.70)
  Sodium, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Sodium, Week 40, n=250, 266 | 139.3 (2.04) | 139.5 (1.84)
  Sodium, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Sodium, Week 44, n=258, 263 | 139.5 (1.95) | 139.6 (1.79)
  Sodium, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Sodium, Week 48, n=247, 262 | 139.4 (1.68) | 139.5 (1.75)
  Urea, Baseline (Day 1), n=283, 283 | 5.30 (1.468) | 5.17 (1.458)
  Urea, Week 4, n=280, 277: number analyzed (Participants) | 280 | 277
  Urea, Week 4, n=280, 277 | 5.33 (1.424) | 5.14 (1.508)
  Urea, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Urea, Week 8, n=212, 278 | 5.32 (1.485) | 5.12 (1.480)
  Urea, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Urea, Week 12, n=270, 276 | 5.28 (1.424) | 5.20 (1.574)
  Urea, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  Urea, Week 16, n=255, 269 | 5.26 (1.385) | 5.20 (1.561)
  Urea, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  Urea, Week 20, n=260, 272 | 5.18 (1.349) | 5.22 (1.483)
  Urea, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  Urea, Week 24, n=261, 268 | 5.38 (1.489) | 5.11 (1.449)
  Urea, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Urea, Week 28, n=253, 268 | 5.32 (1.422) | 5.21 (1.406)
  Urea, Week 32, n=255, 268: number analyzed (Participants) | 255 | 268
  Urea, Week 32, n=255, 268 | 5.43 (1.440) | 5.17 (1.491)
  Urea, Week 36, n=254, 261: number analyzed (Participants) | 254 | 261
  Urea, Week 36, n=254, 261 | 5.31 (1.396) | 5.23 (1.556)
  Urea, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Urea, Week 40, n=250, 266 | 5.40 (1.523) | 5.26 (1.566)
  Urea, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Urea, Week 44, n=258, 263 | 5.38 (1.543) | 5.24 (1.512)
  Urea, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Urea, Week 48, n=247, 262 | 5.37 (1.402) | 5.27 (2.305)

21. Secondary Outcome: Absolute Values for Clinical Chemistry Parameter Over Time Including Week 48: Lipase
Description: Blood samples were collected for the analysis of clinical chemistry parameter-lipase at indicated timepoints.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Units per liter
  Baseline (Day 1), n=283, 283 | 31.0 (21.04) | 30.9 (28.89)
  Week 4, n=278, 276: number analyzed (Participants) | 278 | 276
  Week 4, n=278, 276 | 31.7 (27.17) | 32.6 (24.73)
  Week 8, n=211, 278: number analyzed (Participants) | 211 | 278
  Week 8, n=211, 278 | 31.5 (21.15) | 31.3 (19.96)
  Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Week 12, n=270, 276 | 31.4 (23.94) | 33.6 (23.37)
  Week 16, n=254, 269: number analyzed (Participants) | 254 | 269
  Week 16, n=254, 269 | 30.8 (22.39) | 32.1 (18.99)
  Week 20, n=260, 270: number analyzed (Participants) | 260 | 270
  Week 20, n=260, 270 | 31.3 (23.46) | 31.9 (19.13)
  Week 24, n=260, 268: number analyzed (Participants) | 260 | 268
  Week 24, n=260, 268 | 31.3 (22.60) | 32.2 (21.08)
  Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Week 28, n=253, 268 | 30.3 (18.71) | 33.0 (22.56)
  Week 32, n=254, 268: number analyzed (Participants) | 254 | 268
  Week 32, n=254, 268 | 33.5 (35.38) | 33.2 (32.95)
  Week 36, n=254, 261: number analyzed (Participants) | 254 | 261
  Week 36, n=254, 261 | 31.5 (20.49) | 31.2 (20.03)
  Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Week 40, n=250, 266 | 32.6 (27.07) | 32.1 (22.19)
  Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Week 44, n=258, 263 | 36.3 (45.04) | 33.0 (24.09)
  Week 48, n=247, 261: number analyzed (Participants) | 247 | 261
  Week 48, n=247, 261 | 30.1 (20.31) | 32.6 (28.96)

22. Secondary Outcome: Absolute Values for Clinical Chemistry Parameter Over Time Including Week 48: Creatinine Clearance.
Description: Blood samples were collected for the analysis of clinical chemistry parameter-creatinine clearance at indicated timepoints. Glomerular filtration rate (GFR) will be estimated by the central laboratory using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI).
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mL/min/1.73/m^2
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
mL/min/1.73/m^2
  Baseline (Day 1), n=283, 283 | 94.3 (17.61) | 97.9 (17.70)
  Week 4, n=278, 277: number analyzed (Participants) | 278 | 277
  Week 4, n=278, 277 | 101.2 (16.56) | 96.5 (17.14)
  Week 8, n=211, 278: number analyzed (Participants) | 211 | 278
  Week 8, n=211, 278 | 104.9 (15.64) | 98.1 (17.46)
  Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Week 12, n=270, 276 | 104.8 (16.08) | 98.6 (17.77)
  Week 16, n=254, 269: number analyzed (Participants) | 254 | 269
  Week 16, n=254, 269 | 104.2 (15.03) | 97.6 (16.84)
  Week 20, n=261, 271: number analyzed (Participants) | 261 | 271
  Week 20, n=261, 271 | 105.5 (15.19) | 98.0 (17.67)
  Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  Week 24, n=261, 268 | 105.1 (16.05) | 97.9 (17.33)
  Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Week 28, n=253, 268 | 105.3 (16.18) | 98.8 (17.40)
  Week 32, n=254, 268: number analyzed (Participants) | 254 | 268
  Week 32, n=254, 268 | 105.1 (16.10) | 98.8 (17.39)
  Week 36, n=254, 262: number analyzed (Participants) | 254 | 262
  Week 36, n=254, 262 | 104.7 (15.88) | 98.0 (16.60)
  Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Week 40, n=250, 266 | 104.3 (16.47) | 98.3 (17.25)
  Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Week 44, n=258, 263 | 104.4 (16.73) | 98.9 (16.67)
  Week 48, n=247, 261: number analyzed (Participants) | 247 | 261
  Week 48, n=247, 261 | 103.6 (16.34) | 96.9 (18.21)

23. Secondary Outcome: Absolute Values for Fasting Lipid Panel Overtime Including Week 48
Description: Blood samples were collected at Baseline and at Week 48 to assess fasting lipids which included total cholesterol, high density lipoprotein (HDL)cholesterol, low density lipoprotein (LDL) cholesterol and triglycerides.
Time Frame: Baseline (Day 1) and at Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Millimoles per liter
  Total Cholesterol, Baseline (Day 1), n=268, 275: number analyzed (Participants) | 268 | 275
  Total Cholesterol, Baseline (Day 1), n=268, 275 | 4.44 (0.928) | 4.42 (0.986)
  Total Cholesterol, Week 48, n=240, 239: number analyzed (Participants) | 240 | 239
  Total Cholesterol, Week 48, n=240, 239 | 4.65 (1.021) | 4.46 (0.944)
  HDL cholesterol, Baseline (Day 1), n=268, 275: number analyzed (Participants) | 268 | 275
  HDL cholesterol, Baseline (Day 1), n=268, 275 | 1.249 (0.3761) | 1.302 (0.3851)
  HDL cholesterol, Week 48, n=240, 239: number analyzed (Participants) | 240 | 239
  HDL cholesterol, Week 48, n=240, 239 | 1.359 (0.4096) | 1.376 (0.4335)
  LDL cholesterol, Baseline (Day 1), n=267, 275: number analyzed (Participants) | 267 | 275
  LDL cholesterol, Baseline (Day 1), n=267, 275 | 2.557 (0.7991) | 2.529 (0.7870)
  LDL cholesterol, Week 48, n=238, 237: number analyzed (Participants) | 238 | 237
  LDL cholesterol, Week 48, n=238, 237 | 2.697 (0.9158) | 2.472 (0.7693)
  Triglycerides, Baseline (Day 1), n=268, 275: number analyzed (Participants) | 268 | 275
  Triglycerides, Baseline (Day 1), n=268, 275 | 1.387 (0.9142) | 1.294 (0.7392)
  Triglycerides, Week 48, n=240, 239: number analyzed (Participants) | 240 | 239
  Triglycerides, Week 48, n=240, 239 | 1.323 (0.9333) | 1.341 (0.9059)

24. Secondary Outcome: Number of Participants With Abnormal Urinalysis Parameter Over Time Including Week 48
Description: The dipstick test gives results in a semi-quantitative manner and results for urinalysis parameters (ketones, glucose, bilirubin, occult blood, nitrite and blood protein) can be read as positive, trace, 1+, 2+, 3+ and 4+ indicating proportional concentrations in the urine sample. The urine parameters were graded according to DAIDS scale where Grade 1 indicates mild (trace to 1+), Grade 2 indicates moderate (2+) and Grade 3 indicates severe (3+ or higher). Only participants with abnormal findings for urinalysis at any visit has been presented.
Time Frame: Baseline (Day 1) and at Weeks 4, 24 and 48
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Participants
  Urine bilirubin,Baseline (Day 1),Trace, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine bilirubin,Baseline (Day 1),Trace, n=276, 276 | 0 | 0
  Urine bilirubin, Baseline (Day 1), 1+, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine bilirubin, Baseline (Day 1), 1+, n=276, 276 | 15 | 22
  Urine bilirubin, Baseline (Day 1), 2+, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine bilirubin, Baseline (Day 1), 2+, n=276, 276 | 0 | 1
  Urine bilirubin, Baseline (Day 1), 3+, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine bilirubin, Baseline (Day 1), 3+, n=276, 276 | 0 | 0
  Urine glucose, Baseline (Day 1), Trace, n=282, 282: number analyzed (Participants) | 282 | 282
  Urine glucose, Baseline (Day 1), Trace, n=282, 282 | 0 | 1
  Urine glucose, Baseline (Day 1), 1+, n=282, 282: number analyzed (Participants) | 282 | 282
  Urine glucose, Baseline (Day 1), 1+, n=282, 282 | 2 | 0
  Urine glucose, Baseline (Day 1), 2+, n=282, 282: number analyzed (Participants) | 282 | 282
  Urine glucose, Baseline (Day 1), 2+, n=282, 282 | 0 | 0
  Urine glucose, Baseline (Day 1), 3+, n=282, 282: number analyzed (Participants) | 282 | 282
  Urine glucose, Baseline (Day 1), 3+, n=282, 282 | 1 | 1
  Urine ketones, Baseline (Day 1), Trace, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine ketones, Baseline (Day 1), Trace, n=276, 276 | 30 | 29
  Urine ketones, Baseline (Day 1), 1+, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine ketones, Baseline (Day 1), 1+, n=276, 276 | 4 | 2
  Urine ketones, Baseline (Day 1), 2+, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine ketones, Baseline (Day 1), 2+, n=276, 276 | 0 | 1
  Urine ketones, Baseline (Day 1), 3+, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine ketones, Baseline (Day 1), 3+, n=276, 276 | 0 | 0
  Urine leukocyte esterase,Baseline,Trace,n=276, 276: number analyzed (Participants) | 276 | 276
  Urine leukocyte esterase,Baseline,Trace,n=276, 276 | 22 | 21
  Urine leukocyte esterase, Baseline, 1+, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine leukocyte esterase, Baseline, 1+, n=276, 276 | 12 | 14
  Urine leukocyte esterase, Baseline, 2+, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine leukocyte esterase, Baseline, 2+, n=276, 276 | 9 | 9
  Urine leukocyte esterase, Baseline, 3+, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine leukocyte esterase, Baseline, 3+, n=276, 276 | 3 | 3
  Urine nitrite, Baseline, positive, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine nitrite, Baseline, positive, n=276, 276 | 6 | 9
  Urine occult blood, Baseline, Trace, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine occult blood, Baseline, Trace, n=276, 276 | 13 | 9
  Urine occult blood, Baseline, 1+, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine occult blood, Baseline, 1+, n=276, 276 | 5 | 6
  Urine occult blood, Baseline, 2+, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine occult blood, Baseline, 2+, n=276, 276 | 6 | 3
  Urine occult blood, Baseline, 3+, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine occult blood, Baseline, 3+, n=276, 276 | 3 | 2
  Urine protein, Baseline, Trace, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine protein, Baseline, Trace, n=276, 276 | 25 | 20
  Urine protein, Baseline, 1+, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine protein, Baseline, 1+, n=276, 276 | 4 | 10
  Urine protein, Baseline, 2+, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine protein, Baseline, 2+, n=276, 276 | 3 | 7
  Urine protein, Baseline, 3+, n=276, 276: number analyzed (Participants) | 276 | 276
  Urine protein, Baseline, 3+, n=276, 276 | 0 | 0
  Urine bilirubin, Week 4, Trace, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine bilirubin, Week 4, Trace, n=278, 272 | 0 | 0
  Urine bilirubin, Week 4, 1+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine bilirubin, Week 4, 1+, n=278, 272 | 14 | 28
  Urine bilirubin, Week 4, 2+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine bilirubin, Week 4, 2+, n=278, 272 | 0 | 0
  Urine bilirubin, Week 4, 3+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine bilirubin, Week 4, 3+, n=278, 272 | 0 | 0
  Urine glucose, Week 4, Trace, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine glucose, Week 4, Trace, n=278, 272 | 0 | 0
  Urine glucose, Week 4, 1+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine glucose, Week 4, 1+, n=278, 272 | 0 | 2
  Urine glucose, Week 4, 2+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine glucose, Week 4, 2+, n=278, 272 | 0 | 0
  Urine glucose, Week 4, 3+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine glucose, Week 4, 3+, n=278, 272 | 1 | 0
  Urine ketones, Week 4, Trace, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine ketones, Week 4, Trace, n=278, 272 | 20 | 21
  Urine ketones, Week 4, 1+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine ketones, Week 4, 1+, n=278, 272 | 1 | 5
  Urine ketones, Week 4, 2+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine ketones, Week 4, 2+, n=278, 272 | 0 | 0
  Urine ketones, Week 4, 3+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine ketones, Week 4, 3+, n=278, 272 | 1 | 0
  Urine leukocyte esterase, Week 4, Trace,n=278, 272: number analyzed (Participants) | 278 | 272
  Urine leukocyte esterase, Week 4, Trace,n=278, 272 | 19 | 23
  Urine leukocyte esterase, Week 4, 1+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine leukocyte esterase, Week 4, 1+, n=278, 272 | 9 | 17
  Urine leukocyte esterase, Week 4, 2+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine leukocyte esterase, Week 4, 2+, n=278, 272 | 6 | 6
  Urine leukocyte esterase, Week 4, 3+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine leukocyte esterase, Week 4, 3+, n=278, 272 | 2 | 4
  Urine nitrite, Week 4, positive, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine nitrite, Week 4, positive, n=278, 272 | 2 | 10
  Urine occult blood, Week 4, Trace, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine occult blood, Week 4, Trace, n=278, 272 | 11 | 13
  Urine occult blood, Week 4, 1+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine occult blood, Week 4, 1+, n=278, 272 | 8 | 3
  Urine occult blood, Week 4, 2+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine occult blood, Week 4, 2+, n=278, 272 | 5 | 1
  Urine occult blood, Week 4, 3+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine occult blood, Week 4, 3+, n=278, 272 | 0 | 6
  Urine protein, Week 4, Trace, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine protein, Week 4, Trace, n=278, 272 | 12 | 24
  Urine protein, Week 4, 1+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine protein, Week 4, 1+, n=278, 272 | 4 | 11
  Urine protein, Week 4, 2+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine protein, Week 4, 2+, n=278, 272 | 1 | 3
  Urine protein, Week 4, 3+, n=278, 272: number analyzed (Participants) | 278 | 272
  Urine protein, Week 4, 3+, n=278, 272 | 1 | 1
  Urine bilirubin, Week 24, Trace, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine bilirubin, Week 24, Trace, n=195, 258 | 0 | 0
  Urine bilirubin, Week 24, 1+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine bilirubin, Week 24, 1+, n=195, 258 | 7 | 14
  , Urine bilirubin, Week 24, 2+, n=195, 258: number analyzed (Participants) | 195 | 258
  , Urine bilirubin, Week 24, 2+, n=195, 258 | 0 | 0
  Urine bilirubin, Week 24, 3+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine bilirubin, Week 24, 3+, n=195, 258 | 0 | 0
  Urine glucose, Week 24, Trace, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine glucose, Week 24, Trace, n=195, 258 | 0 | 0
  Urine glucose, Week 24, 1+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine glucose, Week 24, 1+, n=195, 258 | 0 | 0
  Urine glucose, Week 24, 2+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine glucose, Week 24, 2+, n=195, 258 | 1 | 0
  Urine glucose, Week 24, 3+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine glucose, Week 24, 3+, n=195, 258 | 1 | 1
  Urine ketones, Week 24, Trace, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine ketones, Week 24, Trace, n=195, 258 | 13 | 9
  Urine ketones, Week 24, 1+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine ketones, Week 24, 1+, n=195, 258 | 0 | 2
  Urine ketones, Week 24, 2+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine ketones, Week 24, 2+, n=195, 258 | 0 | 0
  Urine ketones, Week 24, 3+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine ketones, Week 24, 3+, n=195, 258 | 0 | 0
  Urine leukocyte esterase,Week 24, Trace,n=195, 258: number analyzed (Participants) | 195 | 258
  Urine leukocyte esterase,Week 24, Trace,n=195, 258 | 15 | 28
  Urine leukocyte esterase, Week 24, 1+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine leukocyte esterase, Week 24, 1+, n=195, 258 | 8 | 12
  Urine leukocyte esterase, Week 24, 2+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine leukocyte esterase, Week 24, 2+, n=195, 258 | 3 | 10
  Urine leukocyte esterase, Week 24, 3+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine leukocyte esterase, Week 24, 3+, n=195, 258 | 1 | 3
  Urine nitrite, Week 24, positive, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine nitrite, Week 24, positive, n=195, 258 | 4 | 5
  Urine occult blood, Week 24, Trace, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine occult blood, Week 24, Trace, n=195, 258 | 9 | 9
  Urine occult blood, Week 24, 1+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine occult blood, Week 24, 1+, n=195, 258 | 3 | 8
  Urine occult blood, Week 24, 2+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine occult blood, Week 24, 2+, n=195, 258 | 3 | 2
  Urine occult blood, Week 24, 3+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine occult blood, Week 24, 3+, n=195, 258 | 1 | 3
  Urine protein, Week 24, Trace, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine protein, Week 24, Trace, n=195, 258 | 11 | 21
  Urine protein, Week 24, 1+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine protein, Week 24, 1+, n=195, 258 | 4 | 7
  Urine protein, Week 24, 2+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine protein, Week 24, 2+, n=195, 258 | 2 | 4
  Urine protein, Week 24, 3+, n=195, 258: number analyzed (Participants) | 195 | 258
  Urine protein, Week 24, 3+, n=195, 258 | 0 | 1
  Urine bilirubin, Week 48, Trace, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine bilirubin, Week 48, Trace, n=261, 259 | 0 | 0
  Urine bilirubin, Week 48, 1+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine bilirubin, Week 48, 1+, n=261, 259 | 9 | 12
  Urine bilirubin, Week 48, 2+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine bilirubin, Week 48, 2+, n=261, 259 | 0 | 0
  Urine bilirubin, Week 48, 3+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine bilirubin, Week 48, 3+, n=261, 259 | 0 | 1
  Urine glucose, Week 48, Trace, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine glucose, Week 48, Trace, n=261, 259 | 0 | 0
  Urine glucose, Week 48, 1+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine glucose, Week 48, 1+, n=261, 259 | 1 | 0
  Urine glucose, Week 48, 2+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine glucose, Week 48, 2+, n=261, 259 | 0 | 0
  Urine glucose, Week 48, 3+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine glucose, Week 48, 3+, n=261, 259 | 2 | 0
  Urine ketones, Week 48, Trace, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine ketones, Week 48, Trace, n=261, 259 | 12 | 13
  Urine ketones, Week 48, 1+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine ketones, Week 48, 1+, n=261, 259 | 0 | 4
  Urine ketones, Week 48, 2+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine ketones, Week 48, 2+, n=261, 259 | 0 | 0
  Urine ketones, Week 48, 3+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine ketones, Week 48, 3+, n=261, 259 | 0 | 0
  Urine leukocyte esterase, Week 48,Trace,n=261, 259: number analyzed (Participants) | 261 | 259
  Urine leukocyte esterase, Week 48,Trace,n=261, 259 | 12 | 15
  Urine leukocyte esterase, Week 48, 1+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine leukocyte esterase, Week 48, 1+, n=261, 259 | 5 | 10
  Urine leukocyte esterase, Week 48, 2+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine leukocyte esterase, Week 48, 2+, n=261, 259 | 4 | 7
  Urine leukocyte esterase, Week 48, 3+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine leukocyte esterase, Week 48, 3+, n=261, 259 | 2 | 2
  Urine nitrite, Week 48, positive, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine nitrite, Week 48, positive, n=261, 259 | 2 | 6
  Urine occult blood, Week 48, Trace, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine occult blood, Week 48, Trace, n=261, 259 | 9 | 8
  Urine occult blood, Week 48, 1+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine occult blood, Week 48, 1+, n=261, 259 | 4 | 6
  Urine occult blood, Week 48, 2+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine occult blood, Week 48, 2+, n=261, 259 | 8 | 3
  Urine occult blood, Week 48, 3+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine occult blood, Week 48, 3+, n=261, 259 | 1 | 0
  Urine protein, Week 48, Trace, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine protein, Week 48, Trace, n=261, 259 | 14 | 23
  Urine protein, Week 48, 1+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine protein, Week 48, 1+, n=261, 259 | 5 | 8
  Urine protein, Week 48, 2+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine protein, Week 48, 2+, n=261, 259 | 6 | 6
  Urine protein, Week 48, 3+, n=261, 259: number analyzed (Participants) | 261 | 259
  Urine protein, Week 48, 3+, n=261, 259 | 0 | 0

25. Secondary Outcome: Number of Participants With Urine Potential of Hydrogen (pH) Over Time Including Week 48
Description: Urine samples were collected for analysis of urine pH. pH is calculated on a scale of 0 to 14, values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH of less than 7 is acidic and a pH of greater than 7 is basic. Normal urine has a slightly acidic pH (5.0-6.0).
Time Frame: Baseline (Day 1) and at Weeks 4, 24 and 48
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Participants
  Baseline (Day 1), pH=5, n=276, 276: number analyzed (Participants) | 276 | 276
  Baseline (Day 1), pH=5, n=276, 276 | 36 | 32
  Baseline (Day 1), pH=5.5, n=276, 276: number analyzed (Participants) | 276 | 276
  Baseline (Day 1), pH=5.5, n=276, 276 | 104 | 101
  Baseline (Day 1), pH=6, n=276, 276: number analyzed (Participants) | 276 | 276
  Baseline (Day 1), pH=6, n=276, 276 | 66 | 62
  Baseline (Day 1), pH=6.5, n=276, 276: number analyzed (Participants) | 276 | 276
  Baseline (Day 1), pH=6.5, n=276, 276 | 29 | 35
  Baseline (Day 1), pH=7, n=276, 276: number analyzed (Participants) | 276 | 276
  Baseline (Day 1), pH=7, n=276, 276 | 27 | 27
  Baseline (Day 1), pH=7.5, n=276, 276: number analyzed (Participants) | 276 | 276
  Baseline (Day 1), pH=7.5, n=276, 276 | 7 | 12
  Baseline (Day 1), pH=8, n=276, 276: number analyzed (Participants) | 276 | 276
  Baseline (Day 1), pH=8, n=276, 276 | 4 | 4
  Baseline (Day 1), pH=8.5, n=276, 276: number analyzed (Participants) | 276 | 276
  Baseline (Day 1), pH=8.5, n=276, 276 | 2 | 1
  Baseline (Day 1), pH>9.0, n=276, 276: number analyzed (Participants) | 276 | 276
  Baseline (Day 1), pH>9.0, n=276, 276 | 1 | 2
  Week 4, pH=5, n=278, 272: number analyzed (Participants) | 278 | 272
  Week 4, pH=5, n=278, 272 | 33 | 41
  Week 4, pH=5.5, n=278, 272: number analyzed (Participants) | 278 | 272
  Week 4, pH=5.5, n=278, 272 | 83 | 81
  Week 4, pH=6, n=278, 272: number analyzed (Participants) | 278 | 272
  Week 4, pH=6, n=278, 272 | 68 | 71
  Week 4, pH=6.5, n=278, 272: number analyzed (Participants) | 278 | 272
  Week 4, pH=6.5, n=278, 272 | 48 | 36
  Week 4, pH=7, n=278, 272: number analyzed (Participants) | 278 | 272
  Week 4, pH=7, n=278, 272 | 25 | 22
  Week 4, pH=7.5, n=278, 272: number analyzed (Participants) | 278 | 272
  Week 4, pH=7.5, n=278, 272 | 10 | 12
  Week 4, pH=8, n=278, 272: number analyzed (Participants) | 278 | 272
  Week 4, pH=8, n=278, 272 | 5 | 5
  Week 4, pH=8.5, n=278, 272: number analyzed (Participants) | 278 | 272
  Week 4, pH=8.5, n=278, 272 | 6 | 1
  Week 4, pH>9.0, n=278, 272: number analyzed (Participants) | 278 | 272
  Week 4, pH>9.0, n=278, 272 | 0 | 3
  Week 24, pH=5, n=195, 258: number analyzed (Participants) | 195 | 258
  Week 24, pH=5, n=195, 258 | 42 | 50
  Week 24, pH=5.5, n=195, 258: number analyzed (Participants) | 195 | 258
  Week 24, pH=5.5, n=195, 258 | 55 | 78
  Week 24, pH=6, n=195, 258: number analyzed (Participants) | 195 | 258
  Week 24, pH=6, n=195, 258 | 47 | 51
  Week 24, pH=6.5, n=195, 258: number analyzed (Participants) | 195 | 258
  Week 24, pH=6.5, n=195, 258 | 19 | 46
  Week 24, pH=7, n=195, 258: number analyzed (Participants) | 195 | 258
  Week 24, pH=7, n=195, 258 | 22 | 16
  Week 24, pH=7.5, n=195, 258: number analyzed (Participants) | 195 | 258
  Week 24, pH=7.5, n=195, 258 | 4 | 13
  Week 24, pH=8, n=195, 258: number analyzed (Participants) | 195 | 258
  Week 24, pH=8, n=195, 258 | 3 | 2
  Week 24, pH=8.5, n=195, 258: number analyzed (Participants) | 195 | 258
  Week 24, pH=8.5, n=195, 258 | 3 | 1
  Week 24, pH>9.0, n=195, 258: number analyzed (Participants) | 195 | 258
  Week 24, pH>9.0, n=195, 258 | 0 | 1
  Week 48, pH=5, n=261, 259: number analyzed (Participants) | 261 | 259
  Week 48, pH=5, n=261, 259 | 54 | 57
  Week 48, pH=5.5, n=261, 259: number analyzed (Participants) | 261 | 259
  Week 48, pH=5.5, n=261, 259 | 81 | 77
  Week 48, pH=6, n=261, 259: number analyzed (Participants) | 261 | 259
  Week 48, pH=6, n=261, 259 | 50 | 61
  Week 48, pH=6.5, n=261, 259: number analyzed (Participants) | 261 | 259
  Week 48, pH=6.5, n=261, 259 | 30 | 27
  Week 48, pH=7, n=261, 259: number analyzed (Participants) | 261 | 259
  Week 48, pH=7, n=261, 259 | 24 | 18
  Week 48, pH=7.5, n=261, 259: number analyzed (Participants) | 261 | 259
  Week 48, pH=7.5, n=261, 259 | 14 | 10
  Week 48, pH=8, n=261, 259: number analyzed (Participants) | 261 | 259
  Week 48, pH=8, n=261, 259 | 5 | 4
  Week 48, pH=8.5, n=261, 259: number analyzed (Participants) | 261 | 259
  Week 48, pH=8.5, n=261, 259 | 2 | 3
  Week 48, pH>9.0, n=261, 259: number analyzed (Participants) | 261 | 259
  Week 48, pH>9.0, n=261, 259 | 1 | 2

26. Secondary Outcome: Change From Baseline for Hematology Parameters: Basophil, Eosinophils, Leukocytes, Lymphocytes, Neutrophils, Monocytes, and Platelets
Description: Blood samples were collected for the analysis of hematology parameters including basophil, eosinophils, leukocytes, lymphocytes, neutrophils, monocytes, and platelets at indicated timepoints. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance Phase dose of IP. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^9 cells per Liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
10^9 cells per Liter
  Basophils, Week 4, n=277, 270: number analyzed (Participants) | 277 | 270
  Basophils, Week 4, n=277, 270 | 0.002 (0.0155) | 0.002 (0.0155)
  Basophils, Week 8, n=210, 272: number analyzed (Participants) | 210 | 272
  Basophils, Week 8, n=210, 272 | 0.002 (0.0161) | 0.001 (0.0153)
  Basophils, Week 12, n=267, 272: number analyzed (Participants) | 267 | 272
  Basophils, Week 12, n=267, 272 | 0.003 (0.0181) | 0.001 (0.0157)
  Basophils, Week 16, n=247, 259: number analyzed (Participants) | 247 | 259
  Basophils, Week 16, n=247, 259 | 0.008 (0.0215) | 0.006 (0.0227)
  Basophils, Week 20, n=247, 259: number analyzed (Participants) | 247 | 259
  Basophils, Week 20, n=247, 259 | 0.013 (0.0250) | 0.010 (0.0271)
  Basophils, Week 24, n=256, 260: number analyzed (Participants) | 256 | 260
  Basophils, Week 24, n=256, 260 | 0.015 (0.0247) | 0.014 (0.0269)
  Basophils, Week 28, n=239, 258: number analyzed (Participants) | 239 | 258
  Basophils, Week 28, n=239, 258 | 0.017 (0.0265) | 0.016 (0.0251)
  Basophils, Week 32, n=246, 263: number analyzed (Participants) | 246 | 263
  Basophils, Week 32, n=246, 263 | 0.022 (0.0266) | 0.017 (0.0227)
  Basophils, Week 36, n=250, 259: number analyzed (Participants) | 250 | 259
  Basophils, Week 36, n=250, 259 | 0.021 (0.0235) | 0.018 (0.0249)
  Basophils, Week 40, n=244, 245: number analyzed (Participants) | 244 | 245
  Basophils, Week 40, n=244, 245 | 0.020 (0.0252) | 0.019 (0.0243)
  Basophils, Week 44, n=249, 260: number analyzed (Participants) | 249 | 260
  Basophils, Week 44, n=249, 260 | 0.018 (0.0246) | 0.018 (0.0265)
  Basophils, Week 48, n=239, 258: number analyzed (Participants) | 239 | 258
  Basophils, Week 48, n=239, 258 | 0.016 (0.0218) | 0.016 (0.0243)
  Eosinophils, Week 4, n=277, 270: number analyzed (Participants) | 277 | 270
  Eosinophils, Week 4, n=277, 270 | 0.024 (0.1099) | 0.013 (0.1220)
  Eosinophils, Week 8, n=210, 272: number analyzed (Participants) | 210 | 272
  Eosinophils, Week 8, n=210, 272 | 0.023 (0.1101) | 0.009 (0.1075)
  Eosinophils, Week 12, n=267, 272: number analyzed (Participants) | 267 | 272
  Eosinophils, Week 12, n=267, 272 | 0.023 (0.1305) | 0.018 (0.1082)
  Eosinophils, Week 16, n=247, 259: number analyzed (Participants) | 247 | 259
  Eosinophils, Week 16, n=247, 259 | 0.037 (0.1425) | 0.022 (0.1262)
  Eosinophils, Week 20, n=247, 259: number analyzed (Participants) | 247 | 259
  Eosinophils, Week 20, n=247, 259 | 0.044 (0.1478) | 0.027 (0.1288)
  Eosinophils, Week 24, n=256, 260: number analyzed (Participants) | 256 | 260
  Eosinophils, Week 24, n=256, 260 | 0.051 (0.1307) | 0.030 (0.1124)
  Eosinophils, Week 28, n=239, 258: number analyzed (Participants) | 239 | 258
  Eosinophils, Week 28, n=239, 258 | 0.061 (0.1367) | 0.037 (0.1393)
  Eosinophils, Week 32, n=246, 263: number analyzed (Participants) | 246 | 263
  Eosinophils, Week 32, n=246, 263 | 0.061 (0.1556) | 0.029 (0.1158)
  Eosinophils, Week 36, n=250, 259: number analyzed (Participants) | 250 | 259
  Eosinophils, Week 36, n=250, 259 | 0.070 (0.1797) | 0.030 (0.1303)
  Eosinophils, Week 40, n=244, 245: number analyzed (Participants) | 244 | 245
  Eosinophils, Week 40, n=244, 245 | 0.062 (0.1623) | 0.035 (0.1155)
  Eosinophils, Week 44, n=249, 260: number analyzed (Participants) | 249 | 260
  Eosinophils, Week 44, n=249, 260 | 0.057 (0.1598) | 0.038 (0.1410)
  Eosinophils, Week 48, n=239, 258: number analyzed (Participants) | 239 | 258
  Eosinophils, Week 48, n=239, 258 | 0.039 (0.1416) | 0.030 (0.1183)
  Leukocytes, Week 4, n=279, 272: number analyzed (Participants) | 279 | 272
  Leukocytes, Week 4, n=279, 272 | 0.57 (1.404) | 0.42 (1.383)
  Leukocytes, Week 8, n=211, 275: number analyzed (Participants) | 211 | 275
  Leukocytes, Week 8, n=211, 275 | 0.18 (1.278) | 0.32 (1.374)
  Leukocytes, Week 12, n=270, 275: number analyzed (Participants) | 270 | 275
  Leukocytes, Week 12, n=270, 275 | 0.07 (1.402) | 0.40 (1.465)
  Leukocytes, Week 16, n=252, 265: number analyzed (Participants) | 252 | 265
  Leukocytes, Week 16, n=252, 265 | 0.32 (1.641) | 0.41 (1.621)
  Leukocytes, Week 20, n=254, 265: number analyzed (Participants) | 254 | 265
  Leukocytes, Week 20, n=254, 265 | 0.27 (1.505) | 0.44 (1.480)
  Leukocytes, Week 24, n=258, 264: number analyzed (Participants) | 258 | 264
  Leukocytes, Week 24, n=258, 264 | 0.34 (1.581) | 0.45 (1.725)
  Leukocytes, Week 28, n=244, 263: number analyzed (Participants) | 244 | 263
  Leukocytes, Week 28, n=244, 263 | 0.34 (1.713) | 0.48 (1.551)
  Leukocytes, Week 32, n=253, 266: number analyzed (Participants) | 253 | 266
  Leukocytes, Week 32, n=253, 266 | 0.28 (1.726) | 0.42 (1.748)
  Leukocytes, Week 36, n=252, 259: number analyzed (Participants) | 252 | 259
  Leukocytes, Week 36, n=252, 259 | 0.34 (1.549) | 0.52 (1.789)
  Leukocytes, Week 40, n=246, 253: number analyzed (Participants) | 246 | 253
  Leukocytes, Week 40, n=246, 253 | 0.16 (1.497) | 0.42 (1.614)
  Leukocytes, Week 44, n=256, 262: number analyzed (Participants) | 256 | 262
  Leukocytes, Week 44, n=256, 262 | 0.22 (1.732) | 0.49 (1.626)
  Leukocytes, Week 48, n=243, 260: number analyzed (Participants) | 243 | 260
  Leukocytes, Week 48, n=243, 260 | 0.09 (1.455) | 0.29 (1.520)
  Lymphocytes, Week 4, n=277, 270: number analyzed (Participants) | 277 | 270
  Lymphocytes, Week 4, n=277, 270 | 0.198 (0.5156) | 0.231 (0.5066)
  Lymphocytes, Week 8, n=210, 272: number analyzed (Participants) | 210 | 272
  Lymphocytes, Week 8, n=210, 272 | 0.054 (0.4812) | 0.155 (0.5088)
  Lymphocytes, Week 12, n=267, 272: number analyzed (Participants) | 267 | 272
  Lymphocytes, Week 12, n=267, 272 | 0.012 (0.4632) | 0.164 (0.5560)
  Lymphocytes, Week 16, n=247, 259: number analyzed (Participants) | 247 | 259
  Lymphocytes, Week 16, n=247, 259 | 0.020 (0.4971) | 0.158 (0.5246)
  Lymphocytes, Week 20, n=247, 259: number analyzed (Participants) | 247 | 259
  Lymphocytes, Week 20, n=247, 259 | 0.030 (0.4889) | 0.146 (0.5292)
  Lymphocytes, Week 24, n=256, 260: number analyzed (Participants) | 256 | 260
  Lymphocytes, Week 24, n=256, 260 | 0.014 (0.5195) | 0.148 (0.5716)
  Lymphocytes, Week 28, n=239, 258: number analyzed (Participants) | 239 | 258
  Lymphocytes, Week 28, n=239, 258 | 0.021 (0.5389) | 0.145 (0.5469)
  Lymphocytes, Week 32, n=246, 263: number analyzed (Participants) | 246 | 263
  Lymphocytes, Week 32, n=246, 263 | 0.021 (0.5195) | 0.129 (0.5812)
  Lymphocytes, Week 36, n=250, 259: number analyzed (Participants) | 250 | 259
  Lymphocytes, Week 36, n=250, 259 | 0.028 (0.5261) | 0.132 (0.5258)
  Lymphocytes, Week 40, n=244, 245: number analyzed (Participants) | 244 | 245
  Lymphocytes, Week 40, n=244, 245 | 0.006 (0.5303) | 0.054 (0.5106)
  Lymphocytes, Week 44, n=249, 260: number analyzed (Participants) | 249 | 260
  Lymphocytes, Week 44, n=249, 260 | -0.021 (0.6176) | 0.098 (0.5139)
  Lymphocytes, Week 48, n=239, 258: number analyzed (Participants) | 239 | 258
  Lymphocytes, Week 48, n=239, 258 | -0.074 (0.5191) | 0.039 (0.5936)
  Monocytes, Week 4, n=277, 270: number analyzed (Participants) | 277 | 270
  Monocytes, Week 4, n=277, 270 | 0.038 (0.1269) | 0.031 (0.1528)
  Monocytes, Week 8, n=210, 272: number analyzed (Participants) | 210 | 272
  Monocytes, Week 8, n=210, 272 | 0.022 (0.1464) | 0.013 (0.1600)
  Monocytes, Week 12, n=267, 272: number analyzed (Participants) | 267 | 272
  Monocytes, Week 12, n=267, 272 | 0.016 (0.1234) | 0.018 (0.1613)
  Monocytes, Week 16, n=247, 259: number analyzed (Participants) | 247 | 259
  Monocytes, Week 16, n=247, 259 | 0.059 (0.1548) | 0.035 (0.1618)
  Monocytes, Week 20, n=247, 259: number analyzed (Participants) | 247 | 259
  Monocytes, Week 20, n=247, 259 | 0.070 (0.1583) | 0.053 (0.1790)
  Monocytes, Week 24, n=256, 260: number analyzed (Participants) | 256 | 260
  Monocytes, Week 24, n=256, 260 | 0.059 (0.1442) | 0.070 (0.1599)
  Monocytes, Week 28, n=239, 258: number analyzed (Participants) | 239 | 258
  Monocytes, Week 28, n=239, 258 | 0.086 (0.1584) | 0.077 (0.1806)
  Monocytes, Week 32, n=246, 263: number analyzed (Participants) | 246 | 263
  Monocytes, Week 32, n=246, 263 | 0.081 (0.1530) | 0.088 (0.1841)
  Monocytes, Week 36, n=250, 259: number analyzed (Participants) | 250 | 259
  Monocytes, Week 36, n=250, 259 | 0.084 (0.1685) | 0.086 (0.1772)
  Monocytes, Week 40, n=244, 245: number analyzed (Participants) | 244 | 245
  Monocytes, Week 40, n=244, 245 | 0.056 (0.1378) | 0.076 (0.1651)
  Monocytes, Week 44, n=249, 260: number analyzed (Participants) | 249 | 260
  Monocytes, Week 44, n=249, 260 | 0.062 (0.1522) | 0.057 (0.1558)
  Monocytes, Week 48, n=239, 258: number analyzed (Participants) | 239 | 258
  Monocytes, Week 48, n=239, 258 | 0.024 (0.1395) | 0.031 (0.1389)
  Neutrophils, Week 4, n=277, 270: number analyzed (Participants) | 277 | 270
  Neutrophils, Week 4, n=277, 270 | 0.313 (1.3508) | 0.130 (1.1869)
  Neutrophils, Week 8, n=210, 272: number analyzed (Participants) | 210 | 272
  Neutrophils, Week 8, n=210, 272 | 0.084 (1.1310) | 0.125 (1.2775)
  Neutrophils, Week 12, n=267, 272: number analyzed (Participants) | 267 | 272
  Neutrophils, Week 12, n=267, 272 | 0.032 (1.3016) | 0.185 (1.3016)
  Neutrophils, Week 16, n=247, 259: number analyzed (Participants) | 247 | 259
  Neutrophils, Week 16, n=247, 259 | 0.215 (1.5752) | 0.211 (1.4233)
  Neutrophils, Week 20, n=247, 259: number analyzed (Participants) | 247 | 259
  Neutrophils, Week 20, n=247, 259 | 0.132 (1.4116) | 0.217 (1.3130)
  Neutrophils, Week 24, n=256, 260: number analyzed (Participants) | 256 | 260
  Neutrophils, Week 24, n=256, 260 | 0.218 (1.4890) | 0.217 (1.4694)
  Neutrophils, Week 28, n=239, 258: number analyzed (Participants) | 239 | 258
  Neutrophils, Week 28, n=239, 258 | 0.193 (1.5833) | 0.221 (1.3274)
  Neutrophils, Week 32, n=246, 263: number analyzed (Participants) | 246 | 263
  Neutrophils, Week 32, n=246, 263 | 0.144 (1.5739) | 0.175 (1.5009)
  Neutrophils, Week 36, n=250, 259: number analyzed (Participants) | 250 | 259
  Neutrophils, Week 36, n=250, 259 | 0.170 (1.3865) | 0.243 (1.4938)
  Neutrophils, Week 40, n=244, 245: number analyzed (Participants) | 244 | 245
  Neutrophils, Week 40, n=244, 245 | 0.055 (1.4372) | 0.259 (1.4739)
  Neutrophils, Week 44, n=249, 260: number analyzed (Participants) | 249 | 260
  Neutrophils, Week 44, n=249, 260 | 0.156 (1.5382) | 0.273 (1.4445)
  Neutrophils, Week 48, n=239, 258: number analyzed (Participants) | 239 | 258
  Neutrophils, Week 48, n=239, 258 | 0.110 (1.3697) | 0.201 (1.3169)
  Platelets, Week 4, n=278, 269: number analyzed (Participants) | 278 | 269
  Platelets, Week 4, n=278, 269 | 5.7 (29.10) | 4.3 (31.11)
  Platelets, Week 8, n=207, 273: number analyzed (Participants) | 207 | 273
  Platelets, Week 8, n=207, 273 | -0.9 (29.09) | 2.2 (35.14)
  Platelets, Week 12, n=269, 271: number analyzed (Participants) | 269 | 271
  Platelets, Week 12, n=269, 271 | 0.8 (32.49) | 6.2 (36.23)
  Platelets, Week 16, n=251, 263: number analyzed (Participants) | 251 | 263
  Platelets, Week 16, n=251, 263 | 1.6 (33.34) | 9.3 (51.53)
  Platelets, Week 20, n=255, 264: number analyzed (Participants) | 255 | 264
  Platelets, Week 20, n=255, 264 | 7.6 (38.18) | 13.4 (39.24)
  Platelets, Week 24, n=256, 261: number analyzed (Participants) | 256 | 261
  Platelets, Week 24, n=256, 261 | 6.5 (36.11) | 14.4 (35.15)
  Platelets, Week 28, n=245, 258: number analyzed (Participants) | 245 | 258
  Platelets, Week 28, n=245, 258 | 8.6 (38.23) | 18.4 (38.56)
  Platelets, Week 32, n=249, 262: number analyzed (Participants) | 249 | 262
  Platelets, Week 32, n=249, 262 | 7.9 (40.22) | 14.6 (34.28)
  Platelets, Week 36, n=248, 259: number analyzed (Participants) | 248 | 259
  Platelets, Week 36, n=248, 259 | 12.1 (38.48) | 18.6 (35.81)
  Platelets, Week 40, n=244, 254: number analyzed (Participants) | 244 | 254
  Platelets, Week 40, n=244, 254 | 8.2 (36.08) | 17.7 (43.30)
  Platelets, Week 44, n=254, 261: number analyzed (Participants) | 254 | 261
  Platelets, Week 44, n=254, 261 | 9.4 (38.42) | 19.3 (47.64)
  Platelets, Week 48, n=240, 255: number analyzed (Participants) | 240 | 255
  Platelets, Week 48, n=240, 255 | 7.7 (39.61) | 16.4 (47.45)

27. Secondary Outcome: Change From Baseline for Hematology Parameters: Erythrocyte Mean Corpuscular Volume
Description: Blood samples were collected for the analysis of hematology parameter including erythrocyte mean corpuscular volume at indicated timepoints. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance phase dose of IP. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Femtoliters
  Week 4, n=279, 273: number analyzed (Participants) | 279 | 273
  Week 4, n=279, 273 | -0.7 (1.66) | 0.2 (1.56)
  Week 8, n=211, 275: number analyzed (Participants) | 211 | 275
  Week 8, n=211, 275 | -2.5 (2.33) | 0.2 (2.06)
  Week 12, n=270, 275: number analyzed (Participants) | 270 | 275
  Week 12, n=270, 275 | -3.8 (2.49) | -0.3 (2.48)
  Week 16, n=254, 265: number analyzed (Participants) | 254 | 265
  Week 16, n=254, 265 | -5.1 (2.63) | -0.2 (2.65)
  Week 20, n=255, 267: number analyzed (Participants) | 255 | 267
  Week 20, n=255, 267 | -5.6 (2.72) | -0.5 (2.55)
  Week 24, n=259, 264: number analyzed (Participants) | 259 | 264
  Week 24, n=259, 264 | -5.6 (2.85) | -0.5 (2.58)
  Week 28, n=246, 265: number analyzed (Participants) | 246 | 265
  Week 28, n=246, 265 | -5.6 (2.97) | -0.9 (2.52)
  Week 32, n=254, 267: number analyzed (Participants) | 254 | 267
  Week 32, n=254, 267 | -5.3 (3.02) | -0.9 (2.55)
  Week 36, n=252, 261: number analyzed (Participants) | 252 | 261
  Week 36, n=252, 261 | -5.3 (3.00) | -0.6 (2.45)
  Week 40, n=246, 255: number analyzed (Participants) | 246 | 255
  Week 40, n=246, 255 | -4.8 (3.02) | -0.1 (2.64)
  Week 44, n=256, 262: number analyzed (Participants) | 256 | 262
  Week 44, n=256, 262 | -4.2 (3.12) | 0.2 (2.81)
  Week 48, n=243, 260: number analyzed (Participants) | 243 | 260
  Week 48, n=243, 260 | -3.7 (3.12) | 1.0 (2.93)

28. Secondary Outcome: Change From Baseline for Hematology Parameters: Erythrocytes
Description: Blood samples were collected for the analysis of hematology parameters including erythrocytes at indicated timepoints. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance phase dose of IP. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^12 cells per Liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
10^12 cells per Liter
  Week 4, n=279, 273: number analyzed (Participants) | 279 | 273
  Week 4, n=279, 273 | 0.08 (0.226) | -0.03 (0.228)
  Week 8, n=211, 275: number analyzed (Participants) | 211 | 275
  Week 8, n=211, 275 | 0.18 (0.249) | 0.02 (0.239)
  Week 12, n=270, 275: number analyzed (Participants) | 270 | 275
  Week 12, n=270, 275 | 0.23 (0.269) | 0.01 (0.273)
  Week 16, n=254, 265: number analyzed (Participants) | 254 | 265
  Week 16, n=254, 265 | 0.30 (0.263) | 0.01 (0.255)
  Week 20, n=255, 267: number analyzed (Participants) | 255 | 267
  Week 20, n=255, 267 | 0.31 (0.272) | -0.01 (0.242)
  Week 24, n=259, 264: number analyzed (Participants) | 259 | 264
  Week 24, n=259, 264 | 0.31 (0.254) | 0.02 (0.242)
  Week 28, n=246, 265: number analyzed (Participants) | 246 | 265
  Week 28, n=246, 265 | 0.29 (0.248) | 0.04 (0.259)
  Week 32, n=254, 267: number analyzed (Participants) | 254 | 267
  Week 32, n=254, 267 | 0.25 (0.283) | 0.01 (0.259)
  Week 36, n=252, 261: number analyzed (Participants) | 252 | 261
  Week 36, n=252, 261 | 0.23 (0.263) | -0.01 (0.250)
  Week 40, n=246, 255: number analyzed (Participants) | 246 | 255
  Week 40, n=246, 255 | 0.23 (0.246) | -0.01 (0.239)
  Week 44, n=256, 262: number analyzed (Participants) | 256 | 262
  Week 44, n=256, 262 | 0.21 (0.234) | -0.06 (0.243)
  Week 48, n=243, 260: number analyzed (Participants) | 243 | 260
  Week 48, n=243, 260 | 0.16 (0.264) | -0.06 (0.257)

29. Secondary Outcome: Change From Baseline for Hematology Parameters: Hematocrit
Description: Blood samples were collected for the analysis of hematology parameters including hematocrit at indicated timepoints. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance phase dose of IP. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Proportion of red blood cells in blood
  Week 4, n=279, 273: number analyzed (Participants) | 279 | 273
  Week 4, n=279, 273 | 0.0046 (0.02082) | -0.0013 (0.02213)
  Week 8, n=211, 275: number analyzed (Participants) | 211 | 275
  Week 8, n=211, 275 | 0.0053 (0.02344) | 0.0026 (0.02314)
  Week 12, n=270, 275: number analyzed (Participants) | 270 | 275
  Week 12, n=270, 275 | 0.0040 (0.02383) | -0.0000 (0.02618)
  Week 16, n=254, 265: number analyzed (Participants) | 254 | 265
  Week 16, n=254, 265 | 0.0035 (0.02338) | -0.0003 (0.02489)
  Week 20, n=255, 267: number analyzed (Participants) | 255 | 267
  Week 20, n=255, 267 | 0.0024 (0.02335) | -0.0033 (0.02323)
  Week 24, n=259, 264: number analyzed (Participants) | 259 | 264
  Week 24, n=259, 264 | 0.0021 (0.02299) | -0.0012 (0.02337)
  Week 28, n=246, 265: number analyzed (Participants) | 246 | 265
  Week 28, n=246, 265 | -0.0003 (0.02262) | -0.0001 (0.02460)
  Week 32, n=254, 267: number analyzed (Participants) | 254 | 267
  Week 32, n=254, 267 | -0.0017 (0.02607) | -0.0032 (0.02503)
  Week 36, n=252, 261: number analyzed (Participants) | 252 | 261
  Week 36, n=252, 261 | -0.0041 (0.02515) | -0.0032 (0.02407)
  Week 40, n=246, 255: number analyzed (Participants) | 246 | 255
  Week 40, n=246, 255 | -0.0014 (0.02461) | -0.0017 (0.02388)
  Week 44, n=256, 262: number analyzed (Participants) | 256 | 262
  Week 44, n=256, 262 | -0.0011 (0.02230) | -0.0045 (0.02328)
  Week 48, n=243, 260: number analyzed (Participants) | 243 | 260
  Week 48, n=243, 260 | -0.0027 (0.02571) | -0.0019 (0.02572)

30. Secondary Outcome: Change From Baseline for Hematology Parameters: Hemoglobin
Description: Blood samples were collected for the analysis of hematology parameter including hemoglobin at indicated timepoints. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance Phase dose of IP. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Grams per liter
  Week 4, n=279, 273: number analyzed (Participants) | 279 | 273
  Week 4, n=279, 273 | 1.8 (6.59) | 0.1 (6.47)
  Week 8, n=211, 275: number analyzed (Participants) | 211 | 275
  Week 8, n=211, 275 | 1.9 (7.29) | 1.3 (7.26)
  Week 12, n=270, 275: number analyzed (Participants) | 270 | 275
  Week 12, n=270, 275 | 2.1 (7.47) | 1.5 (8.28)
  Week 16, n=254, 265: number analyzed (Participants) | 254 | 265
  Week 16, n=254, 265 | 2.9 (6.98) | 1.4 (7.88)
  Week 20, n=255, 267: number analyzed (Participants) | 255 | 267
  Week 20, n=255, 267 | 2.9 (7.43) | 1.4 (7.18)
  Week 24, n=259, 264: number analyzed (Participants) | 259 | 264
  Week 24, n=259, 264 | 2.7 (7.32) | 2.0 (7.11)
  Week 28, n=246, 265: number analyzed (Participants) | 246 | 265
  Week 28, n=246, 265 | 2.7 (6.80) | 3.3 (7.75)
  Week 32, n=254, 267: number analyzed (Participants) | 254 | 267
  Week 32, n=254, 267 | 2.7 (8.08) | 2.9 (7.73)
  Week 36, n=252, 261: number analyzed (Participants) | 252 | 261
  Week 36, n=252, 261 | 2.0 (7.93) | 2.8 (7.73)
  Week 40, n=246, 255: number analyzed (Participants) | 246 | 255
  Week 40, n=246, 255 | 3.2 (7.91) | 3.1 (7.85)
  Week 44, n=256, 262: number analyzed (Participants) | 256 | 262
  Week 44, n=256, 262 | 2.5 (7.66) | 1.8 (7.62)
  Week 48, n=243, 260: number analyzed (Participants) | 243 | 260
  Week 48, n=243, 260 | 1.4 (7.98) | 2.1 (8.33)

31. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Over Time Including Week 48: ALT, ALP, AST and CK
Description: Blood samples were collected for the analysis of clinical chemistry parameters including ALT, ALP, AST and CK. Baseline values is defined as the latest pre-treatment assessment with a non-missing value. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance Phase dose of IP. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
International units per liter
  ALT, Week 4, n=281, 277: number analyzed (Participants) | 281 | 277
  ALT, Week 4, n=281, 277 | 3.7 (49.90) | -1.4 (11.14)
  ALT, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  ALT, Week 8, n=212, 278 | 1.0 (14.28) | -0.9 (11.86)
  ALT, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  ALT, Week 12, n=270, 276 | 1.0 (15.80) | -0.1 (13.27)
  ALT, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  ALT, Week 16, n=255, 269 | 1.2 (16.61) | 1.5 (13.99)
  ALT, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  ALT, Week 20, n=260, 272 | 5.3 (72.80) | 0.2 (17.04)
  ALT, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  ALT, Week 24, n=261, 268 | 3.3 (30.00) | -0.4 (12.75)
  ALT, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  ALT, Week 28, n=253, 268 | 1.9 (18.82) | 0.2 (12.72)
  ALT, Week 32, n=256, 268: number analyzed (Participants) | 256 | 268
  ALT, Week 32, n=256, 268 | 18.1 (293.85) | -0.4 (13.08)
  ALT, Week 36, n=255, 261: number analyzed (Participants) | 255 | 261
  ALT, Week 36, n=255, 261 | -0.1 (14.10) | 1.7 (32.63)
  ALT, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  ALT, Week 40, n=250, 266 | 0.6 (17.42) | 0.0 (14.84)
  ALT, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  ALT, Week 44, n=258, 263 | 1.7 (27.55) | 0.8 (16.75)
  ALT, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  ALT, Week 48, n=247, 262 | -0.2 (22.91) | 0.1 (18.81)
  ALP, Week 4, n=281, 277: number analyzed (Participants) | 281 | 277
  ALP, Week 4, n=281, 277 | 0.3 (11.04) | -1.3 (15.74)
  ALP, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  ALP, Week 8, n=212, 278 | 0.6 (10.41) | -0.5 (17.00)
  ALP, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  ALP, Week 12, n=270, 276 | 1.4 (12.71) | -0.7 (17.40)
  ALP, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  ALP, Week 16, n=255, 269 | 0.8 (10.34) | -0.3 (17.99)
  ALP, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  ALP, Week 20, n=260, 272 | 1.5 (10.20) | -1.1 (17.35)
  ALP, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  ALP, Week 24, n=261, 268 | 1.2 (9.57) | -0.7 (17.03)
  ALP, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  ALP, Week 28, n=253, 268 | 1.4 (10.57) | 0.6 (17.28)
  ALP, Week 32, n=256, 268: number analyzed (Participants) | 256 | 268
  ALP, Week 32, n=256, 268 | 1.9 (15.42) | -0.3 (18.11)
  ALP, Week 36, n=255, 261: number analyzed (Participants) | 255 | 261
  ALP, Week 36, n=255, 261 | 3.3 (20.31) | 1.3 (20.90)
  ALP, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  ALP, Week 40, n=250, 266 | 1.8 (9.84) | 0.7 (18.50)
  ALP, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  ALP, Week 44, n=258, 263 | 1.4 (11.00) | 1.2 (17.62)
  ALP, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  ALP, Week 48, n=247, 262 | 1.1 (12.75) | 0.7 (17.54)
  AST, Week 4, n=281, 277: number analyzed (Participants) | 281 | 277
  AST, Week 4, n=281, 277 | 1.5 (24.47) | -1.6 (14.58)
  AST, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  AST, Week 8, n=212, 278 | 0.7 (19.90) | -2.0 (14.13)
  AST, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  AST, Week 12, n=270, 276 | -0.3 (10.74) | -1.5 (15.34)
  AST, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  AST, Week 16, n=255, 269 | -0.1 (11.31) | 1.0 (16.68)
  AST, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  AST, Week 20, n=260, 272 | 2.3 (32.28) | 0.2 (26.46)
  AST, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  AST, Week 24, n=261, 268 | 2.8 (24.22) | -1.5 (16.00)
  AST, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  AST, Week 28, n=253, 268 | 1.7 (15.85) | -0.9 (16.99)
  AST, Week 32, n=256, 268: number analyzed (Participants) | 256 | 268
  AST, Week 32, n=256, 268 | 14.0 (233.48) | -1.9 (14.68)
  AST, Week 36, n=255, 261: number analyzed (Participants) | 255 | 261
  AST, Week 36, n=255, 261 | -0.1 (12.22) | -0.2 (22.03)
  AST, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  AST, Week 40, n=250, 266 | 0.2 (13.31) | -1.5 (15.24)
  AST, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  AST, Week 44, n=258, 263 | 1.3 (16.49) | -0.5 (18.31)
  AST Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  AST Week 48, n=247, 262 | -0.8 (11.88) | 0.8 (44.70)
  CK, Week 4, n=280, 277: number analyzed (Participants) | 280 | 277
  CK, Week 4, n=280, 277 | 31.1 (456.63) | -27.0 (523.89)
  CK, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  CK, Week 8, n=212, 278 | 53.5 (907.83) | -46.6 (499.91)
  CK, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  CK, Week 12, n=270, 276 | 1.2 (420.32) | -17.2 (605.92)
  CK, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  CK, Week 16, n=255, 269 | -18.0 (316.74) | 40.2 (746.32)
  CK, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  CK, Week 20, n=260, 272 | 19.2 (536.70) | 57.3 (1208.73)
  CK, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  CK, Week 24, n=261, 268 | 47.3 (635.42) | -19.6 (605.13)
  CK, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  CK, Week 28, n=253, 268 | 49.9 (669.37) | -8.5 (705.35)
  CK, Week 32, n=256, 268: number analyzed (Participants) | 256 | 268
  CK, Week 32, n=256, 268 | -24.5 (298.70) | -42.5 (509.77)
  CK, Week 36, n=254, 261: number analyzed (Participants) | 254 | 261
  CK, Week 36, n=254, 261 | 14.7 (515.62) | 12.2 (674.76)
  CK, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  CK, Week 40, n=250, 266 | 24.8 (544.72) | -51.7 (497.70)
  CK, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  CK, Week 44, n=258, 263 | 54.8 (526.28) | -20.1 (652.24)
  CK, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  CK, Week 48, n=247, 262 | -17.8 (309.33) | 121.1 (2682.33)

32. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameter Over Time Including Week 48: Albumin
Description: Blood samples were collected for the analysis of clinical chemistry parameter-albumin. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance Phase dose of IP. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Grams per liter
  Week 4, n=280, 277: number analyzed (Participants) | 280 | 277
  Week 4, n=280, 277 | -0.1 (2.15) | -0.3 (2.14)
  Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Week 8, n=212, 278 | -0.1 (2.32) | -0.3 (2.25)
  Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Week 12, n=270, 276 | -0.1 (2.38) | 0.0 (2.58)
  Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  Week 16, n=255, 269 | 0.2 (2.23) | -0.1 (2.48)
  Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  Week 20, n=260, 272 | 0.2 (2.51) | -0.2 (2.47)
  Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  Week 24, n=261, 268 | 0.5 (2.28) | 0.2 (2.37)
  Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Week 28, n=253, 268 | 0.5 (2.42) | 0.4 (2.32)
  Week 32, n=255, 268: number analyzed (Participants) | 255 | 268
  Week 32, n=255, 268 | 0.7 (2.47) | 0.4 (2.60)
  Week 36, n=254, 261: number analyzed (Participants) | 254 | 261
  Week 36, n=254, 261 | 0.3 (2.44) | 0.3 (2.52)
  Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Week 40, n=250, 266 | 0.9 (2.42) | 0.5 (2.46)
  Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Week 44, n=258, 263 | 0.9 (2.44) | 0.4 (2.49)
  Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Week 48, n=247, 262 | 0.7 (2.40) | 0.5 (2.63)

33. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters Over Time Including Week 48: Bilirubin, Direct Bilirubin and Creatinine
Description: Blood samples were collected for the analysis of clinical chemistry parameters including bilirubin, creatinine and direct bilirubin. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance Phase dose of IP. Baseline value is defined as the latest pre-treatment assessment with a non-missing value. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Micromoles per liter
  Bilirubin, Week 4, n=281, 277: number analyzed (Participants) | 281 | 277
  Bilirubin, Week 4, n=281, 277 | 1.4 (4.74) | -0.3 (3.77)
  Bilirubin, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Bilirubin, Week 8, n=212, 278 | 0.9 (4.04) | -0.5 (4.17)
  Bilirubin, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Bilirubin, Week 12, n=270, 276 | 1.2 (4.15) | -0.7 (4.51)
  Bilirubin, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  Bilirubin, Week 16, n=255, 269 | 1.2 (4.30) | -0.3 (3.61)
  Bilirubin, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  Bilirubin, Week 20, n=260, 272 | 1.1 (4.14) | -0.7 (4.02)
  Bilirubin, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  Bilirubin, Week 24, n=261, 268 | 0.8 (4.12) | -0.4 (3.85)
  Bilirubin, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Bilirubin, Week 28, n=253, 268 | 1.2 (4.41) | -0.7 (3.75)
  Bilirubin, Week 32, n=256, 268: number analyzed (Participants) | 256 | 268
  Bilirubin, Week 32, n=256, 268 | 1.3 (6.44) | -0.6 (4.05)
  Bilirubin, Week 36, n=255, 260: number analyzed (Participants) | 255 | 260
  Bilirubin, Week 36, n=255, 260 | 0.6 (5.36) | -0.7 (4.28)
  Bilirubin, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Bilirubin, Week 40, n=250, 266 | 0.9 (4.31) | -0.8 (4.32)
  Bilirubin, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Bilirubin, Week 44, n=258, 263 | 1.2 (4.34) | -0.4 (4.28)
  Bilirubin, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Bilirubin, Week 48, n=247, 262 | 1.1 (4.18) | -0.3 (4.17)
  Direct bilirubin, Week 4, n=277, 277: number analyzed (Participants) | 277 | 277
  Direct bilirubin, Week 4, n=277, 277 | 0.2 (1.40) | -0.1 (1.33)
  Direct bilirubin, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Direct bilirubin, Week 8, n=212, 278 | 0.2 (1.30) | -0.1 (1.19)
  Direct bilirubin, Week 12, n=269, 273: number analyzed (Participants) | 269 | 273
  Direct bilirubin, Week 12, n=269, 273 | 0.2 (1.22) | 0.0 (1.22)
  Direct bilirubin, Week 16, n=254, 268: number analyzed (Participants) | 254 | 268
  Direct bilirubin, Week 16, n=254, 268 | 0.2 (1.44) | -0.1 (1.14)
  Direct bilirubin, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  Direct bilirubin, Week 20, n=260, 272 | 0.2 (1.57) | -0.1 (1.14)
  Direct bilirubin, Week 24, n=260, 266: number analyzed (Participants) | 260 | 266
  Direct bilirubin, Week 24, n=260, 266 | 0.1 (1.46) | -0.1 (1.10)
  Direct bilirubin, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Direct bilirubin, Week 28, n=253, 268 | 0.2 (1.26) | -0.1 (1.22)
  Direct bilirubin, Week 32, n=256, 268: number analyzed (Participants) | 256 | 268
  Direct bilirubin, Week 32, n=256, 268 | 0.3 (3.39) | -0.1 (1.08)
  Direct bilirubin, Week 36, n=255, 260: number analyzed (Participants) | 255 | 260
  Direct bilirubin, Week 36, n=255, 260 | 0.1 (2.18) | -0.1 (1.16)
  Direct bilirubin, Week 40, n=249, 266: number analyzed (Participants) | 249 | 266
  Direct bilirubin, Week 40, n=249, 266 | 0.1 (1.42) | -0.1 (1.26)
  Direct bilirubin, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Direct bilirubin, Week 44, n=258, 263 | 0.2 (1.41) | -0.1 (1.19)
  Direct bilirubin, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Direct bilirubin, Week 48, n=247, 262 | 0.0 (1.41) | 0.0 (1.19)
  Creatinine, Week 4, n=280, 277: number analyzed (Participants) | 280 | 277
  Creatinine, Week 4, n=280, 277 | -6.07 (9.696) | 0.61 (7.635)
  Creatinine, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Creatinine, Week 8, n=212, 278 | -9.25 (9.936) | -0.24 (8.838)
  Creatinine, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Creatinine, Week 12, n=270, 276 | -9.89 (9.703) | -1.20 (8.710)
  Creatinine, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  Creatinine, Week 16, n=255, 269 | -9.75 (9.572) | -0.33 (8.964)
  Creatinine, Week 20, n=261, 272: number analyzed (Participants) | 261 | 272
  Creatinine, Week 20, n=261, 272 | -10.10 (9.839) | -0.68 (8.700)
  Creatinine, Week 24, n=262, 268: number analyzed (Participants) | 262 | 268
  Creatinine, Week 24, n=262, 268 | -9.73 (9.499) | -0.75 (8.327)
  Creatinine, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Creatinine, Week 28, n=253, 268 | -10.34 (9.731) | -1.33 (8.892)
  Creatinine, Week 32, n=255, 268: number analyzed (Participants) | 255 | 268
  Creatinine, Week 32, n=255, 268 | -9.77 (9.166) | -1.26 (9.243)
  Creatinine, Week 36, n=254, 262: number analyzed (Participants) | 254 | 262
  Creatinine, Week 36, n=254, 262 | -9.57 (9.712) | -0.74 (8.565)
  Creatinine, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Creatinine, Week 40, n=250, 266 | -9.60 (10.656) | -1.10 (7.875)
  Creatinine, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Creatinine, Week 44, n=258, 263 | -9.02 (9.562) | -1.91 (8.306)
  Creatinine, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Creatinine, Week 48, n=247, 262 | -8.97 (9.742) | 5.00 (85.535)

34. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters Over Time Including Week 48
Description: Blood samples were collected for the analysis of clinical chemistry parameters which includes total CO2, chloride, glucose, phosphate, potassium, sodium and urea. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance Phase dose of IP. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Millimoles per liter
  CO2, Week 4, n=280, 276: number analyzed (Participants) | 280 | 276
  CO2, Week 4, n=280, 276 | 0.6 (2.67) | 0.2 (2.32)
  CO2, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  CO2, Week 8, n=212, 278 | 0.2 (2.51) | -0.1 (2.24)
  CO2, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  CO2, Week 12, n=270, 276 | 0.2 (2.56) | -0.1 (2.26)
  CO2, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  CO2, Week 16, n=255, 269 | 0.4 (2.55) | -0.1 (2.72)
  CO2, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  CO2, Week 20, n=260, 272 | 0.3 (2.52) | 0.1 (2.38)
  CO2, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  CO2, Week 24, n=261, 268 | 0.6 (2.84) | 0.4 (2.56)
  CO2, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  CO2, Week 28, n=253, 268 | 0.5 (2.51) | 0.4 (2.39)
  CO2, Week 32, n=255, 268: number analyzed (Participants) | 255 | 268
  CO2, Week 32, n=255, 268 | 0.5 (2.72) | 0.3 (2.37)
  CO2, Week 36, n=253, 261: number analyzed (Participants) | 253 | 261
  CO2, Week 36, n=253, 261 | 0.7 (2.54) | 0.2 (2.35)
  CO2, Week 40, n=249, 265: number analyzed (Participants) | 249 | 265
  CO2, Week 40, n=249, 265 | 0.4 (2.53) | 0.2 (2.61)
  CO2, Week 44, n=257, 263: number analyzed (Participants) | 257 | 263
  CO2, Week 44, n=257, 263 | 0.4 (2.71) | 0.1 (2.37)
  CO2, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  CO2, Week 48, n=247, 262 | 0.0 (2.70) | 0.0 (2.27)
  Chloride, Week 4, n=280, 277: number analyzed (Participants) | 280 | 277
  Chloride, Week 4, n=280, 277 | 0.0 (2.13) | 0.5 (2.17)
  Chloride, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Chloride, Week 8, n=212, 278 | 0.0 (2.05) | 0.3 (2.14)
  Chloride, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Chloride, Week 12, n=270, 276 | 0.0 (2.10) | 0.4 (2.16)
  Chloride, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  Chloride, Week 16, n=255, 269 | -0.2 (2.32) | 0.3 (2.39)
  Chloride, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  Chloride, Week 20, n=260, 272 | -0.3 (2.49) | 0.4 (2.15)
  Chloride, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  Chloride, Week 24, n=261, 268 | -0.2 (2.40) | 0.2 (2.47)
  Chloride, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Chloride, Week 28, n=253, 268 | -0.2 (2.21) | 0.1 (2.18)
  Chloride, Week 32, n=255, 268: number analyzed (Participants) | 255 | 268
  Chloride, Week 32, n=255, 268 | -0.2 (2.37) | 0.3 (2.34)
  Chloride, Week 36, n=254, 261: number analyzed (Participants) | 254 | 261
  Chloride, Week 36, n=254, 261 | -0.1 (2.46) | 0.4 (2.37)
  Chloride, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Chloride, Week 40, n=250, 266 | 0.1 (2.35) | 0.4 (2.20)
  Chloride, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Chloride, Week 44, n=258, 263 | 0.1 (2.40) | 0.7 (2.23)
  Chloride, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Chloride, Week 48, n=247, 262 | 0.0 (2.23) | 0.3 (2.09)
  Phosphate, Week 4, n=279, 277: number analyzed (Participants) | 279 | 277
  Phosphate, Week 4, n=279, 277 | 0.032 (0.1865) | 0.014 (0.1771)
  Phosphate, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Phosphate, Week 8, n=212, 278 | -0.016 (0.1834) | 0.017 (0.1855)
  Phosphate, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Phosphate, Week 12, n=270, 276 | -0.010 (0.1825) | 0.009 (0.1772)
  Phosphate, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  Phosphate, Week 16, n=255, 269 | 0.000 (0.1789) | 0.017 (0.1892)
  Phosphate, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  Phosphate, Week 20, n=260, 272 | -0.029 (0.1932) | 0.016 (0.1764)
  Phosphate, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  Phosphate, Week 24, n=261, 268 | -0.001 (0.1907) | 0.011 (0.1852)
  Phosphate, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Phosphate, Week 28, n=253, 268 | -0.007 (0.1894) | 0.019 (0.1882)
  Phosphate, Week 32, n=255, 268: number analyzed (Participants) | 255 | 268
  Phosphate, Week 32, n=255, 268 | -0.004 (0.1806) | 0.005 (0.2092)
  Phosphate, Week 36, n=254, 261: number analyzed (Participants) | 254 | 261
  Phosphate, Week 36, n=254, 261 | -0.006 (0.1798) | 0.021 (0.1965)
  Phosphate, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Phosphate, Week 40, n=250, 266 | -0.011 (0.1851) | 0.015 (0.1753)
  Phosphate, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Phosphate, Week 44, n=258, 263 | -0.004 (0.1824) | 0.020 (0.1801)
  Phosphate, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Phosphate, Week 48, n=247, 262 | -0.007 (0.1784) | 0.020 (0.2333)
  Potassium, Week 4, n=280, 277: number analyzed (Participants) | 280 | 277
  Potassium, Week 4, n=280, 277 | 0.15 (0.334) | 0.06 (0.368)
  Potassium, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Potassium, Week 8, n=212, 278 | 0.10 (0.348) | 0.08 (0.346)
  Potassium, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Potassium, Week 12, n=270, 276 | 0.09 (0.352) | 0.05 (0.305)
  Potassium, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  Potassium, Week 16, n=255, 269 | 0.10 (0.321) | 0.04 (0.314)
  Potassium, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  Potassium, Week 20, n=260, 272 | 0.09 (0.374) | 0.04 (0.364)
  Potassium, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  Potassium, Week 24, n=261, 268 | 0.12 (0.353) | 0.07 (0.309)
  Potassium, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Potassium, Week 28, n=253, 268 | 0.08 (0.341) | 0.08 (0.350)
  Potassium, Week 32, n=255, 268: number analyzed (Participants) | 255 | 268
  Potassium, Week 32, n=255, 268 | 0.09 (0.334) | 0.06 (0.345)
  Potassium, Week 36, n=254, 261: number analyzed (Participants) | 254 | 261
  Potassium, Week 36, n=254, 261 | 0.10 (0.353) | 0.08 (0.347)
  Potassium, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Potassium, Week 40, n=250, 266 | 0.07 (0.347) | 0.06 (0.345)
  Potassium, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Potassium, Week 44, n=258, 263 | 0.08 (0.353) | 0.06 (0.338)
  Potassium, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Potassium, Week 48, n=247, 262 | 0.01 (0.343) | 0.03 (0.496)
  Sodium, Week 4, n=280, 277: number analyzed (Participants) | 280 | 277
  Sodium, Week 4, n=280, 277 | 0.3 (2.25) | 0.2 (1.95)
  Sodium, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Sodium, Week 8, n=212, 278 | 0.1 (1.98) | 0.1 (1.92)
  Sodium, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Sodium, Week 12, n=270, 276 | 0.3 (1.84) | 0.1 (1.89)
  Sodium, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  Sodium, Week 16, n=255, 269 | 0.2 (2.10) | 0.3 (2.21)
  Sodium, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  Sodium, Week 20, n=260, 272 | 0.2 (2.08) | 0.4 (1.79)
  Sodium, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  Sodium, Week 24, n=261, 268 | 0.2 (2.02) | 0.2 (2.12)
  Sodium, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Sodium, Week 28, n=253, 268 | 0.2 (1.88) | 0.4 (1.82)
  Sodium, Week 32, n=255, 268: number analyzed (Participants) | 255 | 268
  Sodium, Week 32, n=255, 268 | 0.3 (2.13) | 0.3 (2.02)
  Sodium, Week 36, n=254, 261: number analyzed (Participants) | 254 | 261
  Sodium, Week 36, n=254, 261 | 0.2 (2.16) | 0.4 (1.94)
  Sodium, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Sodium, Week 40, n=250, 266 | 0.1 (2.08) | 0.4 (2.13)
  Sodium, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Sodium, Week 44, n=258, 263 | 0.3 (2.30) | 0.4 (2.01)
  Sodium, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Sodium, Week 48, n=247, 262 | 0.2 (2.11) | 0.3 (1.72)
  Urea, Week 4, n=280, 277: number analyzed (Participants) | 280 | 277
  Urea, Week 4, n=280, 277 | 0.04 (1.292) | -0.05 (1.240)
  Urea, Week 8, n=212, 278: number analyzed (Participants) | 212 | 278
  Urea, Week 8, n=212, 278 | 0.04 (1.315) | -0.05 (1.278)
  Urea, Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Urea, Week 12, n=270, 276 | -0.01 (1.287) | 0.04 (1.340)
  Urea, Week 16, n=255, 269: number analyzed (Participants) | 255 | 269
  Urea, Week 16, n=255, 269 | 0.02 (1.394) | 0.01 (1.171)
  Urea, Week 20, n=260, 272: number analyzed (Participants) | 260 | 272
  Urea, Week 20, n=260, 272 | -0.07 (1.359) | 0.04 (1.190)
  Urea, Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  Urea, Week 24, n=261, 268 | 0.09 (1.459) | -0.08 (1.154)
  Urea, Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Urea, Week 28, n=253, 268 | 0.02 (1.412) | 0.02 (1.230)
  Urea, Week 32, n=255, 268: number analyzed (Participants) | 255 | 268
  Urea, Week 32, n=255, 268 | 0.16 (1.364) | -0.03 (1.330)
  Urea, Week 36, n=254, 261: number analyzed (Participants) | 254 | 261
  Urea, Week 36, n=254, 261 | 0.05 (1.451) | 0.04 (1.265)
  Urea, Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Urea, Week 40, n=250, 266 | 0.07 (1.466) | 0.05 (1.312)
  Urea, Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Urea, Week 44, n=258, 263 | 0.12 (1.361) | 0.03 (1.290)
  Urea, Week 48, n=247, 262: number analyzed (Participants) | 247 | 262
  Urea, Week 48, n=247, 262 | 0.09 (1.362) | 0.06 (2.189)

35. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameter Over Time Including Week 48: Lipase
Description: Blood samples were collected for the analysis of clinical chemistry parameter-lipase. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance Phase dose of IP. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Units per liter
  Week 4, n=278, 276: number analyzed (Participants) | 278 | 276
  Week 4, n=278, 276 | 1.6 (23.51) | 1.8 (30.92)
  Week 8, n=211, 278: number analyzed (Participants) | 211 | 278
  Week 8, n=211, 278 | 0.8 (19.07) | 0.4 (27.41)
  Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Week 12, n=270, 276 | 1.3 (18.55) | 2.5 (29.44)
  Week 16, n=254, 269: number analyzed (Participants) | 254 | 269
  Week 16, n=254, 269 | 0.8 (20.27) | 1.2 (27.24)
  Week 20, n=260, 270: number analyzed (Participants) | 260 | 270
  Week 20, n=260, 270 | 1.6 (16.26) | 0.8 (27.96)
  Week 24, n=260, 268: number analyzed (Participants) | 260 | 268
  Week 24, n=260, 268 | 0.9 (18.74) | 0.9 (27.58)
  Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Week 28, n=253, 268 | -0.4 (16.73) | 1.8 (29.09)
  Week 32, n=254, 268: number analyzed (Participants) | 254 | 268
  Week 32, n=254, 268 | 2.9 (29.88) | 2.0 (34.42)
  Week 36, n=254, 261: number analyzed (Participants) | 254 | 261
  Week 36, n=254, 261 | 1.0 (17.45) | -0.1 (28.89)
  Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Week 40, n=250, 266 | 2.3 (22.71) | 0.6 (27.95)
  Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Week 44, n=258, 263 | 5.7 (41.87) | 1.6 (29.05)
  Week 48, n=247, 261: number analyzed (Participants) | 247 | 261
  Week 48, n=247, 261 | 0.7 (16.14) | 1.1 (32.35)

36. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameter Over Time Including Week 48: Creatinine Clearance
Description: Blood samples were collected for the analysis of clinical chemistry parameter-creatinine clearance. GFR will be estimated by the central laboratory using the CKD-EPI. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance Phase dose of IP. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mL/min/1.73/m^2
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
mL/min/1.73/m^2
  Week 4, n=278, 277: number analyzed (Participants) | 278 | 277
  Week 4, n=278, 277 | 6.9 (10.16) | -1.2 (8.72)
  Week 8, n=211, 278: number analyzed (Participants) | 211 | 278
  Week 8, n=211, 278 | 10.0 (11.83) | 0.2 (9.13)
  Week 12, n=270, 276: number analyzed (Participants) | 270 | 276
  Week 12, n=270, 276 | 10.7 (11.49) | 0.9 (9.83)
  Week 16, n=254, 269: number analyzed (Participants) | 254 | 269
  Week 16, n=254, 269 | 10.4 (11.28) | -0.3 (10.23)
  Week 20, n=261, 271: number analyzed (Participants) | 261 | 271
  Week 20, n=261, 271 | 10.9 (11.45) | 0.3 (9.90)
  Week 24, n=261, 268: number analyzed (Participants) | 261 | 268
  Week 24, n=261, 268 | 10.5 (11.38) | 0.2 (9.63)
  Week 28, n=253, 268: number analyzed (Participants) | 253 | 268
  Week 28, n=253, 268 | 10.9 (11.90) | 1.0 (9.90)
  Week 32, n=254, 268: number analyzed (Participants) | 254 | 268
  Week 32, n=254, 268 | 10.6 (11.45) | 1.1 (10.05)
  Week 36, n=254, 262: number analyzed (Participants) | 254 | 262
  Week 36, n=254, 262 | 10.3 (11.94) | 0.2 (10.08)
  Week 40, n=250, 266: number analyzed (Participants) | 250 | 266
  Week 40, n=250, 266 | 10.2 (12.57) | 0.7 (9.19)
  Week 44, n=258, 263: number analyzed (Participants) | 258 | 263
  Week 44, n=258, 263 | 9.8 (11.61) | 1.4 (9.88)
  Week 48, n=247, 261: number analyzed (Participants) | 247 | 261
  Week 48, n=247, 261 | 9.5 (11.35) | -0.7 (10.86)

37. Secondary Outcome: Change From Baseline Values for Fasting Lipid Panel and Glucose Overtime Including Week 48
Description: Blood samples were collected at Baseline and at Week 48 to assess glucose and fasting lipids which included total cholesterol, high density lipoprotein (HDL)cholesterol, low density lipoprotein (LDL) cholesterol and triglycerides. Only fasting data is presented for glucose and lipids. Baseline value is defined as the last available fasting recorded value up to and including the date of first Maintenance Phase dose of IP. Change from Baseline value is calculated as the value at Week 48 visit (if collected while fasting) minus the Baseline value.
Time Frame: Baseline (Day 1) and at Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Millimoles per liter
  Glucose, Week 48, n=248, 251: number analyzed (Participants) | 248 | 251
  Glucose, Week 48, n=248, 251 | 0.02 (1.220) | 0.04 (0.923)
  Total Cholesterol, Week 48, n=240, 239: number analyzed (Participants) | 240 | 239
  Total Cholesterol, Week 48, n=240, 239 | 0.09 (0.658) | 0.05 (0.607)
  HDL cholesterol, Week 48, n=240, 239: number analyzed (Participants) | 240 | 239
  HDL cholesterol, Week 48, n=240, 239 | 0.109 (0.2587) | 0.076 (0.2478)
  LDL cholesterol, Week 48, n=238, 237: number analyzed (Participants) | 238 | 237
  LDL cholesterol, Week 48, n=238, 237 | 0.122 (0.5807) | -0.045 (0.5384)
  Triglycerides, Week 48, n=240, 239: number analyzed (Participants) | 240 | 239
  Triglycerides, Week 48, n=240, 239 | -0.085 (0.7167) | 0.073 (0.8361)

38. Secondary Outcome: Change From Baseline Values in Urine Albumin/Creatinine Ratio and Urine Protein/Creatinine Ratio Over Time Including Week 48
Description: Urine biomarker samples were collected for the analysis of urine albumin/creatinine ratio and urine protein/creatinine ratio. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance Phase dose of IP. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 24 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per mole
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Grams per mole
  Urine albumin/creatinine ratio, Week 4,n=199, 194: number analyzed (Participants) | 199 | 194
  Urine albumin/creatinine ratio, Week 4,n=199, 194 | 0.36 (6.714) | 0.23 (4.062)
  Urine albumin/creatinine ratio, Week 24,n=137, 184: number analyzed (Participants) | 137 | 184
  Urine albumin/creatinine ratio, Week 24,n=137, 184 | 0.30 (4.941) | 1.06 (7.186)
  Urine albumin/creatinine ratio, Week 48,n=181, 184: number analyzed (Participants) | 181 | 184
  Urine albumin/creatinine ratio, Week 48,n=181, 184 | -0.53 (17.469) | 0.19 (3.944)
  Urine protein/creatinine, Week 4, n=211, 215: number analyzed (Participants) | 211 | 215
  Urine protein/creatinine, Week 4, n=211, 215 | -0.16 (18.641) | 0.19 (6.439)
  Urine protein/creatinine, Week 24, n=151, 204: number analyzed (Participants) | 151 | 204
  Urine protein/creatinine, Week 24, n=151, 204 | 2.23 (35.187) | 1.32 (12.171)
  Urine protein/creatinine, Week 48, n=194, 197: number analyzed (Participants) | 194 | 197
  Urine protein/creatinine, Week 48, n=194, 197 | -1.86 (21.898) | 0.26 (8.180)

39. Secondary Outcome: Change From Baseline Values in Urine Creatinine Over Time Including Week 48
Description: Urine biomarker samples were collected for the analysis of urine creatinine. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance Phase dose of IP. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 24 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Micromoles per liter
  Week 4, n=277, 272: number analyzed (Participants) | 277 | 272
  Week 4, n=277, 272 | -519.5 (9558.55) | -429.0 (9540.31)
  Week 24, n=193, 258: number analyzed (Participants) | 193 | 258
  Week 24, n=193, 258 | -597.4 (9405.95) | -17.1 (9575.04)
  Week 48, n=260, 258: number analyzed (Participants) | 260 | 258
  Week 48, n=260, 258 | -1359.2 (9059.43) | -505.4 (8873.05)

40. Secondary Outcome: Change From Baseline Values in Urine Phosphate Over Time Including Week 48
Description: Urine biomarker samples were collected for the analysis of urine phosphate. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance Phase dose of IP. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 24 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Micromoles per liter
  Week 4, n=275, 273: number analyzed (Participants) | 275 | 273
  Week 4, n=275, 273 | 1.842 (18.4414) | -0.693 (18.4830)
  Week 24, n=192, 260: number analyzed (Participants) | 192 | 260
  Week 24, n=192, 260 | 0.585 (19.2777) | -0.689 (16.9500)
  Week 48, n=259, 258: number analyzed (Participants) | 259 | 258
  Week 48, n=259, 258 | 0.043 (17.3741) | 0.304 (16.7073)

41. Secondary Outcome: Change From Baseline Values in Urine Retinol Binding Protein Over Time Including Week 48
Description: Urine biomarker samples were collected for the analysis of urine retinol binding protein. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance Phase dose of IP. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Week 48
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanomoles per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Nanomoles per liter | -0.33 (0.938) | -0.24 (0.932)

42. Secondary Outcome: Change From Baseline Values in Urine Specific Gravity Over Time Including Week 48
Description: Urine biomarker samples were collected for the analysis of urine specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance Phase dose of IP. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value. The urine specific gravity was measured as the ratio of urine density compared with water density.
Time Frame: Baseline (Day 1) and at Weeks 4, 24 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Ratio of urine density to water density
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Ratio of urine density to water density
  Week 4, n=271, 266: number analyzed (Participants) | 271 | 266
  Week 4, n=271, 266 | -0.0004 (0.00837) | -0.0005 (0.00798)
  Week 24, n=191, 252: number analyzed (Participants) | 191 | 252
  Week 24, n=191, 252 | -0.0001 (0.00805) | -0.0002 (0.00825)
  Week 48, n=255, 252: number analyzed (Participants) | 255 | 252
  Week 48, n=255, 252 | -0.0009 (0.00784) | -0.0007 (0.00783)

43. Secondary Outcome: Change From Baseline Values in Urine pH Over Time Including Week 48
Description: Urine samples were collected for analysis of urine pH. pH is calculated on a scale of 0 to 14, values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH of less than 7 is acidic and a pH of greater than 7 is basic. Normal urine has a slightly acidic pH (5.0-6.0). Baseline value is defined as the last available recorded value up to and including the date of first Maintenance Phase dose of IP. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 4, 24 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
pH
  Week 4, n=271, 266: number analyzed (Participants) | 271 | 266
  Week 4, n=271, 266 | 0.12 (0.833) | 0.01 (0.884)
  Week 24, n=191, 252: number analyzed (Participants) | 191 | 252
  Week 24, n=191, 252 | -0.01 (0.889) | -0.07 (0.910)
  Week 48, n=255, 252: number analyzed (Participants) | 255 | 252
  Week 48, n=255, 252 | 0.01 (0.926) | -0.10 (0.988)

44. Secondary Outcome: Number of Participants Who Discontinued or Withdrawn Due to AEs Over Time Including Week 48
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. All Maintenance Phase adverse events (start date occurring on or after the date of first dose of randomized study treatment) leading to withdrawal have been presented.
Time Frame: Up to Week 48
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Participants | 9 | 4

45. Secondary Outcome: Percentage Change From Baseline in Fasting Lipids Overtime Including Week 48
Description: Blood samples were collected at Baseline and at Week 48 to assess fasting lipids which included total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides. Baseline value is defined as the last available recorded fasting value up to and including the date of first Maintenance Phase dose of IP. Percentage change from baseline is calculated as: value at Week 48 (if collected while fasting) minus Baseline value divided by Baseline value multiplied by 100.
Time Frame: Baseline (Day 1) and at Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Millimoles per liter
  Cholesterol, Week 48, Overall, n=240, 239: number analyzed (Participants) | 240 | 239
  Cholesterol, Week 48, Overall, n=240, 239 | 5.09 (15.695) | 2.32 (14.456)
  HDL cholesterol, Week 48, Overall, n=240, 239: number analyzed (Participants) | 240 | 239
  HDL cholesterol, Week 48, Overall, n=240, 239 | 15.448 (78.5208) | 7.361 (20.3088)
  LDL cholesterol, Week 48, Overall, n=238, 237: number analyzed (Participants) | 238 | 237
  LDL cholesterol, Week 48, Overall, n=238, 237 | 7.048 (29.2139) | 0.462 (23.9648)
  Triglycerides, Week 48, Overall, n=240, 239: number analyzed (Participants) | 240 | 239
  Triglycerides, Week 48, Overall, n=240, 239 | 2.633 (44.1663) | 14.252 (62.2823)

46. Secondary Outcome: Number of Participants With Phenotypic Resistance Through Week 48
Description: Plasma samples were collected and analyzed from participants who met confirmed virologic withdrawal criteria. Phenotypic Resistance data for following drugs :CAB,dolutegravir(DTG),elvitegravir (EVG), raltegravir(RAL),delavirdine(DLV),efavirenz(EFV),etravirine(ETR),nevirapine(NVP),RPV,lamivudine(3TC),abacavir(ABC),emtricitabine(FTC),tenofovir(TDF),zidovudine(ZDV),stavudine(d4T),didanosine(ddI),atazanavir(ATV),darunavir(DRV),fosamprenavir(FPV),indinavir(IDV),lopinavir(LPV),nelfinavir(NFV),ritonavir(RTV), saquinavir(SQV) and tipranavir (TPV) in participants meeting CVF criteria is presented.Phenotypic resistance, partially sensitive, and Sensitive were defined based on fold change(FC) value from Monogram as:resistance (FC>clinical higher cutoff/biologic cutoff),partially sensitive (FC=clinical higher cutoff and > clinical lower cutoff),sensitive(FC<=clinical lower cutoff/biologic cutoff). The CVF population comprised of all participants in ITT-E population who met CVF criteria
Time Frame: Week 48
Population: CVF Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 3 | 3
Participants
  INI, CAB, sensitive | 0 | 3
  INI, CAB, partially sensitive | 0 | 0
  INI, CAB, resistant | 3 | 0
  INI, DTG, sensitive | 3 | 3
  INI, DTG, partially sensitive | 0 | 0
  INI, DTG, resistant | 0 | 0
  INI, EVG, sensitive | 0 | 3
  INI, EVG, partially sensitive | 0 | 0
  INI, EVG, resistant | 3 | 0
  INI, RAL, sensitive | 0 | 3
  INI, RAL, partially sensitive | 0 | 0
  INI, RAL, resistant | 3 | 0
  NNRTI, DLV, sensitive | 1 | 3
  NNRTI, DLV, partially sensitive | 0 | 0
  NNRTI, DLV, resistant | 2 | 0
  NNRTI, EFV, sensitive | 1 | 3
  NNRTI, EFV, partially sensitive | 0 | 0
  NNRTI, EFV, resistant | 2 | 0
  NNRTI, ETR, sensitive | 2 | 3
  NNRTI, ETR, partially sensitive | 1 | 0
  NNRTI, ETR, resistant | 0 | 0
  NNRTI, NVP, sensitive | 1 | 3
  NNRTI, NVP, partially sensitive | 0 | 0
  NNRTI, NVP, resistant | 2 | 0
  NNRTI, RPV, sensitive | 1 | 3
  NNRTI, RPV, partially sensitive | 0 | 0
  NNRTI, RPV, resistant | 2 | 0
  NRTI, 3TC, sensitive | 3 | 3
  NRTI, 3TC, partially sensitive | 0 | 0
  NRTI, 3TC, resistant | 0 | 0
  NRTI, ABC, sensitive | 3 | 3
  NRTI, ABC, partially sensitive | 0 | 0
  NRTI, ABC, resistant | 0 | 0
  NRTI, FTC, sensitive | 3 | 3
  NRTI, FTC, partially sensitive | 0 | 0
  NRTI, FTC, resistant | 0 | 0
  NRTI, TDF, sensitive | 1 | 3
  NRTI, TDF, partially sensitive | 2 | 0
  NRTI, TDF, resistant | 0 | 0
  NRTI, ZDV, sensitive | 2 | 3
  NRTI, ZDV, partially sensitive | 0 | 0
  NRTI, ZDV, resistant | 1 | 0
  NRTI, d4T, sensitive | 3 | 3
  NRTI, d4T, partially sensitive | 0 | 0
  NRTI, d4T, resistant | 0 | 0
  NRTI, ddI, sensitive | 3 | 3
  NRTI, ddI, partially sensitive | 0 | 0
  NRTI, ddI, resistant | 0 | 0
  PI, ATV, sensitive | 3 | 3
  PI, ATV, partially sensitive | 0 | 0
  PI, ATV, resistant | 0 | 0
  PI, DRV, sensitive | 3 | 3
  PI, DRV, partially sensitive | 0 | 0
  PI, DRV, resistant | 0 | 0
  PI, FPV, sensitive | 3 | 3
  PI, FPV, partially sensitive | 0 | 0
  PI, FPV, resistant | 0 | 0
  PI, IDV, sensitive | 3 | 3
  PI, IDV, partially sensitive | 0 | 0
  PI, IDV, resistant | 0 | 0
  PI, LPV, sensitive | 3 | 3
  PI, LPV, partially sensitive | 0 | 0
  PI, LPV, resistant | 0 | 0
  PI, NFV, sensitive | 3 | 3
  PI, NFV, partially sensitive | 0 | 0
  PI, NFV, resistant | 0 | 0
  PI, RTV, sensitive | 3 | 3
  PI, RTV, partially sensitive | 0 | 0
  PI, RTV, resistant | 0 | 0
  PI, SQV, sensitive | 3 | 3
  PI, SQV, partially sensitive | 0 | 0
  PI, SQV, resistant | 0 | 0
  PI, TPV, sensitive | 3 | 3
  PI, TPV, partially sensitive | 0 | 0
  PI, TPV, resistant | 0 | 0

47. Secondary Outcome: Number of Participants With Genotypic Resistance Through Week 48
Description: Plasma samples were collected and analyzed from participants who met confirmed virologic withdrawal criteria. Genotypic Resistance data for the following drugs: DTG, EVG, RAL, DLV, EFV, ETR, NVP, RPV, 3TC, ABC, FTC, TDF, ZDV, d4T, ddI, ATV, DRV, FPV, IDV, LPV, NFV, RTV, SQV and TPV in participants meeting CVF criteria has been presented.
Time Frame: Week 48
Population: CVF Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 3 | 3
Participants
  INI, DTG, resistant | 0 | 0
  INI, DTG, resistance possible | 2 | 0
  INI, DTG, sensitive | 1 | 3
  INI, EVG, resistant | 2 | 0
  INI, EVG, resistance possible | 0 | 0
  INI, EVG, sensitive | 1 | 3
  INI, RAL, resistant | 2 | 0
  INI, RAL, resistance possible | 0 | 0
  INI, RAL, sensitive | 1 | 3
  NNRTI, DLV, resistant | 0 | 0
  NNRTI, DLV, resistance possible | 0 | 0
  NNRTI, DLV, sensitive | 3 | 3
  NNRTI, EFV, resistant | 0 | 0
  INI, EFV, resistance possible | 1 | 0
  NNRTI, EFV, sensitive | 2 | 3
  NNRTI, ETR, resistant | 0 | 0
  NNRTI, ETR, resistance possible | 0 | 0
  NNRTI, ETR, sensitive | 3 | 3
  NNRTI, NVP, resistant | 0 | 0
  NNRTI, NVP, resistance possible | 1 | 0
  NNRTI, NVP, sensitive | 2 | 3
  NNRTI, RPV, resistant | 3 | 0
  NNRTI, RPV, resistance possible | 0 | 0
  NNRTI, RPV, sensitive | 0 | 3
  NRTI, 3TC, resistant | 0 | 0
  NNRTI, 3TC, resistance possible | 0 | 0
  NRTI, 3TC, sensitive | 3 | 3
  NRTI, ABC, resistant | 0 | 0
  NRTI, ABC, resistance possible | 0 | 0
  NRTI, ABC, sensitive | 3 | 3
  NRTI, FTC, resistant | 0 | 0
  NRTI, FTC, resistance possible | 0 | 0
  NRTI, FTC, sensitive | 3 | 3
  NRTI, TDF, resistant | 0 | 0
  NRTI, TDF, resistance possible | 0 | 0
  NRTI, TDF, sensitive | 3 | 3
  NRTI, ZDV, resistant | 0 | 0
  NRTI, ZDV, resistance possible | 0 | 0
  NRTI, ZDV, sensitive | 3 | 3
  NRTI, d4T, resistant | 0 | 0
  NRTI, d4T, resistance possible | 0 | 0
  NRTI, d4T, sensitive | 3 | 3
  NRTI, ddI, resistant | 0 | 0
  NRTI, ddI, resistance possible | 0 | 0
  NRTI, ddI, sensitive | 3 | 3
  PI, ATV, resistant | 0 | 0
  PI, ATV, resistance possible | 0 | 0
  PI, ATV, sensitive | 3 | 3
  PI, ATV/r, resistant | 0 | 0
  PI, ATV/r, resistance possible | 0 | 0
  PI, ATV/r, sensitive | 3 | 3
  PI, DRV/r, resistant | 0 | 0
  PI, DRV/r, resistance possible | 0 | 0
  PI, DRV/r, sensitive | 3 | 3
  PI, FPV/r, resistant | 0 | 0
  PI, FPV/r, resistance possible | 0 | 0
  PI, FPV/r, sensitive | 3 | 3
  PI, IDV/r, resistant | 0 | 0
  PI, IDV/r, resistance possible | 0 | 0
  PI, IDV/r, sensitive | 3 | 3
  PI, LPV/r, resistant | 0 | 0
  PI, LPV/r, resistance possible | 0 | 0
  PI, LPV/r, sensitive | 3 | 3
  PI, NFV, resistant | 0 | 0
  PI, NFV, resistance possible | 0 | 0
  PI, NFV, sensitive | 3 | 3
  PI, RTV, resistant | 0 | 0
  PI, RTV, resistance possible | 0 | 0
  PI, RTV, sensitive | 3 | 3
  PI, SQV/r, resistant | 0 | 0
  PI, SQV/r, resistance possible | 0 | 0
  PI, SQV/r, sensitive | 3 | 3
  PI, TPV/r, resistant | 0 | 0
  PI, TPV/r, resistance possible | 1 | 0
  PI, TPV/r, sensitive | 2 | 3

48. Secondary Outcome: Area Under the Curve (AUC) for CAB LA
Description: AUC values are Bayesian pharmacokinetic (PK) parameter estimates obtained from a population PK meta-analysis of the data collected from studies 201584 and 201585# NCT02951052. Blood samples from the current study 201584 were collected at indicated time points to analyse concentration in plasma for CAB LA. The PK Population includes all participants who received CAB and / or RPV and undergo PK sampling during the study, and provide CAB and /or RPV plasma concentration data.
Time Frame: Pre-dose at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48; 1 Week post-dose at Weeks 5, 41, 2 hours post-dose at Weeks 4 and 48
Population: PK Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours*micrograms per milliliter
Groups:
- CAB LA: Participants in this arm received CAB 30 mg once daily for 4 Weeks during Maintenance Phase (Day 1 to Week 100). At Week 4b visit, participants received last dose of oral CAB and first dose CAB LA 600 mg injections. Participants received IM injections of CAB LA 400 mg at Week 8 and every four weeks through Week 100.
Arm/Group | CAB LA
Number analyzed (Participants) | 278
Hours*micrograms per milliliter | 2517.40 [2439.876 to 2597.394]

49. Secondary Outcome: AUC for RPV LA
Description: AUC values are Bayesian PK parameter estimates obtained from a population PK meta-analysis of the data collected from studies 201584 and 201585# NCT02951052. Blood samples from the current study 201584 were collected at indicated time points to analyse concentration in plasma for RPV LA
Time Frame: as for outcome 48
Population: PK Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours*nanograms per milliliter
Arm/Group | CAB LA
Number analyzed (Participants) | 278
Hours*nanograms per milliliter | 63989.13 [61489.692 to 66590.156]

50. Secondary Outcome: Plasma Trough Concentration (Ctrough) for CAB LA Evaluable
Description: Blood samples were collected at indicated time points for PK analysis of CAB LA.
Time Frame: Pre-dose at Weeks 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: PK population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per milliliter
Arm/Group | CAB LA
Number analyzed (Participants) | 278
Microgram per milliliter
  Pre-dose, Week 8, n=250: number analyzed (Participants) | 250
  Pre-dose, Week 8, n=250 | 1.5616 [1.4508 to 1.6808]
  Pre-dose, Week 12, n=237: number analyzed (Participants) | 237
  Pre-dose, Week 12, n=237 | 2.0141 [1.8990 to 2.1362]
  Pre-dose, Week 16, n=215: number analyzed (Participants) | 215
  Pre-dose, Week 16, n=215 | 2.0960 [1.9740 to 2.2255]
  Pre-dose, Week 20, n=233: number analyzed (Participants) | 233
  Pre-dose, Week 20, n=233 | 2.1739 [2.0580 to 2.2963]
  Pre-dose, Week 24, n=227: number analyzed (Participants) | 227
  Pre-dose, Week 24, n=227 | 2.3827 [2.2731 to 2.4976]
  Pre-dose, Week 28, n=220: number analyzed (Participants) | 220
  Pre-dose, Week 28, n=220 | 2.4683 [2.3421 to 2.6013]
  Pre-dose, Week 32, n=219: number analyzed (Participants) | 219
  Pre-dose, Week 32, n=219 | 2.6729 [2.5339 to 2.8196]
  Pre-dose, Week 36, n=215: number analyzed (Participants) | 215
  Pre-dose, Week 36, n=215 | 2.8590 [2.7096 to 3.0165]
  Pre-dose, Week 40, n=210: number analyzed (Participants) | 210
  Pre-dose, Week 40, n=210 | 2.9378 [2.7872 to 3.0966]
  Pre-dose, Week 44, n=217: number analyzed (Participants) | 217
  Pre-dose, Week 44, n=217 | 3.0133 [2.8739 to 3.1595]
  Pre-dose, Week 48, n=197: number analyzed (Participants) | 197
  Pre-dose, Week 48, n=197 | 3.1325 [2.9454 to 3.3315]

51. Secondary Outcome: Ctrough for RPV LA Evaluable
Description: Blood samples were collected at indicated time points for PK analysis of RPV LA.
Time Frame: Pre-dose at Weeks 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: as for outcome 50
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms per milliliter
Groups:
- RPV LA: Participants in this arm received RPV 25 mg once daily for 4 Weeks during Maintenance Phase (Day 1 to Week 100). At Week 4b visit, participants received last dose of oral RPV and first dose CAB LA 900 mg injections. Participants received IM injections of RPV LA 600 mg at Week 8 and every four weeks through Week 100.
Arm/Group | RPV LA
Number analyzed (Participants) | 278
Nanograms per milliliter
  Pre-dose, Week 8, n=251: number analyzed (Participants) | 251
  Pre-dose, Week 8, n=251 | 41.23 [38.74 to 43.88]
  Pre-dose, Week 12, n=236: number analyzed (Participants) | 236
  Pre-dose, Week 12, n=236 | 46.86 [43.82 to 50.12]
  Pre-dose, Week 16, n=217: number analyzed (Participants) | 217
  Pre-dose, Week 16, n=217 | 50.01 [47.06 to 53.15]
  Pre-dose, Week 20, n=233: number analyzed (Participants) | 233
  Pre-dose, Week 20, n=233 | 52.76 [49.79 to 55.91]
  Pre-dose, Week 24, n=228: number analyzed (Participants) | 228
  Pre-dose, Week 24, n=228 | 55.56 [52.48 to 58.82]
  Pre-dose, Week 28, n=220: number analyzed (Participants) | 220
  Pre-dose, Week 28, n=220 | 59.46 [55.43 to 63.79]
  Pre-dose, Week 32, n=220: number analyzed (Participants) | 220
  Pre-dose, Week 32, n=220 | 66.88 [62.95 to 71.05]
  Pre-dose, Week 36, n=215: number analyzed (Participants) | 215
  Pre-dose, Week 36, n=215 | 69.09 [64.90 to 73.55]
  Pre-dose, Week 40, n=210: number analyzed (Participants) | 210
  Pre-dose, Week 40, n=210 | 75.71 [71.38 to 80.29]
  Pre-dose, Week 44, n=216: number analyzed (Participants) | 216
  Pre-dose, Week 44, n=216 | 77.96 [73.87 to 82.28]
  Pre-dose, Week 48, n=197: number analyzed (Participants) | 197
  Pre-dose, Week 48, n=197 | 82.38 [77.82 to 87.22]

52. Secondary Outcome: Maximum Concentration (Cmax) in Plasma for CAB LA Evaluable at Week 41
Description: Blood samples will be collected at indicated time points for PK analysis of CAB LA.
Time Frame: Week 41- 1 Week post dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter
Arm/Group | CAB LA
Number analyzed (Participants) | 236
Micrograms per milliliter | 4.0334 [3.8488 to 4.2269]

53. Secondary Outcome: Cmax in Plasma for RPV LA Evaluable at Week 41
Description: Blood samples will be collected at indicated time points for PK analysis of RPV LA.
Time Frame: Week 41- 1 Week post dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms per milliliter
Arm/Group | RPV LA
Number analyzed (Participants) | 236
Nanograms per milliliter | 106.3 [101.03 to 111.28]

54. Other Pre Specified Outcome: Number of Participants With Different Demographic Parameters for Inter-subject Variability
Description: Blood samples were planned to be collected at indicated time points for PK analysis of CAB LA and RPV LA. Demographic parameters including, but not limited to, age, sex, race, body weight, body mass index, and relevant laboratory parameters were planned to be evaluated as potential predictors of inter subject variability for pharmacokinetic parameters.
Time Frame: Up to Week 48
Population: PK Population. This was an exploratory Outcome Measure. Data will not be analyzed and reported.
Arm/Group | CAB LA | RPV LA
Number analyzed (Participants) | 0 | 0

55. Secondary Outcome: Change From Week 5 in Dimension Scores Using Perception of Injection Questionnaire (PIN)-Last Observation Carried Forward (LOCF)
Description: PIN questionnaire explores bother of pain at injection site and injection site reactions (ISR),anxiety before and after injection, willingness to receive HIV injectable treatment and satisfaction with mode of treatment administration of individuals receiving injection and perceptions associated with receiving injections.This measure contains 21 items: pain at injection site, local site reactions, impact on functioning and willingness to pursue injectable treatment outside clinical trial. Scores range from 1 to 5; questions are phrased to ensure that 1:most favorable perception of vaccination, and 5:most unfavorable.Dimension scores include bother from ISR, leg movement, sleep and acceptability.Score of a domain is calculated as mean of all items with domain.Higher scores represent worse perception of injection.LOCF was primary method of analysis
Time Frame: Weeks 5 and at Weeks 41 and 48
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA (Q4W)
Number analyzed (Participants) | 270
Scores on a scale
  Bother of ISRs, Week 41 | -0.14 (0.551)
  Bother of ISRs, Week 48 | -0.14 (0.639)
  Leg movement, Week 41 | -0.58 (0.880)
  Leg movement, Week 48 | -0.63 (0.964)
  Sleep, Week 41 | -0.57 (0.925)
  Sleep, Week 48 | -0.58 (1.033)
  Acceptance, Week 41 | -0.36 (0.959)
  Acceptance, Week 48 | -0.40 (0.943)
Statistical Analysis 1: Comparison: CAB LA + RPV LA (Q4W); Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney) — Week 41/48 was compared with the 1st visit (Week 5) based on Wilcoxon signed-rank test, respectively. p-values are derived for 'Acceptance' only and not adjusted for multiple testing

56. Secondary Outcome: Percentage of Participants With Extremely or Very Acceptable Pain and Local Reaction: Acceptability Score on PIN Questionnaire
Description: PIN questionnaire explores bother of pain at injection site and injection site reactions (ISR),anxiety before and after injection, willingness to receive HIV injectable treatment, following visit and satisfaction with mode of treatment administration of individuals receiving injection and perceptions associated with receiving injections.This measure contains 21 items: pain at injection site, local site reactions, impact on functioning and willingness to pursue injectable treatment outside clinical trial. Scores range from 1 to 5; questions are phrased to ensure that 1:most favorable perception of vaccination, and 5:most unfavorable.Dimension scores include bother from ISR, leg movement, sleep and acceptability.Score of a domain is calculated as mean of all items with domain.Higher scores represent worse perception of injection.LOCF was primary method of analysis.
Time Frame: Weeks 5, 41 and 48
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Number; unit: Percentage of participants
Arm/Group | CAB LA + RPV LA (Q4W)
Number analyzed (Participants) | 283
Percentage of participants
  Local reactions, Week 5, totally acceptable, n=270: number analyzed (Participants) | 270
  Local reactions, Week 5, totally acceptable, n=270 | 47
  Local reactions,Week 5, very acceptable, n=270: number analyzed (Participants) | 270
  Local reactions,Week 5, very acceptable, n=270 | 29
  Local reactions, Week 5, moderate, n=270: number analyzed (Participants) | 270
  Local reactions, Week 5, moderate, n=270 | 16
  Local reactions, Week 5, little acceptable, n=270: number analyzed (Participants) | 270
  Local reactions, Week 5, little acceptable, n=270 | 6
  Local reactions, Week 5, not at all, n=270: number analyzed (Participants) | 270
  Local reactions, Week 5, not at all, n=270 | 3
  Pain, Week 5, totally acceptable, n=270: number analyzed (Participants) | 270
  Pain, Week 5, totally acceptable, n=270 | 33
  Pain, Week 5, very acceptable, n=270: number analyzed (Participants) | 270
  Pain, Week 5, very acceptable, n=270 | 28
  Pain, Week 5, moderate acceptable, n=270: number analyzed (Participants) | 270
  Pain, Week 5, moderate acceptable, n=270 | 24
  Pain, Week 5, little acceptable, n=270: number analyzed (Participants) | 270
  Pain, Week 5, little acceptable, n=270 | 11
  Pain, Week 5, not at all acceptable, n=270: number analyzed (Participants) | 270
  Pain, Week 5, not at all acceptable, n=270 | 5
  Local reactions, week 41, totally, n=276: number analyzed (Participants) | 276
  Local reactions, week 41, totally, n=276 | 57
  Local reactions, Week 41, very acceptable, n=276: number analyzed (Participants) | 276
  Local reactions, Week 41, very acceptable, n=276 | 29
  Local reactions, Week 41, moderate, n=276: number analyzed (Participants) | 276
  Local reactions, Week 41, moderate, n=276 | 11
  Local reactions, Week 41, little acceptable, n=276: number analyzed (Participants) | 276
  Local reactions, Week 41, little acceptable, n=276 | 3
  Local reactions, Week 41, not at all, n=276: number analyzed (Participants) | 276
  Local reactions, Week 41, not at all, n=276 | 1
  Pain, Week 41, totally acceptable, n=276: number analyzed (Participants) | 276
  Pain, Week 41, totally acceptable, n=276 | 45
  Pain, Week 41, very acceptable, n=276: number analyzed (Participants) | 276
  Pain, Week 41, very acceptable, n=276 | 35
  Pain, Week 41, moderate acceptable, n=276: number analyzed (Participants) | 276
  Pain, Week 41, moderate acceptable, n=276 | 14
  Pain, Week 41, little acceptable, n=276: number analyzed (Participants) | 276
  Pain, Week 41, little acceptable, n=276 | 4
  Pain, Week 41, not at all acceptable, n=276: number analyzed (Participants) | 276
  Pain, Week 41, not at all acceptable, n=276 | 1
  Local reactions, week 48, totally, n=278: number analyzed (Participants) | 278
  Local reactions, week 48, totally, n=278 | 55
  Local reactions, Week 48, very acceptable, n=278: number analyzed (Participants) | 278
  Local reactions, Week 48, very acceptable, n=278 | 31
  Local reactions, Week 48, moderate, n=278: number analyzed (Participants) | 278
  Local reactions, Week 48, moderate, n=278 | 11
  Local reactions, Week 48, little acceptable, n=278: number analyzed (Participants) | 278
  Local reactions, Week 48, little acceptable, n=278 | 2
  Local reactions, Week 48, not at all, n=278: number analyzed (Participants) | 278
  Local reactions, Week 48, not at all, n=278 | 1
  Pain, Week 48, totally acceptable, n=278: number analyzed (Participants) | 278
  Pain, Week 48, totally acceptable, n=278 | 49
  Pain, Week 48, very acceptable, n=278: number analyzed (Participants) | 278
  Pain, Week 48, very acceptable, n=278 | 35
  Pain, Week 48, moderate acceptable, n=278: number analyzed (Participants) | 278
  Pain, Week 48, moderate acceptable, n=278 | 12
  Pain, Week 48 little acceptable, n=278: number analyzed (Participants) | 278
  Pain, Week 48 little acceptable, n=278 | 3
  Pain, Week 48, not at all acceptable, n=278: number analyzed (Participants) | 278
  Pain, Week 48, not at all acceptable, n=278 | 1

57. Secondary Outcome: Change From Baseline in Life Satisfaction (LISAT) Using HIV/AIDs-targeted Quality of Life (HATQoL) Questionnaire
Description: The HATQoL questionnaire was used to assess health related QoL (HRQoL). It comprises of three dimensions: life satisfaction (LISAT), medication worries (MEDWO) and disclosure worries (DISWO). For LISAT domain, each question is scored as 1-5, where 5 corresponds to satisfaction 'all of time' and 1 as 'none of time'. Total score for the LISAT domain (sum of item scores for questions 1a to 1d) is transformed to a 0-100 scale using formula:[100 divided by (20 minus 4)]*(raw total score for LISAT minus 4). Higher the LISAT score, greater satisfaction to life. Transformed dimension score for each domain was summarized and analyzed. LOCF was used as primary method of analysis. Measure type was considered as mean for adjusted mean and dispersion measure as 95% CI. Baseline value is defined as the last available value up to and including the date of first Maintenance phase dose of IP. Change from Baseline value is calculated as value at post-dose visit minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 56
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Scores on a scale
  Week 24, n=252, 253: number analyzed (Participants) | 252 | 253
  Week 24, n=252, 253 | 0.4 [-1.3 to 2.1] | -0.8 [-2.5 to 0.9]
  Week 48, n=253, 258: number analyzed (Participants) | 253 | 258
  Week 48, n=253, 258 | 0.9 [-0.8 to 2.6] | 0.0 [-1.6 to 1.7]
Statistical Analysis 1: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Other; p = 0.307, ANCOVA; Adjusted difference = 1.2, 95% CI 2-sided [-1.1 to 3.6] — Treatment comparison at Week 24 is presented, adjusted for Maintenance Baseline (Day 1) Score, Induction Baseline (Week -20) HIV-1 RNA (<100,000, >=100,000 c/mL), gender at birth, age (<50, >= 50 Years) and race (white, non-white)
Statistical Analysis 2: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Other; p = 0.472, ANCOVA; Adjusted difference = 0.9, 95% CI 2-sided [-1.5 to 3.2] — Treatment comparison at Week 48 is presented, adjusted for Maintenance Baseline (Day 1) Score, Induction Baseline (Week -20) HIV-1 RNA (<100,000, >=100,000 c/mL), gender at birth, age (<50, >= 50 Years) and race (white, non-white)

58. Secondary Outcome: Change From Baseline in HIV Medication, MEDWO Using HATQoL
Description: The HATQoL questionnaire was used to assess HRQoL. It comprises of three dimensions: LISAT, MEDWO and DISWO. For the MEDWO domain, each question is scored as 1-5, where 5 is associated with medication worry 'none of the time' and 1 as 'all of the time'. The total score for the MEDWO domain (sum of item scores for questions 2a to 3e) is transformed to a 0-100 scale using formula: [100 divided by (25 minus 5)]* (raw total score for MEDWO minus 5). Higher MEDWO scores correspond to lower medication worries. Transformed dimension score for each domain was summarized and analyzed. LOCF was used as primary method of analysis. Measure type was considered as mean for adjusted mean and dispersion measure as 95% CI. Baseline value is defined as the last available value up to and including the date of first Maintenance phase dose of IP. Change from Baseline value is calculated as value at post-dose visit minus Baseline value.
Time Frame: Baseline and at Weeks 24 and 48
Population: as for outcome 56
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Scores on a scale
  Week 24, n=252, 253: number analyzed (Participants) | 252 | 253
  Week 24, n=252, 253 | 3.2 [1.6 to 4.7] | 1.4 [-0.1 to 3.0]
  Week 48, n=253, 258: number analyzed (Participants) | 253 | 258
  Week 48, n=253, 258 | 1.4 [-0.3 to 3.1] | 1.3 [-0.4 to 3.0]
Statistical Analysis 1: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Other; p = 0.116, ANCOVA; Adjusted difference = 1.8, 95% CI 2-sided [-0.4 to 3.9] — [estimate comment as in outcome 57, analysis 1]
Statistical Analysis 2: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Other; p = 0.944, ANCOVA; Adjusted difference = 0.1, 95% CI 2-sided [-2.3 to 2.5] — [estimate comment as in outcome 57, analysis 2]

59. Secondary Outcome: Change From Baseline in DISWO Using HATQoL
Description: The HATQoL questionnaire was used to assess HRQoL. It comprises of three dimensions: LISAT, MEDWO and DISWO. For the DISWO domain, each question is scored as 1-5, where 5 is associated with disclosure worry 'none of the time' and 1 as 'all of the time'. The total score for the DISWO domain (sum of item scores for questions 3a to 3e) is transformed to a 0-100 scale using formula: [100 divided by (25 minus 5)]* (raw total score for DISWO minus 5). Higher DISWO total scores correspond to lower disclosure worries. Transformed dimension score for each domain was summarized and analyzed. LOCF was used as primary method of analysis. Measure type was considered as mean for adjusted mean and dispersion measure as 95% CI. Baseline value is defined as the last available value up to and including the date of first Maintenance phase dose of IP. Change from Baseline value is calculated as value at post-dose visit minus Baseline value.
Time Frame: Baseline and at Weeks 24 and 48
Population: as for outcome 56
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Scores on a scale
  Week 24, n=252, 253: number analyzed (Participants) | 252 | 253
  Week 24, n=252, 253 | -0.8 [-3.9 to 2.3] | 0.5 [-2.6 to 3.6]
  Week 48, n=253, 258: number analyzed (Participants) | 253 | 258
  Week 48, n=253, 258 | -3.6 [-6.6 to -0.6] | 1.1 [-1.9 to 4.0]
Statistical Analysis 1: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Other; p = 0.552, ANCOVA; Adjusted difference = -1.3, 95% CI 2-sided [-5.7 to 3.0] — [estimate comment as in outcome 57, analysis 1]
Statistical Analysis 2: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Other; p = 0.033, ANCOVA; Adjusted difference = -4.6, 95% CI 2-sided [-8.9 to -0.4] — [estimate comment as in outcome 57, analysis 2]

60. Secondary Outcome: Change From Baseline in Health Status Using 12-item Short Form Survey (SF-12)
Description: The SF-12 questionnaire consists of 7 questions which measures degree of general health status and mental health distress. Each question is scored 0-5, except for question 2 scored 0-3. HRQoL using SF-12 for physical component summary (PCS) and mental component summary (MCS) were assessed for two treatment groups.Missing component scores was imputed using LOCF.PCS/MCS are calculated using computer software purchased from QualityMetric (http://www.qualitymetric.com).The higher the score, the better will be the health status.Measure type was considered as mean for adjusted mean and dispersion measure as 95% CI. Baseline value is defined as the last available recorded value up to and including the date of first Maintenance phase dose of IP. Change from Baseline value is calculated as value at post-dose visit minus Baseline value.
Time Frame: Baseline and at Weeks 24 and 48
Population: as for outcome 56
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Scores on a scale
  MCS, Week 24, n=251, 253: number analyzed (Participants) | 251 | 253
  MCS, Week 24, n=251, 253 | -0.045 [-0.963 to 0.874] | -1.066 [-1.980 to -0.151]
  MCS, Week 48, n=252, 258: number analyzed (Participants) | 252 | 258
  MCS, Week 48, n=252, 258 | -0.013 [-0.973 to 0.947] | -1.116 [-2.065 to -0.167]
  PCS, Week 24, n=251, 253: number analyzed (Participants) | 251 | 253
  PCS, Week 24, n=251, 253 | -0.019 [-0.568 to 0.531] | -0.201 [-0.748 to 0.347]
  PCS, Week 48, n=252, 258: number analyzed (Participants) | 252 | 258
  PCS, Week 48, n=252, 258 | -0.294 [-0.881 to 0.293] | -0.126 [-0.706 to 0.455]
Statistical Analysis 1: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Other; p = 0.122, ANCOVA; Adjusted difference = 1.021, 95% CI 2-sided [-0.275 to 2.318] — Treatment comparison of SF-12 MCS at Week 24 is presented, adjusted for Maintenance Baseline (Day 1) Score, Induction Baseline (Week -20) HIV-1 RNA (<100,000, >=100,000 c/mL), gender at birth, age (<50, >= 50 Years) and race (white, non-white)
Statistical Analysis 2: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Other; p = 0.109, ANCOVA; Adjusted difference = 1.103, 95% CI 2-sided [-0.248 to 2.453] — Treatment comparison of SF-12 MCS at Week 48 is presented, adjusted for Maintenance Baseline (Day 1) Score, Induction Baseline (Week -20) HIV-1 RNA (<100,000, >=100,000 c/mL), gender at birth, age (<50, >= 50 Years) and race (white, non-white)
Statistical Analysis 3: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Other; p = 0.645, ANCOVA; Adjusted difference = 0.182, 95% CI 2-sided [-0.594 to 0.958] — Treatment comparison of SF-12 PCS at Week 24 is presented, adjusted for Maintenance Baseline (Day 1) Score, Induction Baseline (Week -20) HIV-1 RNA (<100,000, >=100,000 c/mL), gender at birth, age (<50, >= 50 Years) and race (white, non-white)
Statistical Analysis 4: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Other; p = 0.689, ANCOVA; Adjusted difference = -0.169, 95% CI 2-sided [-0.994 to 0.657] — Treatment comparison of SF-12 PCS at Week 48 is presented, adjusted for Maintenance Baseline (Day 1) Score, Induction Baseline (Week -20) HIV-1 RNA (<100,000, >=100,000 c/mL), gender at birth, age (<50, >= 50 Years) and race (white, non-white)

61. Secondary Outcome: Change From Baseline in Total Treatment Satisfaction Using HIV Treatment Satisfaction Questionnaire (HIVTSQs) at Weeks 4b, 24 and 44
Description: HIVTSQs (status version) total treatment satisfaction score is computed with 1-11 items. Items 1-11 are summed to produce score with possible range of 0 to 66. Higher the score, greater improvement in satisfaction with treatment; lower score, greater the deterioration in satisfaction with treatment. A score of 0 represents no change. LOCF was primary method of analysis. Baseline value is defined as the last available value up to and including the date of first Maintenance phase dose of IP. Change from Baseline value is calculated as value at post-dose visit minus Baseline value. Adjusted mean and 95% CI of adjusted mean values has been presented.
Time Frame: Baseline and at Weeks 4b, 24 and 44
Population: as for outcome 56
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Scores on a scale
  Week 4b, n=257, 0: number analyzed (Participants) | 257 | 0
  Week 4b, n=257, 0 | 0.2 [-0.5 to 1.0] |
  Week 24, n=257, 253: number analyzed (Participants) | 257 | 253
  Week 24, n=257, 253 | 1.6 [0.8 to 2.5] | -0.5 [-1.4 to 0.3]
  Week 44, n=257, 256: number analyzed (Participants) | 257 | 256
  Week 44, n=257, 256 | 1.3 [0.5 to 2.1] | 0.5 [-0.3 to 1.4]
Statistical Analysis 1: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Other; p < 0.001, ANCOVA; Adjusted difference = 2.2, 95% CI 2-sided [1.0 to 3.4] — [estimate comment as in outcome 57, analysis 1]
Statistical Analysis 2: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Other; p = 0.217, ANCOVA; Adjusted difference = 0.7, 95% CI 2-sided [-0.4 to 1.9] — Treatment comparison at Week 44 is presented, adjusted for Maintenance Baseline (Day 1) Score, Induction Baseline (Week -20) HIV-1 RNA (<100,000, >=100,000 c/mL), gender at birth, age (<50, >= 50 Years) and race (white, non-white)

62. Secondary Outcome: Change in Treatment Satisfaction Over Time Using HIVTSQc at Week 48
Description: HIVTSQc (change version) total treatment satisfaction score is computed with 1-11 items. Items 1-11 are summed to produce score with possible range:-33 to 33. Higher scores represent greater improvement in treatment satisfaction compared to satisfaction with treatment received during the induction phase; lower scores representedeterioration in satisfaction with treatment. A score of 0 represents no change. LOCF was primary method of analysis. Baseline value is defined as the last available value up to and including the date of first Maintenance phase dose of IP. Change from Baseline value is calculated as value at post-dose visit minus Baseline value.
Time Frame: Week 48
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 263 | 266
Scores on a scale | 29.6 (0.49) | 25.5 (0.48)
Statistical Analysis 1: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Other; p < 0.001, ANOVA; Difference = 4.1, 95% CI 2-sided [2.8 to 5.5] — Treatment comparison of HIVTSQc-total treatment satisfaction score at Week 48 is presented, adjusted for Induction Baseline (Week -20) HIV-1 RNA (<100,000, >=100,000 c/mL), gender at birth, age (<50, >= 50 Years) and race (white, non-white)

63. Secondary Outcome: Change From Baseline in Individual Item Scores of HIVTSQs at Weeks 4b, 24 and 44
Description: HIVTSQs (status version) is a 12 item questionnaire. The individual item scores are ratedas 6 (very satisfied, convenient, flexible, etc.) to 0 (very dissatisfied, inconvenient, inflexible, etc.). Higher scores represent greater treatment satisfaction as compared to the past few weeks. LOCF was used as primary method of analysis. Baseline value is defined as the last available value up to and including the date of first Maintenance phase dose of IP. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline and at Weeks 4b, 24 and 44
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Scores on a scale
  Item 1; Week 4b, n=257, 0: number analyzed (Participants) | 257 | 0
  Item 1; Week 4b, n=257, 0 | -0.0 (0.91) |
  Item 1; Week 24, n=257, 255: number analyzed (Participants) | 257 | 255
  Item 1; Week 24, n=257, 255 | 0.1 (0.96) | -0.0 (0.95)
  Item 1; Week 44, n=257, 258: number analyzed (Participants) | 257 | 258
  Item 1; Week 44, n=257, 258 | 0.0 (1.02) | 0.0 (0.93)
  Item 2; Week 4b, n=257, 0: number analyzed (Participants) | 257 | 0
  Item 2; Week 4b, n=257, 0 | 0.0 (0.61) |
  Item 2; Week 24, n=257, 255: number analyzed (Participants) | 257 | 255
  Item 2; Week 24, n=257, 255 | -0.0 (0.62) | -0.0 (0.87)
  Item 2; Week 44, n=257, 258: number analyzed (Participants) | 257 | 258
  Item 2; Week 44, n=257, 258 | -0.1 (0.61) | 0.1 (0.62)
  Item 3; Week 4b, n=257, 0: number analyzed (Participants) | 257 | 0
  Item 3; Week 4b, n=257, 0 | 0.2 (1.02) |
  Item 3; Week 24, n=257, 255: number analyzed (Participants) | 257 | 255
  Item 3; Week 24, n=257, 255 | -0.1 (1.21) | -0.0 (1.16)
  Item 3; Week 44, n=257, 258: number analyzed (Participants) | 257 | 258
  Item 3; Week 44, n=257, 258 | -0.0 (1.35) | 0.1 (1.22)
  Item 4; Week 4b, n=257, 0: number analyzed (Participants) | 257 | 0
  Item 4; Week 4b, n=257, 0 | 0.1 (1.02) |
  Item 4; Week 24, n=257, 255: number analyzed (Participants) | 257 | 255
  Item 4; Week 24, n=257, 255 | 0.1 (1.03) | -0.0 (1.14)
  Item 4; Week 44, n=257, 258: number analyzed (Participants) | 257 | 258
  Item 4; Week 44, n=257, 258 | 0.0 (1.08) | 0.1 (1.10)
  Item 5; Week 4b, n=257, 0: number analyzed (Participants) | 257 | 0
  Item 5; Week 4b, n=257, 0 | 0.1 (0.98) |
  Item 5; Week 24, n=257, 255: number analyzed (Participants) | 257 | 255
  Item 5; Week 24, n=257, 255 | 0.4 (1.22) | -0.1 (1.05)
  Item 5; Week 44, n=257, 258: number analyzed (Participants) | 257 | 258
  Item 5; Week 44, n=257, 258 | 0.3 (1.28) | 0.0 (1.06)
  Item 6; Week 4b, n=257, 0: number analyzed (Participants) | 257 | 0
  Item 6; Week 4b, n=257, 0 | 0.1 (1.40) |
  Item 6; Week 24, n=257, 255: number analyzed (Participants) | 257 | 255
  Item 6; Week 24, n=257, 255 | 0.3 (1.47) | -0.1 (1.63)
  Item 6; Week 44, n=257, 258: number analyzed (Participants) | 257 | 258
  Item 6; Week 44, n=257, 258 | 0.3 (1.70) | 0.2 (1.48)
  Item 7; Week 4b, n=257, 0: number analyzed (Participants) | 257 | 0
  Item 7; Week 4b, n=257, 0 | 0.0 (0.83) |
  Item 7; Week 24, n=257, 255: number analyzed (Participants) | 257 | 255
  Item 7; Week 24, n=257, 255 | 0.0 (0.79) | 0.0 (1.02)
  Item 7; Week 44, n=257, 258: number analyzed (Participants) | 257 | 258
  Item 7; Week 44, n=257, 258 | 0.1 (0.85) | 0.1 (0.95)
  Item 8; Week 4b, n=257, 0: number analyzed (Participants) | 257 | 0
  Item 8; Week 4b, n=257, 0 | -0.0 (1.06) |
  Item 8; Week 24, n=257, 255: number analyzed (Participants) | 257 | 255
  Item 8; Week 24, n=257, 255 | 0.2 (1.22) | -0.0 (1.11)
  Item 8; Week 44, n=257, 258: number analyzed (Participants) | 257 | 258
  Item 8; Week 44, n=257, 258 | 0.2 (1.27) | 0.1 (1.16)
  Item 9; Week 4b, n=257, 0: number analyzed (Participants) | 257 | 0
  Item 9; Week 4b, n=257, 0 | -0.1 (0.85) |
  Item 9; Week 24, n=257, 255: number analyzed (Participants) | 257 | 255
  Item 9; Week 24, n=257, 255 | 0.0 (0.78) | -0.1 (1.11)
  Item 9; Week 44, n=257, 258: number analyzed (Participants) | 257 | 258
  Item 9; Week 44, n=257, 258 | 0.0 (0.85) | 0.0 (1.01)
  Item 10; Week 4b, n=257, 0: number analyzed (Participants) | 257 | 0
  Item 10; Week 4b, n=257, 0 | -0.1 (1.16) |
  Item 10; Week 24, n=257, 256: number analyzed (Participants) | 257 | 256
  Item 10; Week 24, n=257, 256 | 0.4 (1.28) | -0.1 (1.35)
  Item 10; Week 44, n=257, 259: number analyzed (Participants) | 257 | 259
  Item 10; Week 44, n=257, 259 | 0.4 (1.33) | -0.0 (1.20)
  Item 11; Week 4b, n=257, 0: number analyzed (Participants) | 257 | 0
  Item 11; Week 4b, n=257, 0 | -0.0 (1.02) |
  Item 11; Week 24, n=257, 255: number analyzed (Participants) | 257 | 255
  Item 11; Week 24, n=257, 255 | 0.2 (1.18) | -0.1 (0.99)
  Item 11; Week 44, n=257, 258: number analyzed (Participants) | 257 | 258
  Item 11; Week 44, n=257, 258 | 0.1 (1.18) | 0.0 (0.97)
  Item 12; Week 4b, n=257, 0: number analyzed (Participants) | 257 | 0
  Item 12; Week 4b, n=257, 0 | -0.0 (0.99) |
  Item 12; Week 24, n=257, 255: number analyzed (Participants) | 257 | 255
  Item 12; Week 24, n=257, 255 | -0.4 (1.26) | 0.1 (1.19)
  Item 12; Week 44, n=257, 258: number analyzed (Participants) | 257 | 258
  Item 12; Week 44, n=257, 258 | -0.5 (1.20) | 0.1 (1.29)

64. Secondary Outcome: Change From Baseline in Treatment Acceptance at Weeks 8, 24 and 48 Using "General Acceptance" Dimension of the Chronic Treatment Acceptance (ACCEPT) Questionnaire
Description: ACCEPT questionnaire is generic medication acceptance measure assessing how participants weigh advantages and disadvantages of long-term medication. It consists 25 items, capturing six dimensions. 3 questions focusing on general acceptance of study medication were analyzed. Items scores are rated as 1-5 :1-totally disagree,2-somewhat disagree,3-somewhat agree,4-totally agree and 5-I don't know. The acceptance domain score (ranging from 0 to 100) is calculated using the following formula:100*(mean of recoded items in dimension minus 1) divided by 2.LOCF was primary method of analysis. Measure type is mean for adjusted mean and dispersion measure: 95% CI. Baseline value is defined as the last available value up to and including the date of first Maintenance phase dose of IP. Change from Baseline value is calculated as value at post-dose visit minus Baseline value.
Time Frame: Baseline and at Weeks 8, 24 and 48
Population: as for outcome 56
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA (Q4W) | ABC/ DTG/ 3TC
Number analyzed (Participants) | 283 | 283
Scores on a scale
  Week 8, n=253, 256: number analyzed (Participants) | 253 | 256
  Week 8, n=253, 256 | 3.3 [0.8 to 5.8] | 1.2 [-1.3 to 3.6]
  Week 24, 255, 261: number analyzed (Participants) | 255 | 261
  Week 24, 255, 261 | 3.7 [1.1 to 6.4] | 1.1 [-1.5 to 3.7]
  Week 48, n=255, 262: number analyzed (Participants) | 255 | 262
  Week 48, n=255, 262 | 3.0 [0.4 to 5.6] | 0.8 [-1.7 to 3.4]
Statistical Analysis 1: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Other; p = 0.232, ANCOVA; Adjusted difference = 2.2, 95% CI 2-sided [-1.4 to 5.7] — Treatment comparison at Week 8 is presented, adjusted for Maintenance Baseline (Day 1) Score, Induction Baseline (Week -20) HIV-1 RNA (<100,000, >=100,000 c/mL), gender at birth, age (<50, >= 50 Years) and race (white, non-white)
Statistical Analysis 2: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Other; p = 0.154, ANCOVA; Adjusted difference = 2.7, 95% CI 2-sided [-1.0 to 6.4] — Treatment comparison Week 24 is presented, adjusted for Maintenance Baseline (Day 1) Score, Induction Baseline (Week -20) HIV-1 RNA (<100,000, >=100,000 c/mL), gender at birth, age (<50, >= 50 Years) and race (white, non-white)
Statistical Analysis 3: Comparison: CAB LA + RPV LA (Q4W) vs ABC/ DTG/ 3TC; Test type: Other; p = 0.236, ANCOVA; Adjusted difference = 2.2, 95% CI 2-sided [-1.4 to 5.8] — [estimate comment as in outcome 57, analysis 2]

65. Secondary Outcome: Change From 4b in Tolerability of Injection at Weeks 5, 40 and 41 Using Numeric Rating Scale (NRS) Within CAB LA+RPV LA Arm
Description: The NRS questionnaire is used to assess the tolerability of injections in CAB LA+RPV LA arm only. The questionnaire consists of one single question and will assess maximum level of pain experienced with the most recent injections ranking from no pain (0) to extreme pain (10). Missing scores was imputed using LOCF.
Time Frame: Weeks 4b, 5, 40 and 41
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA (Q4W)
Number analyzed (Participants) | 263
Scores on a scale
  Week 5 | 1.8 (2.78)
  Week 40 | 0.8 (2.72)
  Week 41 | 0.4 (2.69)

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected up to an average of 59 weeks.
Description: AEs and SAEs were collected in Safety population.
Groups:
- CAB LA+RPV LA (Q4W): Participants who received ABC/DTG/3TC for 20 Weeks (Week [-20] to Day 1) in the Induction Phase and who have an HIV-1 ribonucleic acid (RNA) <50 copies per millilter (c/mL) at Week (-4) entered Maintenance Phase (Day 1 to Week 100) to begin oral therapy with CAB 30 milligram (mg) + RPV 25 mg once daily for 4 Weeks. At Week 4b visit, participants received last dose of oral CAB + RPV and first dose CAB LA 600 mg + RPV LA 900 mg injections. Participants received intramuscular (IM) injections of CAB LA 400 mg and RPV LA 600 mg at Week 8 and every four weeks (Q4W) through Week 100. After completion of Maintenance Phase, participants who chose to enter Extension Phase will continue to receive both CAB LA and RPV LA. Participants withdrawn from study treatment who received at least one CAB LA+RPV LA injection were required to enter a 52-week long term follow-up period.
Arm/Group | CAB LA+RPV LA (Q4W) | ABC/ DTG/ 3TC
All-Cause Mortality (participants affected / at risk) | 0/283 | 0/283
Serious Adverse Events (participants affected / at risk) | 18/283 | 12/283
Other Adverse Events (participants affected / at risk) | 252/283 | 138/283
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAB LA+RPV LA (Q4W) (N=283) | ABC/ DTG/ 3TC (N=283)
Hepatitis A (Infections and infestations) | 3 (3) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchitis pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Hydrocholecystis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Priapism (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Rectal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAB LA+RPV LA (Q4W) (N=283) | ABC/ DTG/ 3TC (N=283)
Injection site pain (General disorders) | 227 (1879) | 0 (0)
Nasopharyngitis (Infections and infestations) | 56 (92) | 48 (70)
Upper respiratory tract infection (Infections and infestations) | 38 (50) | 28 (35)
Headache (Nervous system disorders) | 39 (48) | 21 (24)
Diarrhoea (Gastrointestinal disorders) | 32 (40) | 25 (30)
Influenza (Infections and infestations) | 25 (27) | 20 (22)
Injection site nodule (General disorders) | 44 (86) | 0 (0)
Injection site induration (General disorders) | 38 (82) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 23 (23) | 13 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (26) | 13 (14)
Nausea (Gastrointestinal disorders) | 16 (17) | 11 (12)
Gastroenteritis (Infections and infestations) | 15 (18) | 10 (10)
Pyrexia (General disorders) | 21 (33) | 4 (4)
Pharyngitis (Infections and infestations) | 15 (16) | 9 (9)
Injection site swelling (General disorders) | 23 (38) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 16 (18) | 3 (4)
Dizziness (Nervous system disorders) | 15 (17) | 3 (3)
Injection site pruritus (General disorders) | 16 (25) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT02938520/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT02938520/SAP_002.pdf